Obbvie Upadacitinib

M13-545 Protocol Amendment 8 EudraCT 2015-003334-27

#### 1.0 Title Page

# **Clinical Study Protocol M13-545**

A Phase 3, Randomized, Double-Blind Study Comparing Upadacitinib (ABT-494) Once Daily Monotherapy to Methotrexate (MTX) Monotherapy in MTX-Naïve Subjects with Moderately to Severely **Active Rheumatoid Arthritis** 

# Incorporating Administrative Changes 1, 2, 3 and 4, and Amendments 1, 2, 3, 4, 5, 6, 7, and 8

AbbVie Investigational

Product:

Date:

03 December 2020

Upadacitinib

Development Phase:

Study Design:

A 48-week randomized, double-blind, parallel-group, active

comparator-controlled treatment period followed by a long-term extension

period

EudraCT Number: 2015-003334-27

Investigators: Multicenter Trial (Investigator information is on file at AbbVie)

AbbVie\* Sponsor:

> 1 North Waukegan Road North Chicago, IL 60064

> > MD

Sponsor/Emergency

Contact:

Therapeutic Area Medical Director

AbbVie Inc.

1 North Waukegan Road North Chicago, IL 60064 Office: Mobile: Fax: Email:

Emergency 24 hour Number: +1 973-784-6402

This study will be conducted in compliance with the protocol, Good Clinical Practice and all other applicable regulatory requirements, including the archiving of essential documents.

#### **Confidential Information**

No use or disclosure outside AbbVie is permitted without prior written authorization from AbbVie.

<sup>\*</sup> The specific contact details of the AbbVie legal/regulatory entity (person) within the relevant country are provided within the clinical trial agreement with the Investigator/Institution and in the Clinical Trial Application with the Competent Authority.



# 1.1 Protocol Amendment: Summary of Changes

# **Previous Protocol Versions**

| Protocol | Date |
|-----------------------------------------|-------------------|
| Original | 01 October 2015 |
| Amendment 1 | 15 January 2016 |
| Administrative Change 1 | 22 January 2016 |
| Amendment 2 | 29 February 2016 |
| Amendment 2.01 (Japan Only) | 07 March 2016 |
| Amendment 3 | 31 May 2016 |
| Amendment 3.01 (Japan Only) | 25 July 2016 |
| Amendment 4 | 18 August 2016 |
| Amendment 4.01 (Japan Only) | 18 October 2016 |
| Administrative Change 2 | 02 November 2016 |
| Amendment 4.02 (China Only) | 21 December 2016 |
| Amendment 5 | 17 December 2017 |
| Amendment 5.01 (Japan Only) | 06 February 2018 |
| Amendment 5.02 (China Only) | 07 February 2018 |
| Administrative Change 3 | 19 March 2018 |
| Administrative Change 4 | 07 February 2019 |
| Amendment 5.01.01 (Japan Only) | 15 July 2019 |
| Amendment 6 | 16 December 2019 |
| Amendment 6.01 (Japan Only) | 03 March 2020 |
| Amendment 6.02 (VHP and Lithuania Only) | 06 March 2020 |
| Amendment 7 | 01 July 2020 |
| Administrative Change 5 (Japan Only) | 15 September 2020 |

# The purpose of this amendment is to:

- Apply administrative changes throughout the protocol.

  \*Rationale: Revised text to improve consistency and readability, and/or provide clarification.
- Update Section 1.2, Synopsis

**Rationale:** Revised to be consistent with Amendment 7 revisions.

• Update Section 1.3, List of Abbreviations

Rationale: Updated to include new terms, Direct-to Patient (DTP) and Coronavirus Disease – 19 (COVID-19)

• Update Section 3.2, Benefits and Risks

**Rationale:** Revised to include the evaluation of the benefit and risk to subjects participating in the study relative to COVID-19.

- Update Section 5.1, Overall Study Design and Plan: Description *Rationale:* Added provisions for virtual or alternative locations for study visits in the event of a pandemic situation like COVID-19 or any state of emergency (e.g., natural disaster, conflict/combat) to ensure the safety of subjects and site staff, while maintaining the integrity of the study.
- Update Section 5.2.3.2, Prohibited Therapy.

  \*Rationale: Revised Table 1 to update the list of examples of commonly used strong cytochrome 3A inducers.
- Update Section 5.3.1, Efficacy and Safety Measurements Assessed and Flow Chart

Rationale: Added clarifications on study activities that can be performed by phone/video conference or at local clinic/hospital/laboratory or through the optional home healthcare service in the event study visits are impacted by any state of emergency or pandemic situation like COVID-19 to ensure subjects' safety and study continuation, as permitted by IRB/IEC.

- Update Section 5.3.1.1, Study Procedures
  - Outcomes and Questionnaires
     Specified that questionnaires are not eligible for completion by virtual interview in the event that an onsite visit cannot be performed due to a pandemic or state of emergency and will be completed at the next earliest feasible visit.
  - O TB (tuberculosis) Testing/TB Prophylaxis and Chest X-rays (CXR) Specified that chest X-rays can be performed at the next earliest feasible visit unless the Investigator has determined that a CXR is required to ensure that it is safe to continue study drug administration (e.g., subjects



with seroconversion on an annual TB test). In this case, the Investigator should contact the AbbVie Therapeutic Area Medical Director (TA MD) to determine if the subject may continue on study drug and CXR should be performed as soon as restrictions allow at the study site or local hospital/facility.

# • 12-Lead Electrocardiogram (ECG)

Specified that the 12-Lead ECG can be performed at the next earliest feasible visit unless the Investigator has determined that an ECG is required to ensure that it is safe to continue study drug administration. In this case, the ECG should be performed as soon as restrictions allow at the study site or local hospital/facility.

o X-Rays of Hands and Feet

Added provision allowing the X-rays of hands and feet to be performed at the next earliest feasible visit.

# Physical Exam

Added provision allowing the complete physical exam to be performed at the next earliest feasible visit.

 Physician Global Assessment of Disease Activity Visual Analog Scale (VAS)

Specified that Physician Global Assessment of Disease Activity is not eligible for completion by virtual interview in the event that the subject cannot perform an onsite visit due to a pandemic or state of emergency and will be completed by the physician at the next earliest feasible subject's visit.

Tender Joint Count (TJC) and Swollen Joint Count (SJC) Assessments
 Added provision allowing the TJC and SJC to be performed at the next earliest feasible visit by the independent joint assessor, if possible.

# Pregnancy Test

Added provision allowing the urine pregnancy test to be performed at a local laboratory or at home. Updated the reference to contraception requirements for male subjects with a partner of childbearing potential for consistency with Section 5.2.4 "Contraception Recommendations."



# Clinical Laboratory Tests

Added provision allowing the laboratory testing at an alternate local facility, in the event that a state of emergency or pandemic prevents the subject from performing the central laboratory tests and added the requirements to allow the study drug dispensation when laboratory tests are performed at a local laboratory.

- Study Drug Dispensing, Dosing and Compliance
   Added provision allowing Direct-to-Patient (DTP) shipment of study drug and study ancillaries due to state of emergency or pandemic situations.
- New Section: Optional Home Healthcare Service Due to State of Emergency or Pandemic Situation like COVID-19
   Added home healthcare visits as an option in case a study visit on site cannot be performed due to state of emergency or pandemic-related reasons.

**Rationale:** To modify study visits and protocol-specific procedures impacted by the COVID-19 or any pandemic/state of emergency as necessary, to ensure the safety of subjects/site staff and study continuation including alternative locations for data collection, as permitted by IRB/IEC.

• Update Section 5.4.1, Discontinuation of Individual Subjects

**Rationale:** Revised to clarify that subjects will have to discontinue study drug treatment immediately if they develop a gastrointestinal perforation with the exception of appendicitis or mechanical injury to be consistent with the Section 6.1.7 "Toxicity Management."

Clarified that the state of emergency and pandemic-related restrictions may allow mitigation strategies to ensure subject safety and continuity of care as an alternative to study discontinuation/study drug discontinuation and that the AbbVie TA MD should be contacted before discontinuing a subject to ensure all acceptable mitigation steps have been explored.

• Update Section 5.5.1, Treatments Administered

**Rationale:** Added specifications in order to provide the study drug through DTP shipment in the event pandemic situation like COVID-19 or state of emergency prevent the study drug dispensation to the subject onsite, if permitted by local regulations.

- Update Section 6.1.1.3, Adverse Events of Special Interest *Rationale:* Clarified and updated the list of the adverse events of special interest according to the revised sponsor guidelines.
- Update Section 6.1.4, Adverse Event Collection Period

  Rationale: Added supplemental COVID-19 case report forms for missed or virtual visits, study drug interruptions or discontinuations, or adverse events and instructions to collect safety information related to COVID-19
- Update Section 6.1.5, Serious Adverse Event Reporting

  \*Rationale: Updated telephone number to contact the Immunology Safety

  Team for safety concerns.
- Update Section 6.1.6, Pregnancy

  \*Rationale: Updated text to define Pregnancy reporting timeline as 24 hours from site staff awareness according to the sponsor requirements.
- Update Section 6.1.7, Toxicity Management

  Rationale: Added guidance for investigators on the management of subjects

  with suspected or confirmed COVID-19 infection during the study. Clarified

  that the Investigator should also contact the AbbVie TA MD for confirmed ALT

  or AST > 8 × ULN in addition to the immediate study drug interruption.
- Update Section 6.2.2, Reporting

  \*Rationale: Updated text to define Product Complaint reporting timeline as 24 hours from site staff awareness according to the sponsor requirements.
- Update Section 7.0, Protocol Deviations.
   Rationale: Added language to include provision for modifications due to protocol deviations that may be due to pandemic like COVID-19 or state of emergency situations in order to guide investigators to notify IRB/EC when deviations occur.
- Update Section 9.2, Ethical Conduct of the Study
   Rationale: Inclusion of information regarding COVID-19 or any pandemic/state of emergency-related acceptable protocol modifications.
- Update Section 9.3, Subject Information and Consent



**Rationale:** Added provision that in the event of a pandemic situation or state of emergency, verbal consent may be obtained in addition to the study informed consent in accordance with local regulations.

• Update Section 10.1 Source Documents

**Rationale:** Noted that remote monitoring may be employed as needed, due to COVID-19 or any pandemic/state of emergency.

- Update Appendix A, Responsibilities of the Clinical Investigator
   Rationale: Clarified that clinical research studies sponsored by AbbVie are subject to the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) Good Clinical Practices (GCP).
- Update Appendix B, List of Protocol Signatories.

Rationale: Updated list of current Protocol Signatories.



# 1.2 Synopsis

| AbbVie Inc. | Protocol Number: M13-545 |
|---|---|
| Name of Study Drug: Upadacitinib (ABT-494) | Phase of Development: 3 |
| Name of Active Ingredient: Upadacitinib (ABT-494) | Date of Protocol Synopsis: 03 December 2020 |

**Protocol Title:** A Phase 3, Randomized, Double-Blind Study Comparing Upadacitinib (ABT-494) Once Daily Monotherapy to Methotrexate (MTX) Monotherapy in MTX-Naïve Subjects with Moderately to Severely Active Rheumatoid Arthritis

# **Objectives:**

#### Period 1

- 1. To compare the safety and efficacy of upadacitinib 7.5 mg once daily (QD) monotherapy (for subjects in Japan only), 15 mg QD monotherapy, and 30 mg QD monotherapy versus weekly methotrexate (MTX) monotherapy for the treatment of signs and symptoms of rheumatoid arthritis (RA) in MTX-naïve subjects with moderately to severely active RA.
- 2. To compare the efficacy of upadacitinib 15 mg QD monotherapy and upadacitinib 30 mg QD monotherapy versus weekly MTX monotherapy for prevention of structural progression in MTX-naive subjects with moderately to severely active RA.

#### Period 2

To evaluate the long-term safety, tolerability, and efficacy of upadacitinib 7.5 mg QD (for subjects in Japan only), 15 mg QD, and 30 mg QD in subjects with RA who have completed Period 1.

Investigators: Multicenter
Study Sites: Approximately 330

**Study Population:** Adult female and male subjects who are at least 18 years of age with a duration of symptoms consistent with RA for  $\geq 6$  weeks who also fulfill the 2010 ACR/European League Against Rheumatism (EULAR) classification criteria for RA and no prior or limited MTX treatment. Eligible study subjects must have  $\geq 6$  swollen joints (based on 66 joint counts) and  $\geq 6$  tender joints (based on 68 joint counts) at Screening and Baseline Visits, and high-sensitivity C-reactive protein (hsCRP)  $\geq 5$  mg/L (central lab, upper limit of normal [ULN] 2.87 mg/L) at Screening.

Number of Subjects to be Enrolled: Approximately 975 subjects

#### Methodology:

This is a Phase 3 multicenter study that includes two periods and a Japan sub-study. Period 1 is a 48-week randomized, double-blind, parallel-group, active comparator controlled treatment period designed to compare the safety and efficacy of upadacitinib 7.5 mg QD monotherapy (for subjects in Japan only), 15 mg QD monotherapy, and 30 mg QD monotherapy versus MTX monotherapy in adult MTX-naïve subjects with moderately to severely active RA. Period 1 is also designed to compare the efficacy of upadacitinib 15 mg QD monotherapy and 30 mg QD monotherapy versus MTX monotherapy for the prevention of structural progression. Period 2 is a long-term extension to evaluate the long-term safety, tolerability, and efficacy of upadacitinib (7.5, 15, or 30 mg QD) in subjects with RA who have completed Period 1.



# Methodology (Continued):

Starting with Amendment 6, subjects receiving upadacitinib 15 mg and 30 mg QD will receive open-label upadacitinib 15 mg QD. Subjects receiving MTX will receive open-label MTX.

The study duration will include a 35-day screening period, a 48-week randomized, double-blind, parallel-group, active-comparator controlled treatment period (Period 1); a 212-week extension period (blinded until the last subject completes the last visit of Period 1) (Period 2); and a 30-day follow-up (call or site visit).

Subjects will be randomized in a 1:1:1 ratio to treatment Groups 2, 3 and 4 below, except for subjects from Japan, who will be randomized in a 2:1:1:1 ratio to Groups 1, 2, 3 and 4:

- Group 1: Upadacitinib 7.5 mg QD monotherapy (subjects in Japan only; N = 75)
- Group 2: Upadacitinib 15 mg QD monotherapy (N = 300) (includes 37 subjects from Japan)
- Group 3: Upadacitinib 30 mg QD monotherapy (N = 300) (includes 37 subjects from Japan)
- Group 4: MTX monotherapy (N = 300) (includes 37 subjects from Japan)

Each subject will be instructed to take 2 capsules once weekly (MTX and/or matching placebo) and 1 tablet once daily (upadacitinib or matching placebo) to maintain blinding. MTX and matching placebo will be assigned via the Interactive Response Technology (IRT) system, and distributed as identical capsules in blister packs, to provide the correct total dose for each individual subject and to maintain blinding during and after MTX titration (Period 1 and Period 2). Detailed dosing instructions can be found in the Subject Dosing Diary and Instructions. Starting with Amendment 6 subjects receiving MTX will receive open-label MTX tablets in quantities sufficient to cover their respective dose.

Subjects who are assigned to upadacitinib 7.5 mg QD, 15 mg QD, or 30 mg QD will start on their respective upadacitinib dose at Baseline. Subjects who are assigned to the MTX treatment group will start oral MTX treatment at 10 mg/week and will be titrated up to 20 mg/week (increase by 5 mg every 4 weeks), as tolerated, by Week 8 (minimum 15 mg/week final dose required, with documentation of intolerance of > 15 mg/week). (For subjects in Japan: start at 7.5 mg/week with titration up to 10 mg/week at Week 4 and to 15 mg/week, as tolerated, by Week 8; minimum of 7.5 mg/week for final dose is required, with documentation of intolerance of > 7.5 mg/week). After completion of MTX (or placebo) titration, a single dose reduction of study drug (by 5 mg of MTX) is allowed for safety reasons, up to Week 26, as long as the subject remains on  $\geq 15$  mg/week of MTX (or matching placebo) weekly (for subjects in Japan:  $\geq 7.5$  mg/week). In addition, all subjects should take a dietary supplement of oral folic acid (or equivalent) throughout study participation. Folic acid dosing and timing of regimen should be followed according to Investigator's discretion. Rescue therapy has been defined for Weeks 12 through 24, Week 26, and Weeks 36 through 40. Starting at the Week 48 Visit (after Week 48 assessments have been performed) and thereafter, initiation of or change in background RA medication(s), including corticosteroids, non-steroidal anti-inflammatory drugs (NSAIDs), acetaminophen/paracetamol, and csDMARDs (concomitant use of up to 2 csDMARDs except the combination of MTX and leflunomide) is allowed as per local label.

Rescue therapy for those subjects who meet the following criteria from Week 12 through Week 24 are as follows:

• Those who do not achieve ≥ 20% improvement in both TJC and SJC compared with baseline at two consecutive visits starting at Week 12 will continue on their blinded therapy and the Investigator should optimize (initiate or increase) background RA medications: NSAIDs, corticosteroids (oral ≤ 10 mg/day prednisone equivalent or prednisone equivalent ≤ 0.5 mg/kg/day for 3 consecutive days) and/or low-potency analgesics.



# Methodology (Continued):

Rescue therapy for those subjects who meet the following criteria at Week 26 are as follows:

- 1. Subjects who were originally randomized to MTX:
  - Those who do not achieve CR by CDAI:
    - o but achieve ≥ 20% improvement in both TJC and SJC compared with baseline will continue on blinded MTX and the Investigator should optimize (initiate or increase) background RA medications: NSAIDs, corticosteroids (oral ≤ 10 mg/day prednisone equivalent and up to 2 local injections), low-potency analgesics and csDMARDs (only 1 of the following: sulfasalazine, hydroxychloroquine or chloroquine) throughout the remainder of Period 1 and until the study is unblinded.
    - o and do not achieve ≥ 20% improvement in both TJC and SJC compared with baseline will be re-randomized in a 1:1 ratio to receive blinded upadacitinib 15 mg QD or upadacitinib 30 mg QD (for subjects in Japan: randomize 1:1:1 to receive upadacitinib 7.5 mg QD, 15 mg QD, or 30 mg QD) while continuing MTX treatment in a blinded manner and will remain on upadacitinib plus MTX throughout the remainder of Period 1 and until the study is unblinded.
  - Those who achieve Clinical Remission (CR) by clinical disease activity index (CDAI) (CDAI ≤ 2.8) at Week 26 will continue blinded treatment with MTX throughout the remainder of Period 1 and until the study is unblinded (the study is unblinded when all subjects have completed Period 1).
- 2. Subjects who were originally randomized to upadacitinib:
  - Those who do not achieve CR by CDAI:
    - but achieve ≥ 20% improvement in both TJC and SJC compared with baseline will continue on blinded upadacitinib and the Investigator should optimize (initiate or increase the dose) background RA medications: NSAIDs, corticosteroids (oral ≤ 10 mg/day prednisone equivalent and up to 2 local injections), low-potency analgesics and csDMARDs (only 1 of the following: sulfasalazine, hydroxychloroquine or chloroquine) throughout the remainder of Period 1 and until the study is unblinded.
    - o and do not achieve ≥ 20% improvement in both TJC and SJC compared with baseline will add MTX 10 mg/week (7.5 mg for Japan) to upadacitinib in a blinded manner and will remain on upadacitinib plus MTX 10 mg/week (7.5 mg for Japan) throughout the remainder of Period 1 and until the study is unblinded.
  - Those who achieve Clinical Remission (CR) by CDAI (CDAI ≤ 2.8) at Week 26 will continue blinded treatment with upadacitinib throughout the remainder of Period 1 and until the study is unblinded (the study is unblinded when all subjects have completed Period 1).



# Methodology (Continued):

Rescue therapy for those subjects who meet the following criteria from Week 36 through Week 40 are as follows:

• Starting at Week 36, those who do not achieve ≥ 20% improvement in both TJC and SJC compared with baseline at two consecutive visits will continue on their blinded therapy and the Investigator should optimize (initiate or increase) background RA medications: NSAIDs, corticosteroids (oral ≤ 10 mg/day prednisone equivalent or prednisone equivalent ≤ 0.5 mg/kg/day for 3 consecutive days, and up to 2 local injections), low-potency analgesics and csDMARDs (only 1 of the following: sulfasalazine, hydroxychloroquine or chloroquine)

An unblinded analysis will be conducted after all subjects have completed Week 24 for the purpose of regulatory submission. To maintain integrity of the trial and avoid introduction of bias, study sites and subjects will remain blinded for the duration of Period 1. Additional unblinded analyses may be conducted after the Week 24 analysis.

Each subject will undergo a maximum of 3 scheduled visits for x-ray examination of bilateral hands and feet during Period 1 (unless unscheduled repeat imaging is needed due to failure to meet the quality requirements) at Screening, Week 24, and Week 48/Premature Discontinuation. One additional x-ray examination of bilateral hands and feet may be needed depending on the time of premature study drug discontinuation for those subjects that continue the study.

Subjects who complete the Week 48 Visit (end of Period 1) will enter the long-term extension, Period 2 (212 weeks). Subjects will continue study treatment per assignment at the end of Period 1 in a blinded fashion. When the last subject completes the last visit of Period 1 (Week 48), study drug assignment in both periods may be unblinded to the Sponsor and sites, and subjects would then be dispensed study drug in an open-label fashion until the completion of Period 2. All subjects will continue study treatment to which they were assigned at the time of study unblinding. Dose changes of open-label study drugs are not permitted during unblinded Period 2. Background therapies may be adjusted as per the discretion of the investigator (refer to Section 5.2.3.1 for additional details on permitted background therapy in Period 2).

Each subject will undergo a maximum of 3 scheduled visits for x-ray examination of bilateral hands and feet during Period 2 (unless unscheduled repeat imaging is needed due to failure to meet the quality requirements) at Week 96, Week 192, and Week 260. Subjects who prematurely discontinue from Period 2 will undergo an x-ray of hands and feet unless the previous x-ray was performed within the previous 24 weeks.

Starting with Amendment 6, subjects receiving upadacitinib 15 mg and 30 mg QD will receive open-label upadacitinib 15 mg QD. Subjects receiving MTX will receive open-label MTX.

Study visits may be impacted by state of emergency or pandemic like COVID-19. If visits cannot be conducted onsite due to travel restrictions or other pandemic or state of emergency related reasons, virtual visits, visits at alternative locations, or changes in the visit frequency and timing of study procedures, among others may be performed. Every effort should be made to ensure the safety of subjects and site staff, while maintaining the integrity of the study.



# Diagnosis and Main Criteria for Inclusion/Exclusion:

#### **Main Inclusion:**

- 1. Adult male or female, at least 18 years old.
- 2. Duration of symptoms consistent with RA for ≥ 6 weeks who also fulfill the 2010 ACR/EULAR classification criteria for RA.
- 3. Naïve to MTX or, if already on MTX, have received no more than 3 weekly MTX doses with requirement to complete a 4-week MTX washout before the first dose of study drug.
- 4. Subjects with prior exposure to csDMARDs other than MTX may be enrolled if completed the washout period as specified below or should be at least five times the mean terminal elimination half-life of a drug:
  - ≥ 4 weeks prior to first dose of study drug for minocycline, penicillamine, sulfasalazine, hydroxychloroquine, chloroquine, azathioprine, gold formulations, cyclophosphamide, tacrolimus, cyclosporine, mycophenolate;
  - ≥ 8 weeks prior to first dose of study drug for leflunomide if no elimination procedure was followed, or adheres to an elimination procedure (i.e., 11 days with colestyramine, or 30 days washout with activated charcoal or as per local label).
- 5. Subject meets both of the following disease activity criteria:
  - a.  $\geq 6$  swollen joints (based on 66 joint counts) and  $\geq 6$  tender joints (based on 68 joint counts) at Screening and Baseline Visits; and
  - b.  $hsCRP \ge 5 \text{ mg/L}$  (central lab, ULN 2.87 mg/L) at Screening Visit.
- 6. ≥ 1 bone erosion on x-ray (by local reading) OR in the absence of a documented bone erosion, both positive rheumatoid factor and positive anti-cyclic citrullinated peptide autoantibodies are required at Screening.

# **Main Exclusion:**

- 1. Intolerant to MTX.
- 2. Prior exposure to any JAK inhibitor (including but not limited to tofacitinib, baricitinib, and filgotinib).
- 3. Prior exposure to any bDMARD(s).
- 4. History of any arthritis with onset prior to age 17 years or current diagnosis, inflammatory joint disease other than RA (including but not limited to gout, systemic lupus erythematosus, psoriatic arthritis, axial spondyloarthritis including ankylosing spondylitis and non-radiographic axial SpA, reactive arthritis, overlap connective tissue diseases, scleroderma, polymyositis, dermatomyositis, fibromyalgia [currently with active symptoms]. Current diagnosis of secondary Sjogren's Syndrome is permitted.
- 5. Laboratory values meeting the following criteria within the Screening period prior to the first dose of study drug: serum aspartate transaminase > 2 × ULN; serum alanine transaminase > 2 × ULN; estimated glomerular filtration rate by simplified 4-variable Modification of Diet in Renal Disease formula < 40 mL/min/1.73 m²; total white blood cell count < 2,500/ $\mu$ L; absolute neutrophil count < 1,500/ $\mu$ L; platelet count < 100,000/ $\mu$ L; absolute lymphocyte count < 800/ $\mu$ L; and hemoglobin < 10 g/dL.



**Investigational Product:** Upadacitinib (ABT-494)

**Doses:** 30 mg QD

15 mg QD

7.5 mg QD (for Japan only)

**Mode of Administration:** Oral

**Reference Therapy:** MTX, matching placebo for upadacitinib, matching placebo for MTX

**Dose:** MTX 10 mg/week titrated up to 20 mg/week given as a single dose

every week. For subjects in Japan, MTX 7.5 mg/week titrated up to

15 mg/week given as a single dose every week.

**Mode of Administration:** Oral

**Duration of Treatment:** up to 260 weeks (Period 1: 48 weeks; Period 2: 212 weeks)

#### Criteria for Evaluation:

## Efficacy:

#### Period 1

The primary endpoint in Period 1 is the proportion of subjects achieving ACR50 response at Week 12 (US/FDA regulatory purposes) or the proportion of subjects achieving Clinical Remission (CR) (EU/EMA regulatory purposes) at Week 24. For Japan/PMDA regulatory purposes, the primary endpoints are the proportion of subjects achieving ACR20 response at Week 12 and change from baseline in modified Total Sharp Score (mTSS) at Week 24.

ACR20/50 response rate will be determined based on 20%/50% or greater improvement in TJC and SJC and ≥ 3 of the 5 measures of Patient's Assessment of Pain (Visual Analog Scale [VAS]), Patient's Global Assessment of Disease Activity (VAS), Physician's Global Assessment of Disease Activity (VAS), Health Assessment Questionnaire Disability Index (HAQ-DI), or hsCRP.

CR is defined as Disease Activity Score (DAS) 28 (C-reactive protein [CRP]) < 2.6.

Modified Total Sharp Score (mTSS) is the van der Heijde mTSS.



#### **Criteria for Evaluation (Continued):**

## **Efficacy (Continued):**

## Period 1 (Continued)

Ranked key secondary endpoints for US/FDA regulatory purposes are:

- 1. Change from baseline in DAS28 (CRP) at Week 12;
- 2. Change from baseline in HAQ-DI at Week 12;
- 3. Change from baseline in modified Total Sharp Score (mTSS) at Week 24;
- 4. Proportion of subjects achieving Low Disease Activity (LDA) based on DAS28 (CRP) ≤ 3.2 at Week 12;
- 5. Proportion of subjects achieving CR based on DAS28 (CRP) < 2.6 at Week 24;
- 6. Change from baseline in Short Form-36 (SF-36) Physical Component Score (PCS) at Week 12.

Ranked key secondary endpoints (at Week 24) for EU/EMA regulatory purposes are:

- 1. Change from baseline in DAS28 (CRP);
- 2. Change from baseline in HAQ-DI;
- 3. ACR50 response rate;
- 4. Change from baseline in modified Total Sharp Score (mTSS);
- 5. Proportion of subjects achieving LDA based on DAS28 (CRP)  $\leq$  3.2;
- 6. Change from baseline in SF-36 PCS;
- 7. Proportion of subjects with no radiographic progression (defined as change from baseline in mTSS ≤ 0) at Weeks 24.

Ranked key secondary endpoints for Japan/PMDA regulatory purposes are:

- 1. Change from baseline in DAS28 (CRP) at Week 12;
- 2. Change from baseline in HAQ-DI at Week 12;
- 3. Proportion of subjects achieving LDA based on DAS28 (CRP)  $\leq$  3.2 at Week 12;
- 4. Proportion of subjects achieving CR based on DAS28 (CRP) < 2.6 at Week 24;
- 5. Change from baseline in SF-36 PCS at Week 12.

Other key secondary endpoints for US/FDA regulatory purposes are:

- 1. ACR20 response rate at Week 12;
- 2. ACR70 response rate at Week 12;
- 3. Proportion of subjects with no radiographic progression at Week 24.

Other key secondary endpoints for EU/EMA regulatory purposes are:

- 1. ACR20 response rate at Week 24;
- 2. ACR70 response rate at Week 24.

Other key secondary endpoints for Japan/PMDA regulatory purposes are:

- 1. ACR50 response rate at Week 12;
- 2. ACR70 response rate at Week 12;
- 3. Proportion of subjects with no radiographic progression at Week 24.

# **Criteria for Evaluation (Continued):**

#### **Efficacy (Continued):**

# Period 1 (Continued)

# Additional endpoints are:

- ACR20/50/70 response rates at all visits;
- Change from baseline in individual components of ACR response at all visits;
- Change from baseline in DAS28(CRP) and DAS28 (erythrocyte sedimentation rate [ESR]) at all
  visits;
- Change from baseline in CDAI and SDAI at all visits;
- Proportion of subjects achieving LDA or CR by DAS28(CRP), DAS28(ESR), Simplified Disease Activity Index (SDAI), and Clinical Disease Activity Index (CDAI) at all visits;
- Change from baseline in morning stiffness (severity and duration) at all visits;
- Proportion of subjects with change from baseline in HAQ-DI  $\leq$  -0.22 at all visits;
- Proportion of subjects with change from baseline in HAQ-DI  $\leq$  -0.3 at all visits;
- ACR/EULAR Boolean remission at all visits;
- Change from baseline in EQ-5D-5L at Weeks 12, 24, and 48;
- Change from baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) at Weeks 12, 24, and 48;
- Change from baseline in Work Productivity and Activity Impairment (WPAI) at Weeks 12, 24, and 48;
- Change from baseline in SF-36 at Weeks 12, 24, and 48;
- Change from baseline in mTSS at Weeks 24 and 48;
- Proportion of subjects with no radiographic progression (defined as change from baseline in mTSS ≤ 0) at Weeks 24 and 48;
- Change from baseline in radiographic joint space narrowing and erosion scores at Weeks 24 and 48.

| | DAS28 (CRP) and<br>DAS28 (ESR) | SDAI | CDAI |
|-----|--------------------------------|--------|-------|
| LDA | ≤ 3.2 | ≤ 11.0 | ≤ 10 |
| CR | < 2.6 | ≤ 3.3 | ≤ 2.8 |



#### **Criteria for Evaluation (Continued):**

#### **Efficacy (Continued):**

#### Period 2

Assessments to evaluate efficacy of treatment in Period 2 will be analyzed for the following measures at Weeks 60, 72, 84, 96, every 12 weeks through Week 240, and Week 260/PD:

- ACR20/50/70 response rates;
- Change from baseline in individual ACR components;
- Change from baseline in DAS28 (CRP);
- Change from baseline in DAS28 (ESR);
- Change from baseline in CDAI and SDAI;
- Proportion of subjects achieving LDA and proportion of subjects achieving CR based on DAS28 (CRP), DAS28 (ESR), SDAI, and CDAI criteria (as defined for Period 1);
- Change from baseline in morning stiffness (severity and duration);
- Proportion of subjects with change from baseline in HAQ-DI  $\leq$  -0.22;
- Proportion of subjects with change from baseline in HAQ-DI  $\leq -0.3$ ;
- ACR/EULAR Boolean remission at all visits
- Concomitant corticosteroid use.

Additionally, assessment for the evaluation of radiographic changes in Period 2 will occur at Week 96 and every 96 weeks thereafter (or Premature Discontinuation Visit):

- Change from baseline in mTSS;
- Proportion of subjects with no radiographic progression (defined as change from baseline mTSS of ≤ 0);
- Change from baseline in radiographic joint space narrowing and erosion scores.

#### Pharmacokinetic (Period 1 Only):

Blood samples for assay of upadacitinib and possibly other medications in plasma will be collected at Weeks 2, 4, 12, 16, 20, 24, 32, 36, 40, and 48/Premature Discontinuation.

#### Exploratory Research Variables and Validation Studies (Optional) (Period 1 Only):

Prognostic, predictive, and pharmacodynamics biomarkers signatures may be evaluated. Samples for pharmacogenetic, epigenetic, transcriptomic, and proteomic and targeted protein investigations will be collected at various time points. Assessments will include but may not be limited to nucleic acids, proteins, metabolites, or lipids.

# Safety:

Safety evaluations include adverse event (AE) monitoring, physical examinations, vital sign measurements, electrocardiogram (ECG), and clinical laboratory testing (hematology, chemistry, and urinalysis) as a measure of safety and tolerability for the entire study duration.



# **Statistical Methods:**

#### **Efficacy:**

All efficacy analyses will be carried out using the Full Analysis Set population, which includes all randomized subjects who receive at least one dose of study drug.

# Period 1 Efficacy

# Analysis of the Primary and Key Secondary Endpoints:

For the global analysis, comparisons of the primary and key secondary efficacy endpoints will be made between the upadacitinib 15 mg QD and 30 mg QD groups versus the MTX group for all subjects (excluding the Japan specific upadacitinib 7.5 mg treatment arm). The overall type I error rate of the primary and key secondary endpoints for the two doses will be strongly controlled.

For the Japan sub-study, comparisons of the primary and key secondary efficacy endpoints will be made between the upadacitinib 7.5 mg QD, 15 mg QD and 30 mg QD groups versus the MTX group for subjects enrolled in Japan only.

For binary endpoints, frequencies and percentages will be reported for each treatment group. Pairwise comparisons between each upadacitinib group and the MTX group will be conducted using the Cochran-Mantel-Haenszel test adjusting for main stratification factors.

For continuous endpoints, the mean, standard deviation, median, and range will be reported for each treatment group. Pairwise comparisons between each of the upadacitinib treatment groups and the MTX group will be carried out using the analysis of covariance model with treatment group as the fixed factor, and the corresponding baseline value and the main stratification factors as the covariates.

For mTSS-based endpoints, both linear extrapolation and as observed analysis will be conducted. For other endpoints, non-responder imputation approach will serve as the primary analysis approach for key binary endpoints and multiple imputations will serve as the primary analysis approach for key continuous endpoints. Sensitivity analyses based on observed cases will also be conducted for key endpoints.

# Long-Term Efficacy for Period 1 and Period 2 Combined:

Long-term efficacy by time point will be summarized using descriptive statistics.

#### Pharmacokinetic:

A non-linear mixed-effects modeling approach will be used to estimate the population central values and the empirical Bayesian estimates of the individual values of upadacitinib oral clearance (CL/F) and volume of distribution (V/F). Additional parameters may be estimated if useful in the interpretation of the data.

#### Safety:

Safety analyses will be carried out using the Safety Analysis Set, which includes all subjects who receive at least one dose of study drug. Analyses will be conducted for Period 1 alone, as well as for Period 1 and Period 2 combined. Safety will be assessed by AEs, physical examination, laboratory assessments, ECG, and vital signs. Frequency tables and lists of subjects with treatment-emergent AEs by preferred term as in the Medical Dictionary for Regulatory Activities dictionary, by system organ class, by severity, and by relationship to the study drug as assessed by the Investigator will be provided. The changes from baseline in vital signs, physical examination results, and clinical laboratory values will be analyzed in a descriptive manner. Shift of laboratory values from baseline to defined time points will be tabulated.



# 1.3 List of Abbreviations and Definition of Terms

# **Abbreviations**

ACR American College of Rheumatology

AE adverse event

ALC absolute lymphocyte count
ALT alanine transaminase
ANC absolute neutrophil count
anti-CCP anti-cyclic citrullinated peptide

AP anteroposterior

AST aspartate transaminase

AUC Area under the plasma concentration-time curve

BCG Bacille Calmette-Guérin

bDMARD biologic disease-modifying anti-rheumatic drug

BID twice daily (Latin: bis in die)

BUN blood urea nitrogen
CBC complete blood count
CD4, CD8 cluster of differentiation
CDAI clinical disease activity index

CL/F apparent clearance

C<sub>max</sub> Maximum Observed Plasma Concentration

CPK creatine phosphokinase
COVID-19 Coronavirus Disease – 2019

CR clinical remission
CRF case report form
CRP C-reactive protein

csDMARD conventional synthetic disease-modifying anti-rheumatic drug

CSR clinical study report

CXR chest x-ray

CYP3A cytochrome P450 3A
DAS disease activity score

DMARD disease-modifying anti-rheumatic drug

DMC Data Monitoring Committee

DNA Deoxyribonucleic acid



M13-545 Protocol Amendment 8 EudraCT 2015-003334-27

DTP Direct-to-Patient ECG electrocardiogram

eCRF electronic case report form EDC electronic data capture

EDTA Edetic acid (ethylenediaminetetraacetic acid)

ePRO electronic patient-reported outcome

EQ-5D-5L EuroQoL-5D-5L

ESR erythrocyte sedimentation rate

EU European Union

EULAR European League Against Rheumatism

FACIT-F Functional Assessment of Chronic Illness Therapy - Fatigue

FAS full analysis set

FSH follicle stimulating hormone
GCP Good Clinical Practice
GFR glomerular filtration rate

HAQ-DI Health Assessment Questionnaire – Disability Index

HBc Ab/anti-HBc Hepatitis B core antibody
HBs Ab/anti-HBs Hepatitis B surface antibody
HBs Ag Hepatitis B surface antigen

HBV Hepatitis B virus
HCV Hepatitis C virus

HCV Ab Hepatitis C virus antibody

HDL-C high-density lipoprotein cholesterol
HIV human immunodeficiency virus
hsCRP high-sensitivity C-reactive protein

IAG Imaging Acquisition Guide ICF informed consent form

ICH International Conference on Harmonization

IEC independent ethics committee
IGRA interferon-gamma release assay
IMP investigational medicinal product
INR international normalized ratio

IR inadequate responder
IRB institutional review board



M13-545 Protocol Amendment 8 EudraCT 2015-003334-27

IRT interactive response technology

IUD intrauterine device

IUS intrauterine hormone-releasing system

JAK Janus kinase

LDA low disease activity

LDL-C low-density lipoprotein cholesterol
MACE major adverse cardiovascular event
MDRD modification of diet in renal disease

MedDRA Medical Dictionary for Regulatory Activities

mTSS modified total sharp score

MTX methotrexate

MTX-IR methotrexate inadequate responder

NA no assessment

NMSC non-melanoma skin cancer

NONMEM non-linear mixed-effects modeling

NRI non-responder imputation
NRS numerical rating scale

NSAID non-steroidal anti-inflammatory drug

OC observed cases

OLE open-label extension
PA posterior-anterior

PCR polymerase chain reaction
PCS physical component summary
PD premature discontinuation

PhGA Physician's Global Assessment of Disease Activity

PK pharmacokinetic

PPD purified protein derivative
PRN as needed (Latin: pro re nata)
PRO patient-reported outcome

PT preferred term

PtGA Patient's Global Assessment of Disease Activity

QD once daily (Latin: quaque die)

RA rheumatoid arthritis

RAVE® EDC system from Medidata



M13-545 Protocol Amendment 8 EudraCT 2015-003334-27

RBC red blood cell

RCT randomized controlled trial

RF rheumatoid factor
RNA Ribonucleic acid
SAE serious adverse event
SAP statistical analysis plan
SDAI simple disease activity index

SF-36 Short Form-36
SJC swollen joint count
SOC system organ class

SUSAR suspected unexpected serious adverse reaction

T2T treat-to-target TB tuberculosis

TEAE treatment-emergent adverse event

TJC tender joint count
TNF tumor necrosis factor

TNF-IR anti-tumor necrosis factor inadequate responder

TSJ tender and swollen joints

Tyk2 Tyrosine kinase 2
ULN upper limit of normal

V/F apparent volume of distribution

VAS visual analog scale

VTE venous thromboembolic events

VZV Varicella zoster virus WBC white blood cell

WPAI Work Productivity and Activity Impairment

#### 2.0 **Table of Contents** 1.0 Title Page......1 Protocol Amendment: Summary of Changes ......2 1.1 1.2 Synopsis .......8 1.3 2.0 3.0 3.1 Differences Statement......31 Benefits and Risks......32 3.2 **Study Objectives ......32** 4.0 5.0 Investigational Plan......33 5.1 5.2 5.2.1 5.2.2 5.2.3 Prior, Concomitant, and Prohibited Therapy ......50 5.2.3.1 Permitted Background RA Therapy.....50 Prohibited Therapy......52 5.2.3.2 5.2.3.3 Rescue Therapy......56 5.2.4 Contraception Recommendations .......58 5.3 Efficacy Pharmacokinetic, Pharmacodynamic, Exploratory Research and Validation Studies, and Safety 5.3.1 Study Procedures ......64 5.3.1.1 Collection and Handling of Optional Samples for Exploratory 5.3.1.2 5.3.2 5.3.2.1 Collection of Samples for Analysis ......92 5.3.2.2 Measurement Methods......93 5.3.3 Efficacy Variables.....93 5.3.3.1 Period 1 Variables 93



| 5.3.3.1.1 | Primary Variables93 |
|-----------|---------------------------------------------------------|
| 5.3.3.1.2 | Key Secondary Variables94 |
| 5.3.3.1.3 | Additional Variables96 |
| 5.3.3.2 | Period 2 Variables |
| 5.3.4 | Safety Variables98 |
| 5.3.5 | Pharmacokinetic Variables |
| 5.3.6 | Exploratory Research Variables and Validation Studies98 |
| 5.4 | Removal of Subjects from Therapy or Assessment99 |
| 5.4.1 | Discontinuation of Individual Subjects |
| 5.4.2 | Discontinuation of Entire Study |
| 5.5 | Treatments |
| 5.5.1 | Treatments Administered |
| 5.5.2 | Identity of Investigational Product |
| 5.5.2.1 | Packaging and Labeling |
| 5.5.2.2 | Storage and Disposition of Study Drugs |
| 5.5.3 | Method of Assigning Subjects to Treatment Groups104 |
| 5.5.4 | Selection and Timing of Dose for Each Subject |
| 5.5.5 | Blinding |
| 5.5.5.1 | Blinding of Investigational Product |
| 5.5.5.2 | Blinding of Data for Data Monitoring Committee |
| 5.5.6 | Treatment Compliance |
| 5.5.7 | Drug Accountability |
| 5.6 | Discussion and Justification of Study Design |
| 5.6.1 | Discussion of Study Design and Choice of Control Groups |
| 5.6.2 | Appropriateness of Measurements |
| 5.6.3 | Suitability of Subject Population |
| 5.6.4 | Selection of Doses in the Study |
| 6.0 | Complaints112 |
| 6.1 | Medical Complaints |
| 6.1.1 | Definitions |
| 6.1.1.1 | Adverse Event |
| 6.1.1.2 | Serious Adverse Events |
| 6.1.1.3 | Adverse Events of Special Interest |



| W113-343 | Protocol Amendment |
|----------|--------------------|
| EudraCT | 2015-003334-27 |

| 6.1.2 | Adverse Event Severity |
|---|---|
| 6.1.3 | Relationship to Study Drug |
| 6.1.4 | Adverse Event Collection Period |
| 6.1.5 | Serious Adverse Event Reporting |
| 6.1.6 | Pregnancy |
| 6.1.7 | Toxicity Management |
| 6.1.8 | Data Monitoring Committee |
| 6.1.9 | Cardiovascular Adjudication Committee |
| 6.2 | Product Complaint |
| 6.2.1 | Definition |
| 6.2.2 | Reporting127 |
| 7.0 | Protocol Deviations127 |
| 8.0 | Statistical Methods and Determination of Sample |
| | Size129 |
| 8.1 | Statistical and Analytical Plans |
| 8.1.1 | Analysis Populations 129 |
| 8.1.1.1 | Full Analysis Set |
| 8.1.1.2 | Per Protocol Analysis Set |
| 8.1.1.3 | Safety Analysis Set |
| 8.1.2 | Subject Accountability, Disposition and Study Drug Exposure |
| 8.1.2.1 | Subject Accountability |
| 8.1.2.2 | Subject Disposition |
| 8.1.2.3 | Study Drug Exposure |
| 8.1.3 | Analysis of Demographic and Baseline Characteristics |
| 8.1.4 | Efficacy Analysis |
| 8.1.4.1 | Efficacy Analysis for Period 1 |
| 8.1.4.1.1 | Primary Efficacy Variables |
| 8.1.4.1.2 | Key Secondary Efficacy Variables |
| 8.1.4.1.3 | Other Efficacy Variables |
| 8.1.4.1.4 | Multiplicity Control for the Primary and Ranked Key Secondary Endpoints |
| 8.1.4.1.5 | Imputation Methods |
| 8.1.4.2 | Long-Term Efficacy for Period 1 and Period 2 Combined |
| | ~ |

# Upadacitinib M13-545 Protocol Amendment 8 EudraCT 2015-003334-27

| 8.1.5 | Safety Analysis | 135 |
|---|---|---|
| 8.1.5.1 | General Considerations | 135 |
| 8.1.5.2 | Analysis of Adverse Events | 135 |
| 8.1.5.2.1 | Treatment-Emergent Adverse Events (TEAE) | 135 |
| 8.1.5.2.2 | Serious Adverse Events and Death | 137 |
| 8.1.5.3 | Analysis of Laboratory, Vital Sign, and ECG Data | 137 |
| 8.1.6 | Pharmacokinetic and Exposure-Response Analyses | 137 |
| 8.2 | Determination of Sample Size | 139 |
| 8.3 | Randomization Methods | 140 |
| 9.0 | Ethics | 140 |
| 9.1 | Independent Ethics Committee (IEC) or Institutional Review Board (IRB) | 140 |
| 9.2 | Ethical Conduct of the Study | 141 |
| 9.3 | Subject Information and Consent | 142 |
| 9.3.1 | Informed Consent Form and Explanatory Material | 143 |
| 9.3.2 | Revision of the Consent Form and Explanatory Material | 143 |
| 10.0 | Source Documents and Case Report Form | |
| | Completion | 143 |
| 10.1 | Source Documents | 143 |
| 10.2 | Case Report Forms | 144 |
| 11.0 | Data Quality Assurance | 147 |
| 12.0 | Use of Information | 147 |
| 13.0 | Completion of the Study | 148 |
| 14.0 | Investigator's Agreement | 149 |
| 15.0 | Reference List | 150 |
| List of Ta | ables | |
| Table 1. | Examples of Commonly Used Strong CYP3A Inhibitors and Inducers | 54 |
| Table 2. | Clinical Laboratory Tests | 83 |
| Table 3. | Identity of Investigational Product | 103 |



Upadacitinib
M13-545 Protocol Amendment 8
EudraCT 2015-003334-27

| Table 4. | Specific Toxicity Management Guidelines for Abnormal Laboratory Values | 123 |
|---|---|---|
| List of Fig | ures | |
| Figure 1. | Period 1 Study Design | 39 |
| Figure 2. | Period 2 Study Design | |
| Figure 3. | Handling of X-Rays of Hands and Feet after Baseline (Period 1) | 76 |
| Figure 4. | Criteria for HBV DNA PCR Qualitative Testing | 86 |
| Figure 5. | Adverse Event Collection | 117 |
| List of App | pendices | |
| Appendix A. | Responsibilities of the Clinical Investigator | 153 |
| Appendix B. | List of Protocol Signatories | 155 |
| Appendix C. | Local Requirements | 156 |
| Appendix D. | Study Activities (Period 1) | 162 |
| Appendix E. | Study Activities – Optional Samples for Exploratory Research and Validation Studies (Period 1 Only) | 168 |
| Appendix F. | Study Activities (Period 2) | |
| Appendix G. | Physician's Global Assessment of Disease Activity Example | |
| Appendix H. | Joint Evaluation Worksheet Example | |
| Appendix I. | Latent TB Risk Assessment Form Example | |
| Appendix J. | Patient's Global Assessment of Disease Activity Example | |
| Appendix K. | Patient's Assessment of Pain Example | |
| Appendix L. | Health Assessment Questionnaire (HAQ-DI) Example | 178 |
| Appendix M. | Patient's Assessment of Severity and Duration of Morning Stiffness Example | |
| Appendix N. | EuroQoL-5D Example | |
| Appendix O. | Functional Assessment of Chronic Illness Therapy – Fatigue (FACIT-F) Scale Example | |
| Appendix P. | Work Productivity and Activity Impairment Questionnaire:<br>Specific Health Problem (WPAI:SHP) Questionnaire Example | |



Upadacitinib
M13-545 Protocol Amendment 8
EudraCT 2015-003334-27

| Appendix Q. | Short Form-36 (SF-36 <sup>TM</sup> ) Health Status Survey Questionnaire | |
|---|---|---|
| | Example | 189 |
| Appendix R. | Rheumatology Common Toxicity Criteria v.2.0 Example | 195 |



# 3.0 Introduction

# **Rheumatoid Arthritis**

Rheumatoid arthritis (RA) is a chronic systemic inflammatory disease of unknown etiology. The hallmark feature of RA is an inflammatory process manifested by persistent symmetric polyarthritis of synovial joints which can ultimately lead to bone erosions, deformity, and disability. Left untreated, or inadequately treated, progressive functional impairment with increasing disability occurs leading to a reduction in quality of life. The prevalence of RA in the general population is approximately 1%, and increases with age in both genders, with women being more prone to developing RA than men. Early therapy with disease-modifying anti-rheumatic drugs (DMARDs) is the standard of care, including conventional synthetic DMARDs (csDMARDs) (e.g., methotrexate [MTX], sulfasalazine, hydroxychloroquine, and leflunomide), and biologic DMARDs (bDMARDs) (e.g., anti-tumor necrosis factor [TNF] and non-anti-TNF biologics).

The European League Against Rheumatism (EULAR) recommends a Treat-to-Target (T2T) approach to initiate therapy immediately after diagnosis of RA with a goal of achieving clinical remission (CR) or low disease activity (LDA), as these are associated with improved long-term outcomes. Also, in line with recent advances in early diagnosis, new classification criteria have been developed. The 2010 American College of Rheumatology (ACR)/EULAR classification criteria redefined the paradigm of RA by focusing on features at earlier stages of disease that are associated with persistent and/or erosive disease, rather than defining the disease by its late-stage features.

Despite major progress in the treatment of RA, there still remains a large unmet medical need, as only a small percentage of RA patients reach or maintain a status of LDA or CR over time or need to discontinue due to safety or tolerability issues. <sup>5,6</sup> Novel therapies are therefore needed to complement the available interventions to address the unmet need. <sup>5-7</sup>



# **JAK Inhibitor**

Evidence suggests that inhibition of Janus kinase (JAK)-mediated pathways is a promising approach for the treatment of patients with this chronic disease. AbbVie is developing a small molecule inhibitor of JAK, upadacitinib (ABT-494), that may address the current needs.

The JAK family is composed of 4 family members: JAK1, 2, 3, and Tyrosine kinase 2 (Tyk2). These cytoplasmic tyrosine kinases are associated with membrane cytokine receptors such as common gamma-chain receptors and the glycoprotein 130 transmembrane proteins. Activation of JAK pathways initiates expression of survival factors, cytokines, chemokines, and other molecules that facilitate leukocyte cellular trafficking and cell proliferation which contribute to inflammatory and autoimmune disorders.

Hence, the JAK family has evoked considerable interest in the area of inflammatory diseases leading to the development of various JAK inhibitors with different selectivity profiles against JAK1, JAK2, JAK3, and Tyk2 which have demonstrated efficacy in individuals with RA. <sup>10-14</sup> Tofacitinib, the first in this class, has been approved in the United States and in other countries for treating moderately to severely active RA patients. Although tofacitinib, a non-selective JAK inhibitor, improves the clinical signs and symptoms, and inhibits structural progression in RA patients, questions regarding the safety profile remain, including serious infections, herpes zoster reactivation, malignancies, and hematologic adverse events (AEs).

The second generation of JAK inhibitors, with different selectivity profiles against JAK1, JAK2, JAK3, and Tyk2, are in development. Upadacitinib is a novel selective JAK1 inhibitor being developed for the treatment of adult patients with moderately to severely active RA. In an in vitro setting, upadacitinib potently inhibits JAK1 activity, but to a lesser degree, inhibits the other isoforms, JAK2 and JAK3. The enhanced selectivity of upadacitinib against JAK1 may offer an improved benefit-risk profile in patients with RA. The clinical hypothesis is that upadacitinib should be effective in decreasing joint



inflammation and damage associated with RA by interfering with JAK1-mediated signaling pathways (i.e., interleukin-6) without causing excessive anemia due to its reduced activity against JAK2 (IC<sub>50</sub> 120 nM), which is essential for erythropoietin signaling. Upadacitinib is also less potent against JAK3 (IC<sub>50</sub> 2.3 μM), an important component of lymphocyte activation and function. As such, treatment with upadacitinib, a selective JAK1 inhibitor with reduced JAK3 inhibition, could result in a decreased risk for infection (including viral reactivation) and/or malignancy compared to a pan JAK inhibitor or less selective JAK inhibitors.

# **Phase 2 Studies with Upadacitinib**

The Phase 2 program for upadacitinib consisted of 2 randomized controlled trials (RCTs), both on stable background MTX therapy, in subjects with moderately to severely active RA and one open-label extension (OLE) study (Study M13-538; NCT02049138) for those subjects who had completed either one of the RCTs. Study M13-550 (NCT01960855) enrolled subjects who had an inadequate response to anti-TNF therapy and Study M13-537 (NCT02066389) enrolled subjects who had shown an inadequate response to MTX. A total of 4 twice daily (BID) and 1 once daily (QD) dose regimens of upadacitinib immediate release capsules (3 mg BID, 6 mg BID, 12 mg BID, 18 mg BID, and 24 mg QD) were evaluated.

In TNF-inadequate responder (TNF-IR) subjects, who represent the population with the greatest unmet need, the primary endpoint of ACR20 response rate at Week 12 was significantly greater at all doses of upadacitinib (up to 73%) compared with placebo (35%). In addition, numerically higher proportions of subjects achieved ACR50 and ACR70 responses and LDA (based on Disease Activity Score [DAS]28 C-Reactive Protein [CRP] and Clinical Disease Activity Index [CDAI]) in the upadacitinib dose groups versus placebo.

In MTX-inadequate responder (MTX-IR) subjects, the primary endpoint of ACR20 response rate at Week 12 was significantly greater (up to 82%) at all but the lowest dose



of upadacitinib compared with placebo (50%). At all doses of upadacitinib compared to placebo, significantly higher proportions of subjects achieved LDA and CR at Week 12.

Safety data from these two studies (N = 575) showed that the types and frequencies of AEs during upadacitinib treatment were consistent with subjects with moderately to severely active RA receiving immunomodulatory therapy. The incidences of AEs were numerically higher in the upadacitinib dose groups, with a trend toward higher rates with higher doses of upadacitinib. The most frequently reported AEs ( $\geq 5\%$ ) in the upadacitinib treated subjects were urinary tract infection, headache, upper respiratory tract infection, and nausea. There were 6 subjects (1.3% of total combined populations) with herpes zoster reactivation distributed across the upadacitinib dose groups, and 2 subjects (1.9%) in the placebo groups. In these two 12 week studies, a total of 2 subjects in the upadacitinib treatment groups reported malignancies. One subject reported nonmelanoma skin cancers (NMSC) (basal cell and squamous cell carcinoma) and 1 subject was diagnosed with lung cancer after the final scheduled visit, and subsequently died 14 weeks after study completion. These events were reported by the Investigators as not possibly related to study drug. Elevations of liver function tests were sporadic with no clear dose-response relationship observed. As observed with other JAK inhibitors, treatment with upadacitinib resulted in an increase in lipids (low-density lipoprotein cholesterol [LDL-C] and high-density lipoprotein cholesterol [HDL-C]). Among subjects with laboratory evidence of systemic inflammation (as evidenced by high-sensitivity C-reactive protein [hsCRP] > upper limit of normal [ULN]), treatment with lower doses of upadacitinib (3 mg BID and 6 mg BID) was associated with improvements in mean hemoglobin relative to placebo. At higher doses, there was a reduction in mean hemoglobin; however, the mean hemoglobin levels remained within normal range throughout the treatment period.

# 3.1 Differences Statement

Study M13-545 differs from other upadacitinib studies as it is the first study to evaluate the safety and efficacy (clinical and structural) of upadacitinib in subjects diagnosed with active RA who are naïve to MTX therapy.



# 3.2 Benefits and Risks

Despite the availability of various RA therapies, including csDMARDs and bDMARDs, many patients still do not respond adequately to these treatments, or gradually lose response over time. Upadacitinib is a novel selective JAK1 inhibitor with the ability to decrease joint inflammation and damage mediated by JAK1 signaling while having minimal inhibitory effects on JAK2 and JAK3. This could potentially minimize some of the reported safety concerns with non-selective JAK inhibition which are thought to be mediated by inhibition of JAK2 and JAK3 signaling pathways. The Phase 2 program with upadacitinib demonstrated efficacy for improvement in signs and symptoms of RA and the safety results were consistent with those known to be associated with JAK inhibition. Taken together, the safety and efficacy data from the Phase 2 program support further development of upadacitinib in Phase 3 in subjects with RA.

In view of the COVID-19 pandemic, the benefit:risk profile of various immunomodulatory therapies on COVID-19 is being evaluated. At this time, the effects of upadacitinib on the course of COVID-19 are not well defined.

# 4.0 Study Objectives

# Period 1

- 1. To compare the safety and efficacy of upadacitinib 7.5 mg QD monotherapy (for subjects in Japan only), 15 mg QD monotherapy, and 30 mg QD monotherapy versus weekly MTX monotherapy for the treatment of signs and symptoms of RA in MTX-naïve subjects with moderately to severely active RA.
- 2. To compare the efficacy of upadacitinib 15 mg QD monotherapy and upadacitinib 30 mg QD monotherapy versus weekly MTX monotherapy for prevention of structural progression in MTX-naive subjects with moderately to severely active RA.



# Period 2

To evaluate the long-term safety, tolerability, and efficacy of upadacitinib 7.5 mg QD (for subjects in Japan only), 15 mg QD, and 30 mg QD in subjects with RA who have completed Period 1.

# 5.0 Investigational Plan

# 5.1 Overall Study Design and Plan: Description

This is a Phase 3 multicenter study that includes two periods and a Japan sub-study. Period 1 is a 48-week randomized, double-blind, parallel-group, active comparator controlled treatment period designed to compare the safety and efficacy of upadacitinib 7.5 mg QD monotherapy (for subjects in Japan only), 15 mg QD monotherapy, and 30 mg QD monotherapy versus MTX monotherapy in adult MTX-naïve subjects with moderately to severely active RA. Period 1 is also designed to compare the efficacy of upadacitinib 15 mg QD monotherapy and 30 mg QD monotherapy versus MTX monotherapy for the prevention of structural progression. Period 2 is a long-term extension to evaluate the long-term safety, tolerability, and efficacy of upadacitinib (7.5, 15, or 30 mg QD) in subjects with RA who have completed Period 1. Starting with Amendment 6, subjects receiving upadacitinib 15 mg and 30 mg QD will receive open-label upadacitinib 15 mg QD. Subjects receiving MTX will receive open-label MTX.

The study is designed to enroll approximately 975 subjects at approximately 330 study centers worldwide to meet scientific and regulatory objectives without enrolling an undue number of subjects in alignment with ethical considerations. Therefore, if the target number of subjects has been enrolled, there is a possibility that additional subjects in screening may not be enrolled.

The study duration will include a 35-day screening period, a 48-week randomized, double-blind, parallel-group, active-comparator controlled treatment period (Period 1); a



212 week long-term extension period (blinded until the last subject completes the last visit of Period 1) (Period 2); and a 30-day follow-up (call or site visit).

Subjects will be randomized in a 1:1:1 ratio to treatment Groups 2, 3 and 4 below, except for subjects from Japan, who will be randomized in a 2:1:1:1 ratio to Groups 1, 2, 3 and 4:

- Group 1: Upadacitinib 7.5 mg QD monotherapy (subjects in Japan only; N = 75)
- Group 2: Upadacitinib 15 mg QD monotherapy (N = 300) (includes 37 subjects from Japan)
- Group 3: Upadacitinib 30 mg QD monotherapy (N = 300) (includes 37 subjects from Japan)
- Group 4: MTX monotherapy (N = 300) (includes 37 subjects from Japan)

Each subject will be instructed to take 2 capsules once weekly (MTX and/or matching placebo) and 1 tablet once daily (upadacitinib or matching placebo) to maintain blinding. MTX and matching placebo will be assigned via the Interactive Response Technology (IRT) system, and distributed as identical capsules in blister packs, to provide the correct total dose for each individual subject and to maintain blinding during and after MTX titration (Period 1 and Period 2). Detailed dosing instructions can be found in the Subject Dosing Diary and Instructions. Starting with Amendment 6 subjects receiving MTX will receive open-label MTX tablets in quantities sufficient to cover their respective dose.

Subjects who are assigned to upadacitinib 7.5 mg QD, 15 mg QD, or 30 mg QD will start on their respective upadacitinib dose at Baseline. Subjects who are assigned to the MTX treatment group will start oral MTX treatment at 10 mg/week and will be titrated up to 20 mg/week (increase by 5 mg every 4 weeks), as tolerated, by Week 8 (minimum 15 mg/week final dose required, with documentation of intolerance of > 15 mg/week). (For subjects in Japan: start at 7.5 mg/week with titration up to 10 mg/week at Week 4 and to 15 mg/week, as tolerated, by Week 8; minimum of 7.5 mg/week for final dose is required, with documentation of intolerance of > 7.5 mg/week). After completion of MTX (or placebo) titration, a single dose reduction of study drug (by 5 mg of MTX) is



allowed for safety reasons, up to Week 26, as long as the subject remains on ≥ 15 mg/week of MTX (or matching placebo) weekly (for subjects in Japan: ≥ 7.5 mg/week). In addition, all subjects should take a dietary supplement of oral folic acid (or equivalent) throughout study participation. Folic acid dosing and timing of regimen should be followed according to Investigator's discretion. Rescue therapy has been defined for Weeks 12 through 24, Week 26, and Weeks 36 through 40. Starting at the Week 48 Visit (after Week 48 assessments have been performed) and thereafter, initiation of or change in background RA medication(s), including corticosteroids, non-steroidal anti-inflammatory drugs (NSAIDs), acetaminophen/paracetamol, and csDMARDs (concomitant use of up to 2 csDMARDs except the combination of MTX and leflunomide) is allowed as per local label.

Rescue therapy for those subjects who meet the following criteria from Week 12 through Week 24 are as follows:

Starting at Week 12 through Week 24, those who do not achieve  $\geq$  20% improvement in both TJC and SJC compared with baseline at two consecutive visits will continue on their blinded therapy and the Investigator should optimize (initiate or increase) background RA medications: NSAIDs, corticosteroids (oral  $\leq$  10 mg/day prednisone equivalent or prednisone equivalent  $\leq$  0.5 mg/kg/day for 3 consecutive days) and/or low-potency analgesics.

Rescue therapy for those subjects who meet the following criteria at Week 26 are as follows:

- 1. Subjects who were originally randomized to MTX:
  - Those who do not achieve CR by CDAI:
    - but achieve ≥ 20% improvement in both TJC and SJC compared with baseline will continue on blinded MTX and the Investigator should optimize (initiate or increase) background RA medications: NSAIDs, corticosteroids (oral ≤ 10 mg/day prednisone equivalent and up to 2 local injections), low-potency analgesics and csDMARDs (only 1 of the



- following: sulfasalazine, hydroxychloroquine or chloroquine) throughout the remainder of Period 1 and until the study is unblinded.
- o and do not achieve ≥ 20% improvement in both TJC and SJC compared with baseline will be re-randomized in a 1:1 ratio to receive blinded upadacitinib 15 mg QD or upadacitinib 30 mg QD (for subjects in Japan: randomize 1:1:1 to receive upadacitinib 7.5 mg QD, 15 mg QD, or 30 mg QD) while continuing MTX treatment in a blinded manner and will remain on upadacitinib plus MTX throughout the remainder of Period 1 and until the study is unblinded.
- Those who achieve Clinical Remission (CR) by clinical disease activity index (CDAI) (CDAI ≤ 2.8) at Week 26 will continue blinded treatment with MTX throughout the remainder of Period 1 and until the study is unblinded (the study is unblinded when all subjects have completed Period 1).
- 2. Subjects who were originally randomized to upadacitinib:
  - Those who do not achieve CR by CDAI:
    - o but achieve ≥ 20% improvement in both TJC and SJC compared with baseline will continue on blinded upadacitinib and the Investigator should optimize (initiate or increase) background RA medications: NSAIDs, corticosteroids (oral ≤ 10 mg/day prednisone equivalent and up to 2 local injections), low potency analgesics and csDMARDs (only 1 of the following: sulfasalazine, hydroxychloroquine or chloroquine) throughout the remainder of Period 1 and until the study is unblinded.
    - and do not achieve ≥ 20% improvement in both TJC and SJC compared with baseline will add MTX 10 mg/week (7.5 mg for Japan) to upadacitinib in a blinded manner and will remain on upadacitinib plus MTX 10 mg/week (7.5 mg for Japan) throughout the remainder of Period 1 and until the study is unblinded.
  - Those who achieve Clinical Remission (CR) by CDAI (CDAI ≤ 2.8) at Week 26 will continue blinded treatment with upadacitinib throughout the remainder of Period 1 and until the study is unblinded (the study is unblinded when all subjects have completed Period 1).


Rescue therapy for those subjects who meet the following criteria from Week 36 through Week 40 are as follows:

• Starting at Week 36 through Week 40, those who do not achieve ≥ 20% improvement in both TJC and SJC compared with baseline at two consecutive visits will continue on their blinded therapy and the Investigator should optimize (initiate or increase) background RA medications: NSAIDs, corticosteroids (oral ≤ 10 mg/day prednisone equivalent or prednisone equivalent ≤ 0.5 mg/kg/day for 3 consecutive days and up to 2 local injections), low-potency analgesics and csDMARDs (only 1 of the following: sulfasalazine, hydroxychloroquine or chloroquine).

An unblinded analysis will be conducted after all subjects have completed Week 24 for the purpose of regulatory submission. To maintain integrity of the trial and avoid introduction of bias, study sites and subjects will remain blinded for the duration of Period 1. Additional unblinded analyses may be conducted after the first unblinded analysis for regulatory purposes.

Each subject will undergo a maximum of 3 scheduled visits for x-ray examination of bilateral hands and feet during Period 1 (unless unscheduled repeat imaging is needed due to failure to meet the quality requirements) at Screening, Week 24, and Week 48/Premature Discontinuation. One additional x-ray examination of bilateral hands and feet may be needed depending on the time of premature study drug discontinuation for those subjects that continue the study (refer to Section 5.3.1.1 for additional details).

Subjects who complete the Week 48 Visit (end of Period 1) will enter the long-term extension, Period 2 (212 weeks). Subjects will continue study treatment per assignment at the end of Period 1 in a blinded fashion. When the last subject completes the last visit of Period 1 (Week 48), study drug assignment in both periods may be unblinded to the Sponsor and sites, and subjects would then be dispensed study drug in an open-label fashion until the completion of Period 2. All subjects will continue study treatment to which they were assigned at the time of study unblinding. Dose changes of open-label



study drugs are not permitted during unblinded Period 2. Background therapies may be adjusted as per the discretion of the investigator (refer to Section 5.3.1.1 for additional details on permitted background therapy in Period 2).

Each subject will undergo a maximum of 3 scheduled visits for x-ray examination of bilateral hands and feet during Period 2 (unless unscheduled repeat imaging is needed due to failure to meet the quality requirements) at Week 96, Week 192, and Week 260. Subjects who prematurely discontinue from Period 2 will undergo an x-ray of hands and feet unless the previous x-ray was performed within the previous 24 weeks.

Starting with Amendment 6, subjects receiving upadacitinib 15 mg and 30 mg QD will receive open-label upadacitinib 15 mg QD. Subjects receiving MTX will receive open-label MTX.

Study design schematics of Period 1 and Period 2 are shown in Figure 1 and Figure 2, respectively.

Figure 1. Period 1 Study Design



 $MTX = methotrexate; \ n = number; \ QD = once \ daily; \ SJC = swollen \ joint \ count; \ TJC = tender \ joint \ count; \ W = week$ 

- \* Evaluation for inadequate responders to determine need for rescue therapy at Week 26; refer to Section 5.2.3.3.
- † Evaluation for inadequate responders to determine need for rescue therapy at Weeks 12 24 and Weeks 36 40; refer to Section 5.2.3.3.

Note: The follow-up period is only for subjects who do not enter Period 2.

Figure 2. Period 2 Study Design

# MTX-Naïve /Structure (M13-545) Continued



csDMARD = conventional synthetic disease modifying anti-rheumatic drug; NSAIDs = non-steroidal anti-inflammatory drugs; QD = once daily; RA = rheumatoid arthritis; W = week

Note: Period 2 will remain blinded until the last subject completes Week 48 (Period 1). Subjects who prematurely discontinue from Period 2 will undergo an x-ray of hands and feet unless the previous x-ray was performed within the previous 24 weeks.

Starting with Amendment 6, subjects receiving upadacitinib 15 mg and 30 mg QD will receive open-label upadacitinib 15 mg QD. Subjects receiving MTX will receive open-label MTX.

# **Screening Period**

Within 35 days prior to the Baseline Visit, subjects will receive a full explanation of the study design and study procedures, provide a written informed consent, and undergo the screening procedures outlined in Appendix D. Lab values can be re-tested once during



the screening period. If the re-tested lab value(s) remain exclusionary, the subject will be considered a screen failure with no additional re-screening possible. Redrawing samples if initial samples were unable to be analyzed would not count as a retest since initial result was never obtained.

Subjects that initially screen fail for the study are permitted to re-screen once following re-consent. For additional re-screening, AbbVie Therapeutic Area Medical Director approval is required. All screening procedures with the possible exceptions noted below will be repeated during re-screening. The subject must meet all the inclusion and none of the exclusion criteria at the time of re-screening in order to qualify for the study. There is no minimum period of time a subject must wait to re-screen for the study. If the subject had a complete initial screening evaluation including the assessment of an Interferon-Gamma Release Assay (IGRA; QuantiFERON Tuberculosis [TB] Gold In Tube test) or a purified protein derivative (PPD) test (or equivalent), or chest x-ray and electrocardiogram (ECG), these tests will not be required to be repeated for re-screening provided the conditions noted in Section 5.2 are met and no more than 90 days have passed.

#### Period 1 (48-Week Randomized, Double-Blind Treatment Period)

Period 1 will begin at the Baseline Visit (Day 1) and will end at the Week 48 Visit. At the Baseline Visit, subjects who meet all the inclusion criteria and none of the exclusion criteria described in Section 5.2.1 and Section 5.2.2 will be enrolled into the study and randomized to double-blind treatment. During this period of the study, subjects will visit the study site at Weeks 2, 4, 8, 12, 16, 20, 24, 26, 28, 32, 36, 40, and 48. A  $\pm$  3 day window is permitted around scheduled study visits until Week 32 and then  $\pm$  7 days for the remainder of the period. The last dose of study drug in Period 1 is taken the day prior to the Week 48 Visit. Subjects who complete Period 1, but decide not to continue in Period 2 should complete a 30 day follow-up visit after the last dose of study drug.



## Period 2 (Long-Term Extension Period [212 Weeks])

Period 2 will begin at Week 48 Visit after all assessments have been completed. During Period 2, subjects will visit the study site at Weeks 60, 72, 84, 96, every 12 weeks through Week 240, and Week 260/PD. A ± 7-day window is permitted around scheduled study visits. Starting at Week 48, subjects who fail to show at least 20% improvement in both TJC and SJC compared to baseline at 2 consecutive visits, despite optimization of background RA therapies (see Section 5.2.3.1 for permitted background RA therapies), will be discontinued from study drug. Therefore, the earliest discontinuation would be at Week 60, after completion of all Week 60 study visit activities.

Starting with Amendment 6, subjects receiving upadacitinib 15 mg and 30 mg QD will receive open-label upadacitinib 15 mg QD. Subjects receiving MTX will receive open-label MTX.

# Discontinuation of Study Drug and Continuation of Study Participation (Period 1 and Period 2)

Subjects may discontinue study drug treatment, but may choose to continue to participate in the study (refer to Section 5.4.1 for additional details). Subjects who prematurely discontinue study drug should complete a Premature Discontinuation visit (PD visit) as soon as possible, preferably within 2 weeks, and preferably prior to initiation of another therapy. To minimize missing data for efficacy and safety assessments, subjects who prematurely discontinue study drug treatment should continue to be followed for all regularly scheduled visits as outlined in the Activity Schedule (Appendix D and Appendix F), unless subjects have decided to discontinue study participation entirely (withdrawal of informed consent). Subjects should be advised on the continued scientific importance of their data even if they discontinue treatment with study drug early. Following discontinuation of study drug, the subject should be treated in accordance with the investigator's best clinical judgment irrespective of whether the subject decides to continue participation in the study. In addition, all future rescue- and efficacy-driven discontinuation criteria no longer apply. This includes 20% TJC/SJC calculations at Weeks 12 – 24, Weeks 36 – 40 and Week 48 and thereafter, as well as CDAI calculation



at Week 26, if applicable. If at any point a subject no longer wants to provide assessments (withdrawal of informed consent) following discontinuation of study drug, a second PD visit is not required.

# Premature Discontinuation of Study (Withdrawal of Informed Consent) (Period 1 and Period 2)

Subjects may withdraw from the study completely (withdrawal of informed consent) for any reason at any time (refer to Section 5.4.1 for additional details). If a subject prematurely discontinues study drug treatment and study participation (withdrawal of informed consent) the procedures outlined for the Premature Discontinuation Visit (PD Visit) should be completed as soon as possible, preferably within 2 weeks of study drug discontinuation and preferably prior to initiation of another therapy. In addition, if the subject is willing, a 30-day follow-up visit (or phone call if a visit is not possible) may occur to determine the status of any ongoing AEs/SAEs or the occurrence of any new AEs/SAEs.

#### Follow-Up Visit

A Follow-Up Visit will occur approximately 30 days after the last dose of study drug to obtain information on any new or ongoing AE/SAEs, and to collect vital signs and clinical laboratory tests.

Subjects will complete the Follow-Up Visit when they have either:

- Completed the last visit of Period 1 (Week 48), but decided not to participate in the extension Period 2; OR
- Completed the last visit of Period 2 (Week 260); OR
- Prematurely discontinued study drug and/or study participation. This visit
  may be a telephone call if a site visit is not possible. Vital signs and laboratory
  test may not be required. The Follow-Up Visit is not applicable for subjects
  who discontinued study drug and continued study participation and completed
  at least one study visit at least approximately 30 days after last dose.



#### Protocol Modifications due to State of Emergency or Pandemic like COVID-19

Study visits may be impacted by a pandemic situation (including the COVID-19 pandemic) or any state of emergency. If visits cannot be conducted onsite due to travel restrictions or other pandemic-related reasons, virtual visits, visits at alternative locations, or changes in the visit frequency and timing of study procedures, among others may be performed. Additional details are provided in the subsequent sections. Every effort should be made to ensure the safety of subjects and site staff, while maintaining the integrity of the study.

# 5.2 Selection of Study Population

It is anticipated that approximately 975 subjects with moderately to severely active RA will be randomized at approximately 330 study centers, globally.

A subject may be enrolled in this study provided that he/she has met all of the inclusion criteria specified in Section 5.2.1 and none of the exclusion criteria specified in Section 5.2.2 of this protocol.

#### 5.2.1 Inclusion Criteria

- 1. Adult male or female, at least 18 years old.
- Duration of symptoms consistent with RA for ≥ 6 weeks who also fulfill the 2010 ACR/EULAR classification criteria for RA.
- 3. Naïve to MTX or, if already on MTX, have received no more than 3 weekly MTX doses with requirement to complete a 4-week MTX washout before the first dose of study drug.
- 4. Subjects with prior exposure to csDMARDs other than MTX may be enrolled if completed the washout period as specified below or should be at least five times the mean terminal elimination half-life of a drug:



- ≥ 4 weeks prior to first dose of study drug for minocycline, penicillamine, sulfasalazine, hydroxychloroquine, chloroquine, azathioprine, gold formulations, cyclophosphamide, tacrolimus, cyclosporine, mycophenolate;
- ≥ 8 weeks prior to first dose of study drug for leflunomide if no elimination procedures was followed, or adhere to an elimination procedure (i.e., 11 days with colestyramine, or 30 days washout with activated charcoal or as per local label).
- 5. Subject meets both of the following disease activity criteria:
  - a. ≥ 6 swollen joints (based on 66 joint counts) and ≥ 6 tender joints (based on 68 joint counts) at Screening and Baseline Visits; and
  - b.  $hsCRP \ge 5 \text{ mg/L}$  (central lab, ULN 2.87 mg/L) at Screening Visit.
- 6. ≥ 1 bone erosion on x-ray (by local reading) OR in the absence of documented bone erosion, both positive rheumatoid factor (RF) and positive anti-cyclic citrullinated peptide (anti-CCP) autoantibodies are required at Screening.
- 7. Stable dose of non-steroidal anti-inflammatory drugs (NSAIDs), acetaminophen, oral corticosteroids (equivalent to prednisone ≤ 10 mg/day), or inhaled corticosteroids for stable medical conditions are allowed but must have been at a stable dose ≥ 1 week prior to the first dose of study drug.
- 8. Subjects must have discontinued all high-potency opiates prior at least 1 week to the first dose of study drug (refer to Section 5.2.3.2 for prohibited medications).
- 9. Women of childbearing potential (refer to Section 5.3.1.1), must not have a positive pregnancy test at the Screening or Baseline Visits. *Note: Subjects with borderline pregnancy tests at Screening must have a serum pregnancy test ≥ 3 days later to document continued lack of a positive result.*
- 10. If female, subject must be postmenopausal, OR permanently surgically sterile, OR for women of childbearing potential practicing at least one protocol-specified method of birth control (refer to Section 5.2.4), that is effective from Study Day 1 through at least 180 days after the last dose of study drug.

- Additional local requirements may apply. Refer to Appendix C for local requirements.
- 11. Male subjects who are sexually active with female partner(s) of childbearing potential must agree from Study Day 1 through 180 days after the last dose of study drug to practice the protocol-specified contraception (refer to Section 5.2.4).
  - Additional local requirements may apply. Refer to Appendix C for local requirements.
- 12. Subjects must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.

#### **Rationale for Inclusion Criteria**

| 1 - 8 | To select the appropriate subject population |
|---|---|
| 9 – 11 | Upadacitinib is teratogenic in both rats and rabbits. The effect of upadacitinib on human pregnancy and reproduction is unknown. |
| 12 | In accordance with harmonized Good Clinical Practice (GCP) |

#### 5.2.2 Exclusion Criteria

- 1. Intolerant to MTX.
- 2. Prior exposure to any JAK inhibitor (including but not limited to tofacitinib, baricitinib, and filgotinib).
- 3. Prior exposure to any bDMARD(s).
- 4. History of any arthritis with onset prior to age 17 years or current diagnosis of inflammatory joint disease other than RA (including but not limited to gout, systemic lupus erythematosus, psoriatic arthritis, axial spondyloarthritis including ankylosing spondylitis and non-radiographic axial spondyloarthritis, reactive arthritis, overlap connective tissue diseases, scleroderma, polymyositis,



- dermatomyositis, fibromyalgia [currently with active symptoms]). Current diagnosis of secondary Sjogren's Syndrome is permitted.
- 5. Has been treated with intra-articular, intramuscular, intravenous, trigger point or tender point, intra-bursa, or intra-tendon sheath corticosteroids in the preceding 8 weeks prior to the first dose of study drug.
- 6. Has been treated with any investigational drug within 30 days or five half-lives of the drug (whichever is longer) prior to the first dose of study drug or is currently enrolled in another clinical study.
- 7. Female who is pregnant, breastfeeding or considering becoming pregnant during the study or for approximately 180 days after the last dose of study drug.
- 8. Male subject who is considering fathering a child or donating sperm during the study or for approximately 180 days after the last dose of study drug.
- 9. Any active or recurrent viral infection that, based on the Investigator's clinical assessment, makes the subject an unsuitable candidate for the study, including hepatitis B virus (HBV) or hepatitis C virus (HCV), recurrent or disseminated (even a single episode) herpes zoster, disseminated (even a single episode) herpes simplex, or known history of human immunodeficiency virus (HIV). Active HBV and HCV are defined as:
  - HBV: hepatitis B surface antigen (HBs Ag) positive (+) or detected sensitivity on the HBV deoxyribonucleic acid (DNA) polymerase chain reaction (PCR) qualitative test for Hepatitis B core antibody (HBc Ab) positive (+) subjects; (and for Hepatitis B surface antibody positive [+] subjects in Japan only);
  - HCV: HCV ribonucleic acid (RNA) detectable in any subject with anti-HCV antibody (HCV Ab).
- 10. Subject has active TB or meets TB exclusionary parameters (refer to Section 5.3.1.1 for specific requirements for TB testing).



- 11. Systemic use of known strong cytochrome P450 3A (CYP3A) inhibitors or strong CYP3A inducers from Screening through the end of the study (refer to Table 1 for examples of commonly used strong CYP3A inhibitors and inducers).
- 12. Receipt of any live vaccine within 4 weeks prior to the first dose of study drug, or expected need of live vaccination during study participation including at least 4 weeks after the last dose of study drug.
- 13. History of any malignancy except for successfully treated NMSC or localized carcinoma in situ of the cervix.
- 14. History of clinically significant (per Investigator's judgment) drug or alcohol abuse within the last 6 months.
- 15. History of gastrointestinal perforation (other than appendicitis or penetrating injury), diverticulitis, or significantly increased risk for GI perforation per investigator judgment.
- 16. Conditions that could interfere with drug absorption including but not limited to short bowel syndrome.
- 17. Subject has been a previous recipient of an organ transplant.
- 18. History of clinically significant medical conditions or any other reason that in the opinion of the Investigator would interfere with the subject's participation in this study or would make the subject an unsuitable candidate to receive study drug.
- 19. Active infection(s) requiring treatment with parenteral anti-infectives within 30 days, or oral anti-infectives within 14 days prior the first dose of study drug.
- 20. History of an allergic reaction or significant sensitivity to constituents of the study drug(s) (and their excipients) and/or other products in the same class.
- 21. Laboratory values meeting the following criteria within the Screening period prior to the first dose of study drug:
  - Serum aspartate transaminase (AST)  $> 2 \times ULN$
  - Serum alanine transaminase (ALT)  $> 2 \times ULN$



- Estimated glomerular filtration rate (GFR) by simplified 4-variable Modification of Diet in Renal Disease (MDRD) formula < 40 mL/min/1.73 m<sup>2</sup>
- Total white blood cell count (WBC)  $< 2,500/\mu$ L
- Absolute neutrophil count (ANC)  $< 1,500/\mu L$
- Platelet count  $< 100,000/\mu L$
- Absolute lymphocyte count < 800/μL
- Hemoglobin < 10 g/dL
- 22. History of any of the following cardiovascular conditions:
  - Moderate to severe congestive heart failure (New York Heart Association class III or IV),
  - Recent (within past 6 months) cerebrovascular accident, myocardial infarction, coronary stenting;
  - Uncontrolled hypertension as defined by a persistent, confirmed systolic blood pressure (BP) > 160 mmHg or diastolic BP > 100 mmHg.
  - Any other condition which, in the opinion of the Investigator, would put the subject at risk by participating in the protocol.
- 23. Clinically relevant or significant ECG abnormalities, including ECG with QT interval corrected for heart rate (QTc) using Fridericia's correction formula (QTcF) > 500 msec.
- 24. For subjects in Japan only: Positive result of beta-D-glucan (screening for pneumocystis jiroveci infection).

#### **Rationale for Exclusion Criteria**

| 1-2 | To select the appropriate subject population |
|---|---|
| 7 – 8 | Upadacitinib is teratogenic in both rats and rabbits. The effect of upadacitinib on human pregnancy and reproduction is unknown. |
| 3-6, 9-24 | To ensure safety of the subjects throughout the study |



## 5.2.3 Prior, Concomitant, and Prohibited Therapy

Any medication or vaccine (including over-the-counter or prescription medicines, vitamins and/or herbal supplements including folic acid) that the subject is receiving within 28 days prior to Screening, or receives during the study, must be recorded along with the reason for use, date(s) of administration including start and end dates, and dosage information including dose, route and frequency on the appropriate electronic case report form (eCRF). Also, medications including but not limited to DMARDs taken for RA (based on subject recollection and available medical records), should be entered into the appropriate eCRF.

The AbbVie Therapeutic Area Medical Director should be contacted if there are any questions regarding concomitant or prior therapies.

# 5.2.3.1 Permitted Background RA Therapy

Subjects should continue on their stable doses of NSAIDs, acetaminophen/paracetamol, oral corticosteroids (equivalent to prednisone  $\leq 10$  mg/day), or inhaled corticosteroids.

- If taking any of the above on a scheduled basis, they should continue to take them as they did at study entry with no change in dose or frequency, including on study visit days.
- If not taking any of the above at baseline, these must not be initiated except where permitted by protocol-defined rescue therapy.
- If taking any of the above, including low potency analgesics, i.e., tramadol, codeine, hydrocodone, or propoxyphene at baseline on an as-needed basis (PRN), they should continue to use them for the same reason and same dose each time but they should not be taken within the 24 hours prior to any study visit to avoid bias in outcome measurements.

In the event of tolerability (or other safety) issues, the doses of these medications may be decreased or discontinued with substitution of another permitted medication from that class (see Section 5.2.3.2 for prohibited therapies). PRN use of inhaled corticosteroids is permitted at any time.



In Period 1, starting at Week 26 (after Week 26 assessments have been performed) and thereafter, intra-articular, intramuscular, intravenous, trigger point or tender point, intrabursa, and intra-tendon sheath injections of corticosteroids, dosage and frequency per standard of care, are allowed. To avoid confounding effects of systemic absorption of intra-articular corticosteroids, joint injections should be avoided, if possible, within 21 days prior to the next scheduled study visit. For the analysis of the TJC and SJC, injected joints will be considered "not assessable" for 3 months from the time of the intra-articular injection. Refer to Section 5.2.3.3 for rescue therapy at Week 26.

In Period 2, starting at Week 48 (after Week 48 assessments have been performed) and thereafter, initiation of or change in corticosteroids (including: oral, intra-articular, trigger point or tender point, intra-bursa, intra-tendon sheath, intramuscular and intravenous) is allowed. In addition, the initiation of or change in NSAIDs, acetaminophen/paracetamol and low potency narcotics is also permitted to optimize concomitant RA medications. Adding one of the following, sulfasalazine, hydroxychloroquine, or chloroquine, is also permitted, as per local label. Period 2 may be unblinded after all subjects complete Period 1, at which time the Investigator will know if the subject is taking MTX or MTX placebo. If subject is not taking MTX, he/she may add a maximum of 2 csDMARDs, including MTX, leflunomide, sulfasalazine, hydroxychloroquine, or chloroquine, but not MTX plus leflunomide. For RA flare treatment, no more than 3 consecutive days of high-dose systemic corticosteroids (maximum dose of 0.5 mg/kg/day of prednisone or its equivalent) are allowed, after which subject should resume his/her usual daily oral corticosteroid dose.

#### **Traditional Chinese Medicine**

Traditional oral Chinese medicine cannot be initiated or changed during the study as these may interfere with upadacitinib metabolism and exposure and may impact efficacy and safety of upadacitinib treatment.



# 5.2.3.2 Prohibited Therapy

Local label recommendations for contraindicated concomitant therapies with MTX (i.e., trimethoprim-sulfamethoxazole) should be followed.

#### **JAK Inhibitor**

Prior exposure to JAK inhibitors and concurrent use during the study (including but not limited to tofacitinib [Xeljanz<sup>®</sup>], baricitinib, and filgotinib) is not allowed.

#### **Corticosteroids**

Oral corticosteroids > 10 mg prednisone/day, or equivalent, are NOT allowed in Period 1. Intra-articular, intramuscular, intravenous, trigger point or tender point, intra-bursa, and intra-tendon sheath corticosteroids are NOT allowed up to Week 26. There are exceptions if rescue therapy is needed between Weeks 12 and 24. Refer to Section 5.2.3.3.

## **Biologic Therapies**

All biologic therapies are prohibited during the study (i.e., Periods 1 and 2).

Subjects with prior exposure to bDMARDs are excluded from participation in this study.

Examples of biologic therapies include but are not limited to the following:

- Humira® (adalimumab)
- Enbrel® (etanercept)
- Remicade® (infliximab)
- Orencia® (abatacept)
- Kineret<sup>®</sup> (anakinra)
- Rituxan® (rituximab)
- Cimzia<sup>®</sup> (certolizumab pegol)
- Simponi<sup>®</sup> (golimumab)
- Actemra® (tocilizumab)



- Raptiva® (efalizumab)
- Tysabri<sup>®</sup> (natalizumab)
- Stelara® (ustekinumab)
- Benlysta® (belimumab)
- Dupixent® (dupilumab)
- Taltz<sup>®</sup> (ixekizumab)
- Cosentyx® (secukinumab)
- Entyvio® (vedolizumab)

## csDMARD Therapies

Subjects must be naïve to MTX; however, those who have received not more than 3 weekly doses of MTX may be enrolled if they complete a 4-week washout of the MTX before the first dose of study drug (Inclusion Criterion 3, Section 5.2.1).

Subjects must have discontinued all csDMARDs prior to Baseline Visit as specified in the washout procedures (Inclusion Criterion 4, Section 5.2.1).

# **Strong CYP3A Inhibitors or Inducers**

Systemic use of known strong CYP3A inhibitors or strong CYP3A inducers is excluded from the Screening Visit through the end of the study (i.e., Periods 1 and 2). The most common strong CYP3A inhibitors and inducers are listed in Table 1.



Table 1. Examples of Commonly Used Strong CYP3A Inhibitors and Inducers

| Strong CYP3A Inhibitors | Strong CYP3A Inducers |
|-----------------------------|-----------------------|
| Boceprevir | Avasimibe |
| Cobicistat | Carbamazepine |
| Clarithromycin | Phenytoin |
| Conivaptan | Rifampin |
| Grapefruit (fruit or juice) | Rifapentine |
| Indinavir | St. John's Wort |
| Itraconazole | |
| Ketoconazole | |
| Lopinavir/Ritonavir | |
| Mibefradil | |
| Nefazodone | |
| Nelfinavir | |
| Posaconazole | |
| Ritonavir | |
| Saquinavir | |
| Telaprevir | |
| Telithromycin | |
| Troleandomycin | |
| Voriconazole | |

In Period 2, when study drug has been unblinded, systemic use of known strong CYP3A inhibitors or strong CYP3A inducers is permitted for subjects not receiving upadacitinib.

#### **Opiates**

High potency opiates are not permitted during the study (i.e., Periods 1 and 2), with the exception of analgesic care related to AEs or SAEs and subjects must have discontinued high potency opiates at least 1 week prior to the first dose of study drug, including (but not limited to):

- oxycodone
- oxymorphone
- fentanyl
- levorphanol
- buprenorphine



- methadone
- hydromorphone
- morphine
- meperidine

#### **Investigational Drugs**

Subjects who have been treated with any investigational drug within 30 days or five half-lives of the drug (whichever is longer) prior to the first dose of study drug are excluded from participation in this study. Investigational drugs are also prohibited during the study.

#### **Vaccines**

Although not mandated by the protocol, vaccines recommended by local guidelines should be considered. If the subject and investigator choose to administer live vaccines, these vaccinations must be completed (per local label) 4 weeks before first dose of study drug with appropriate precautions. Live vaccinations are prohibited during Period 1, including at least 30 days (or longer if required locally) after last dose of study drug.

Examples of live vaccines include, but are not limited to, the following:

- Monovalent live influenza A (H1N1) (intranasal);
- Seasonal trivalent live influenza (intranasal);
- Zostavax (herpes zoster, live attenuated);
- Rotavirus;
- Varicella (chicken pox);
- Measles-mumps-rubella or measles mumps rubella varicella;
- Oral polio vaccine;
- Smallpox;
- Yellow fever;
- Bacille Calmette-Guérin (BCG);



#### • Typhoid.

In Period 2, if a live vaccine must be administered during study participation, study drug must be held for at least 30 days prior to the vaccination and at least 30 days after the vaccination (or longer if required locally).

If the live herpes zoster vaccine is to be administered and there is no known history of primary varicella (chicken pox), preexisting immunity to varicella should be confirmed with antibody testing prior to administration of the herpes zoster vaccine. If varicella antibody testing is negative, the live herpes zoster vaccine should not be administered.

Administration of inactivated (non-live) vaccines is permitted during the study according to local practice guidelines. Examples of common vaccines that are inactivated, toxoid or biosynthetic, include but are not limited to: injectable influenza vaccine, pneumococcal, Shingrix (zoster vaccine, recombinant, adjuvanted) and, pertussis (Tdap) vaccines.

If the nasal Influenza vaccine is administered, the vaccine must be administered at least 4 weeks prior to first dose of study drug.

# 5.2.3.3 Rescue Therapy

Rescue therapy for those subjects who meet the following criteria from Week 12 through Week 24 are as follows:

• Those who do not achieve ≥ 20% improvement in both TJC and SJC compared with baseline at two consecutive visits starting at Week 12 will continue on their blinded therapy and the Investigator should optimize (initiate or increase) background RA medications: NSAIDs, corticosteroids (oral ≤ 10 mg/day prednisone equivalent or prednisone equivalent ≤ 0.5 mg/kg/day for 3 consecutive days) and/or low-potency analgesics.

Rescue therapy for those subjects who meet the following criteria at Week 26 are as follows:



- 1. Subjects who were originally randomized to MTX:
  - Those who do not achieve CR by CDAI:
    - o but achieve ≥ 20% improvement in both TJC and SJC compared with baseline will continue on blinded MTX and the Investigator should optimize (initiate or increase) background RA medications: NSAIDs, corticosteroids (oral ≤ 10 mg/day prednisone equivalent and up to 2 local injections), low-potency analgesics and csDMARDs (only 1 of the following: sulfasalazine, hydroxychloroquine or chloroquine) throughout the remainder of Period 1 and until the study is unblinded.
    - o and do not achieve ≥ 20% improvement in both TJC and SJC compared with baseline will be re-randomized in a 1:1 ratio to receive blinded upadacitinib 15 mg QD or upadacitinib 30 mg QD (for subjects in Japan: randomize 1:1:1 to receive upadacitinib 7.5 mg QD, 15 mg QD, or 30 mg QD) while continuing MTX treatment in a blinded manner and will remain on upadacitinib plus MTX throughout the remainder of Period 1 and until the study is unblinded.
  - Those who achieve Clinical Remission (CR) by CDAI (CDAI ≤ 2.8) at
    Week 26 will continue blinded treatment with MTX throughout the remainder
    of Period 1 and until the study is unblinded (the study is unblinded when all
    subjects have completed Period 1).
- 2. Subjects who were originally randomized to upadacitinib:
  - Those who do not achieve CR by CDAI:
    - o but achieve ≥ 20% improvement in both TJC and SJC compared with baseline will continue on blinded upadacitinib and the Investigator should optimize (initiate or increase the dose) background RA medications: NSAIDs, corticosteroids (oral ≤ 10 mg/day prednisone equivalent and up to 2 local injections), low potency analgesics and csDMARDs (only 1 of the following: sulfasalazine, hydroxychloroquine or chloroquine) throughout the remainder of Period 1 and until the study is unblinded.
    - but do not achieve ≥ 20% improvement in both TJC and SJC compared with baseline will add MTX 10 mg/week (7.5 mg for Japan) to upadacitinib in a blinded manner and will remain on upadacitinib plus



MTX 10 mg/week (7.5 mg for Japan) throughout the remainder of Period 1 and until the study is unblinded.

• Those who achieve CR by CDAI (CDAI ≤ 2.8) at Week 26 will continue blinded treatment with upadacitinib throughout the remainder of Period 1 and until the study is unblinded (the study is unblinded when all subjects have completed Period 1).

Rescue therapy for those subjects who meet the following criteria from Week 36 through Week 40 are as follows:

• Those who do not achieve ≥ 20% improvement in both TJC and SJC compared with baseline at two consecutive visits starting at Week 36 will be rescued with optimizing (initiate or increase) background RA medications: NSAIDs, corticosteroids (oral ≤ 10 mg/day prednisone equivalent or prednisone equivalent ≤ 0.5 mg/kg/day for 3 consecutive days and up to 2 local injections), low-potency analgesics and csDMARDs (only 1 of the following: sulfasalazine, hydroxychloroquine or chloroquine).

# 5.2.4 Contraception Recommendations

#### **Contraception Recommendation for Females**

A woman who is postmenopausal or permanently surgically sterile (bilateral oophorectomy, bilateral salpingectomy or hysterectomy) is not considered to be a woman of childbearing potential and is not required to follow contraception recommendations. Postmenopausal is defined as:

- Age ≥ 55 years with no menses for 12 or more months without an alternative medical cause; or
- Age < 55 years with no menses for 12 or more months without an alternative medical cause AND an FSH level > 40 mIU/mL.



If the female subject is < 55 years of age:

AND has had no menses for  $\geq$  12 months AND has no history of permanent surgical sterilization (defined above), FSH should be tested at Screening.

- If FSH is not tested, it is assumed that the subject is of childbearing potential and protocol-specified contraception is required.
- If the FSH is tested and the result is consistent with post-menopausal status, contraception is not required.
- If the FSH is tested and the result is consistent with pre-menopausal status, contraception is required and a serum pregnancy test must be performed (see Section 5.3.1.1 pregnancy test).

For a female subject at any age:

- Female subjects with menses within the past 12 months are of childbearing potential and FSH is therefore not required but contraception is required.
- Female subjects who are surgically sterile (defined above) are not of childbearing potential and therefore no FSH testing or contraception is required.

A woman who does not meet the definition of postmenopausal or permanently surgically sterile is considered of childbearing potential and is required to practice at least one of the following highly effective methods of birth control that is effective from Study Day 1 (or earlier) through at least 180 days after the last dose of study drug.

- Combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal, injectable) associated with the inhibition of ovulation, initiated at least 30 days prior to Study Day 1.
- Progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation, initiated at least 30 days prior to Study Day 1.
- Bilateral tubal occlusion/ligation.



- Vasectomized partner(s), provided the vasectomized partner has received medical confirmation of the surgical success and is the sole sexual partner of the women of childbearing potential trial participant.
- Intrauterine device (IUD).
- Intrauterine hormone-releasing system (IUS).
- True abstinence (if acceptable per local requirements): Refraining from heterosexual intercourse when this is in line with the preferred and usual lifestyle of the subject (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable).

If required per local practices, male or female condom with or without spermicide OR cap, diaphragm or sponge with spermicide should be used in addition to one of the highly effective birth control methods listed above (excluding true abstinence).

It is important to note that contraception recommendations described above are specifically intended to prevent pregnancy during and after exposure to the investigational therapies, upadacitinib and MTX. In Period 2, starting at Week 48, concomitant csDMARDs (i.e., sulfasalazine, hydroxychloroquine, chloroquine and leflunomide) can be prescribed, per standard of care. The duration of contraception after discontinuation of these prescribed csDMARDs should be based on the local label.

If during the course of the study a woman becomes surgically sterile or post-menopausal and complete documentation is available, contraception measures as defined above are no longer required.

Additional local requirements may apply. Refer to Appendix C for local requirements (Canada and Colombia).

#### **Contraception Recommendation for Males**

There are no contraception requirements for male subjects receiving upadacitinib only, or their female partner(s).



For a male subject receiving MTX who has a female partner who is postmenopausal or permanently sterile, no contraception is required.

A male subject receiving MTX who is sexually active with female partner(s) of childbearing potential must agree from Study Day 1 through 180 days after the last dose of MTX study drug to practice contraception with:

- Condom use and female partner(s) using at least one of the contraceptive measures (as defined in the protocol for female study subjects of childbearing potential).
- True abstinence: Refraining from heterosexual intercourse-when this is in line with the preferred and usual lifestyle of the subject. (Note: Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable).

Additionally, male subjects receiving MTX must agree not to donate sperm from Study Day 1 through 180 days after the last dose of MTX study drug.

Male subjects receiving MTX are responsible for informing his partner(s) of the risk of becoming pregnant and for reporting any pregnancy to the study doctor.

It is important to note that contraception and sperm donation recommendations described above are specifically intended to prevent pregnancy during and after exposure to the investigational therapy, MTX. In Period 2, starting at Week 48, concomitant csDMARDs (i.e., sulfasalazine, hydroxychloroquine, chloroquine and leflunomide) can be prescribed, per standard of care. The duration of contraception and requirement not to donate sperm after discontinuation of these prescribed csDMARDs should be based on the local label.

Additional local requirements may apply. Refer to Appendix C for local requirements (Canada and Colombia).



# 5.3 Efficacy Pharmacokinetic, Pharmacodynamic, Exploratory Research and Validation Studies, and Safety Assessments/Variables

# 5.3.1 Efficacy and Safety Measurements Assessed and Flow Chart

Study procedures described are listed in the following section of this protocol and are summarized in tabular format in Appendix D, Appendix E, and Appendix F.

Study visits may be impacted by cases of state of emergency or pandemic situations like COVID-19. This may include changes such as virtual visits, visits at alternative locations, or changes in the visit frequency and timing of study procedures, among others. Additional details are provided in Section 5.3.1.1.

Every effort should be made to ensure the safety of subjects and site staff, while maintaining the integrity of the study.

Supplemental study case report forms should be completed in the event of missed/virtual visits, or study drug interruptions or discontinuations related to COVID-19.

Study Visits and/or activities should be performed as scheduled whenever possible. During a state of emergency or pandemic situation, if it is not possible for all study procedures to be performed as specified due to travel restrictions or other reasons, the following modifications are allowed:

- If permitted by local regulations, the IRB/IEC and the subject, study visits may be conducted in a subject's home residence (see Section 5.3.1.1 Sub-Section "Optional Home Healthcare Service Due to State of Emergency or Pandemic Situation like COVID-19").
- The following study activities may be performed virtually by phone/video conference:
  - Adverse event assessment
  - Concomitant therapy assessment including compliance to contraception requirements, if applicable

- Latent TB risk assessment
- Communication of in-home urine pregnancy test result
- Dispense study drug and subject dosing diary (see Section 5.3.1.1 Sub-Section "Study Drug Dispensing, Dosing, and Compliance" for details about the Direct-to-Patient shipment)
- Review of subject dosing diary, compliance to IP administrations
- During a virtual visit, the following activities should not be performed:
  - Patient questionnaires
  - X-rays (bilateral hands/feet)
  - Vital signs and body weight
  - Physical exam
  - Physician Global Assessment (PhGA)
  - o TJC68/SJC66
- The following study activities may be performed by a local clinic/hospital/laboratory:
  - QuantiFERON-TB Gold test or equivalent (and/or local PPD skin test)
  - Chest x-ray, if the Investigator has determined, based on clinical judgement, that a CXR is required to ensure that it is safe to continue study drug administration (e.g., subjects with seroconversion on an annual TB test).
    - In this case, CXR should be performed as soon as restrictions allow at the study site or local hospital/facility. Otherwise, the CXR will be performed at the next earliest feasible visit.
  - 12-lead ECG, if the Investigator has determined, based on clinical judgement, that an ECG is required to ensure that it is safe to continue study drug administration In this case, ECG should be performed as soon as restrictions allow at the study site or local hospital/facility. Otherwise, the ECG will be performed at the next earliest feasible visit.
  - Local urine pregnancy test
  - Lab tests (blood chemistry, hematology, urinalysis)
  - $\circ$  ESR



All procedures performed at local facilities must be performed by appropriately qualified personnel.

- Lab draws should be obtained as close as possible to the scheduled visit.
- The study site should keep records of all visits/study activities performed virtually by phone/video or through the optional Home Healthcare Service or by a local clinic/hospital/laboratory.

# 5.3.1.1 Study Procedures

The study procedures outlined in Appendix D and Appendix F are discussed in detail in this section, with the exception of exploratory research and validation studies (discussed in Section 5.3.1.2), drug concentration measurements (discussed in Section 5.3.2), the collection of prior and concomitant medication information (discussed in Section 5.2.3), and the collection of AE information (discussed in Section 6.0). All study data will be recorded in source documents and on the appropriate eCRFs.

#### **Informed Consent**

At the Screening Visit, the subject will sign and date a study specific, IEC/IRB approved, informed consent form for the study (i.e., includes both Periods 1 and 2) before any study procedures are performed or any medications are withheld from the subject in order to participate in this study. Separate written consent will be required for each subject in order to participate in the optional exploratory research and validation studies. The separate written consent may be part of the main consent form. Subjects can withdraw informed consent at any time.

Details regarding how informed consent will be obtained and documented are provided in Section 9.3.

#### **Inclusion/Exclusion Criteria**

Subjects will be evaluated to ensure they meet all inclusion criteria and have none of the exclusion criteria at both Screening and Baseline Visits.



#### **Medical and Surgical History**

A complete non-RA-related medical and surgical history, including history of alcohol and nicotine use, will be taken from each subject during the Screening Visit. Additionally, a list of each subject's specific RA-related medical and surgical history will be recorded at Screening. History of herpes zoster, herpes zoster vaccination, and hepatitis B vaccination status will be recorded as part of the medical history. An updated medical history will be obtained prior to study drug administration at Baseline, to ensure the subject is still eligible for enrollment.

A detailed medical history with respect to TB risk factors will be documented in the study source documentation. This information will include BCG vaccination, cohabitation with individuals who have had TB, and travel to, residence in, or work in TB endemic locations.

#### **Patient Questionnaires**

Subjects will complete the following questionnaires as specified in Appendix D and Appendix F; a validated translation will be provided in their local language, as applicable:

#### Period 1

- Patient's Global Assessment of Disease Activity Visual Analog Scale (VAS) (Appendix J)
- Patient's Assessment of Pain VAS (Appendix K)
- Health Assessment Questionnaire Disability Index (HAQ-DI) to assess the physical function and health-related quality of life of each subject (Appendix L)
- Patient's Assessment of Severity and Duration of Morning Stiffness Numerical Rating Scale (NRS) (Appendix M)\*
- EuroQoL-5D-5L (EQ-5D-5L) (Appendix N)
- Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F)
   (Appendix O)



- Work Productivity and Activity Impairment (WPAI) (Appendix P)
- Short Form-36 (SF-36) (Appendix Q)

#### Period 2

- Patient's Global Assessment of Disease Activity VAS (Appendix J)
- Patient's Assessment of Pain VAS (Appendix K)
- HAQ-DI to assess the physical function and health-related quality of life of each subject (Appendix L)
- Patient's Assessment of Severity and Duration of Morning Stiffness NRS (Appendix M)\*
- \* Paper; all other patient-reported outcomes (PROs) collected electronically.

The subject should complete the questionnaires before site personnel perform any clinical assessments and before any interaction with site personnel has occurred to avoid biasing the subject's response.

Due to a state of emergency or pandemic situation like COVID-19, subject visits may be conducted via phone or video conference. In these situations, questionnaires will be completed by the subject at the next feasible visit.

#### TB Testing/TB Prophylaxis

The TB screening tests are diagnostic test results to be interpreted in the context of the subject's epidemiology, history, exam findings, etc., and it is the responsibility of the Investigator to determine if a subject has previous, active, or latent TB.

At Screening, all subjects will be assessed for evidence of increased risk for TB by a risk assessment form (Appendix I) and tested for TB infection by QuantiFERON-TB Gold test. The PPD skin test should be utilized only when a QuantiFERON-TB Gold test is not possible for any reason (unless both tests are required per local guidelines). The site staff will complete the TB risk assessment form and enter the data into an appropriate eCRF.



If a subject had a negative QuantiFERON-TB Gold (and/or PPD) test (or IGRA equivalent such as T-SPOT TB test) within 90 days prior to Screening and source documentation is available, the test does not need to be repeated, provided nothing has changed in the subject's medical history to warrant a repeat test. These cases may be discussed with the AbbVie Therapeutic Area Medical Director. The results of the TB test(s) will be retained at the site as the original source documentation.

For subjects with a negative TB test result at Screening or most recent evaluation, an annual TB re-test will be performed. The TB test(s) to be performed depends on local guidelines and whether or not the site has capacity to perform QuantiFERON-TB Gold testing (see below). If an annual TB test is newly positive (seroconversion), a chest x-ray (CXR) needs to be performed as soon as possible to aid in distinguishing active versus latent TB. Expert consultation can be considered per Investigator's discretion. Any positive TB test result after the patient has started study drug should be reported as an adverse event (AE).

#### TB Test:

- For regions that require both PPD and QuantiFERON-TB Gold testing, both will be performed. A positive TB test is defined by local guidelines (for example, in some countries, both PPD and QuantiFERON-TB Gold are performed, and if either one is positive, the TB test is considered positive).
- In the absence of local guidelines defining a positive result when both PPD and QuantiFERON-TB Gold tests are performed, then the QuantiFERON-TB Gold test result will be the TB test result (QuantiFERON supersedes PPD).
- If a site has the capacity to perform both PPD and QuantiFERON-TB Gold tests, and local guidelines require only one test to be performed, then the QuantiFERON-TB Gold is the preferred test. At a site with capacity to perform both tests, whatever TB test method (i.e., PPD or QuantiFERON-TB Gold or other IGRA) was performed at screening, then the subject should have their annual TB test performed with the same test method.
- If QuantiFERON-TB Gold test is NOT possible (or if both the QuantiFERON-TB Gold test and the PPD skin test are required per local



guidelines): the PPD skin test (also known as a TB skin test) will be performed according to standard clinical practice. The TB skin test should be read by a licensed healthcare professional between 48 and 72 hours after administration. A subject who does not return within 72 hours will need to be rescheduled for another skin test. The reaction will be measured in millimeters (mm) of induration and induration ≥ 5 mm for RA subjects is considered a positive reaction. The absence of induration will be recorded as "0 mm" not "negative." Subjects who have had an ulcerating reaction to the TB skin test in the past should not be re-exposed and the TB Skin Test should be considered positive with no requirement for subsequent testing with either PPD or QuantiFERON-TB Gold test.

- If the QuantiFERON-TB Gold test is indeterminate, then the investigator should perform a local QuantiFERON-TB Gold test (or through the central laboratory if not locally available) to rule out a positive test result. If testing remains indeterminate or is positive, then the subject is considered to be positive for the purpose of this study. If the testing result is negative, then the patient is considered to be negative.
- Interpretation of a positive annual TB test in low risk subjects: In cases where the QuantiFERON-TB Gold test by the central laboratory is positive and the Investigator considers the subject at low risk for TB and has no clinical suspicion of TB, the Investigator may perform a local QuantiFERON-TB Gold test (or repeat testing through the central laboratory if not locally available) to confirm the positive test result. If the repeat testing result is negative, the Investigator may consider the test to be negative based on his/her clinical judgment; if the repeat testing result is positive or indeterminate, the test is considered positive.
- An equivalent Interferon Gamma Release Assay (IGRA) (such as T-SPOT TB test) may be substituted for the QuantiFERON-TB Gold test.
- Subjects with documentation of prior positive result of QuantiFERON-TB Gold Test (or equivalent) and/or PPD are not required to repeat either test during the study and should be considered positive. Annual TB questionnaire should be completed for ALL subjects.



EudraCT 2015-003334-27

Subjects with a negative TB test and CXR not suggestive of active TB or prior TB exposure may be enrolled.

Subjects with a positive TB test must be assessed for evidence of active TB versus latent TB, including signs and symptoms and CXR. Subjects with no signs or symptoms and a CXR not suggestive of active TB may be enrolled after initiation of TB prophylaxis (see below). Subjects with evidence of active TB may not be enrolled.

#### TB Prophylaxis:

At Screening, if the subject has evidence of a latent TB infection (positive TB test and the subject has a CXR not suggestive of active TB), prophylactic treatment must be initiated at least 2 weeks prior to administration of study drug (or per local guidelines, whichever is longer). The prophylaxis needs to be completed; however, the full course of prophylaxis does not need to be completed prior to the first dose of study drug. If the Investigator deems that it is necessary, consultation with a TB expert could be considered.

#### Note: Rifampicin or Rifapentine is Not Allowed for TB prophylaxis

In Period 2, when study drug has been unblinded, rifampicin or rifapentine are allowed for TB prophylaxis for subjects not receiving upadacitinib.

Subjects with a prior history of latent TB that have documented completion of a full course of anti-TB therapy within 1 year prior to first study drug administration will be allowed to enter the study provided nothing has changed in the subject's medical history to warrant repeat treatment.

Obtain a CXR annually for subjects with newly identified TB risk factors as determined by the TB risk assessment form (Appendix I), or for subjects living in areas endemic for TB or for subjects with newly positive PPD or QuantiFERON-TB Gold test.

For subjects with seroconversion on an annual TB test, if a CXR cannot be done due to state of emergency or pandemic situation like COVID-19, the Investigator should contact



the AbbVie TA MD to determine if the subject may continue on study drug. CXR should be performed as soon as restrictions allow at the study site or local hospital/facility.

Subjects with a documented completion of a full course of anti-TB therapy greater than 1 year prior to first study drug administration may be allowed to enter the study only after consultation with the AbbVie Therapeutic Area Medical Director.

Newly initiated prophylactic treatment should be captured in the eCRF and in the source documents. Prior therapy should be captured in the eCRF.

During the study, subjects with new evidence of latent TB should initiate prophylactic treatment immediately per local guidelines. Study drug(s) should **not** be withheld and Isoniazid and/or rifampin/rifapentine should be initiated and 2 to 4 weeks later (per local guidelines), subject should be re-evaluated (unscheduled visit) for signs and symptoms of isoniazid toxicity.

In Period 2, when study drug has been unblinded, rifampicin or rifapentine are allowed for TB prophylaxis for subjects not receiving upadacitinib.

If the subject is experiencing signs or symptoms suspicious for TB or something has changed in the subject's medical history to warrant a repeat test before the next scheduled annual TB re-test, the case (including the TB test results) must be discussed with the AbbVie Therapeutic Area Medical Director.

# Chest X-Ray (CXR)

A CXR (posterior-anterior and lateral views) is required:

• For all subjects at Screening to rule out the presence of TB or other clinically relevant findings. The CXR will not be required if the subject had a previous normal CXR (posterior-anterior and lateral views) within 90 days of Screening, provided all source documentation is available at the site as outlined below and provided nothing has changed in the subject's medical history to warrant a repeat test.



 Annually for subjects with newly identified TB risk factors as determined by the TB risk assessment form (Appendix I) or for subjects living in areas endemic for TB or for subjects with newly positive PPD and/or QuantiFERON-TB Gold test.

Due to a state of emergency or pandemic situation like COVID-19, subject visits may be conducted via phone or video conference. In these situations, if a visit requires completion of a CXR, the CXR will be performed at the next earliest feasible visit, unless the Investigator has determined, based on clinical judgement, that a CXR is required to ensure that it is safe to continue study drug administration. In this case, CXR should be performed as soon as restrictions allow at the study site or local hospital/facility.

Subjects can have a repeat CXR at any time during the study as warranted, based on the opinion of the Investigator.

A radiologist or pulmonologist must perform an assessment of the CXR. The Principal Investigator will indicate the clinical significance of any findings and will sign and date the report. In the assessment of the CXR, the Principal Investigator or his/her delegate must indicate the presence or absence of (1) calcified granulomas, (2) pleural scarring/thickening, and (3) signs of active TB. If the CXR demonstrates changes suggestive of previous TB (e.g., calcified nodule, fibrotic scar, apical or basilar pleural thickening) or other findings that are clinically significant, the Principal Investigator should contact the AbbVie Therapeutic Area Medical Director before enrolling the subject.

#### 12-Lead ECG

For all subjects, a resting 12-lead ECG will be performed at Screening and every 48 weeks thereafter, as specified in Appendix D and Appendix F. A qualified physician will interpret the clinical significance of any abnormal finding, sign, and date each ECG. ECG with QT interval corrected for heart rate using Fridericia's correction formula (QTcF) should be reported (or calculated) and documented in the source documents and later transcribed on to the appropriate eCRF if QTcF prolongation is observed. A valid QTcF cannot be calculated in subjects who have a pacemaker or supraventricular or



ventricular conduction abnormalities. In case of QTcF prolongation, the baseline QTcF will need to be entered into the appropriate eCRF for comparison as well. In addition, any clinically significant findings will be documented in the source documents and later transcribed on to the appropriate eCRF. Each signed original ECG will be monitored by the responsible site monitor and kept with subject's source documents onsite.

For subjects with a normal ECG taken within 90 days of Screening, a repeat ECG at Screening will not be required, provided source documentation is available and provided nothing has changed in the subject's medical history to warrant a repeat test. If there are other findings that are clinically significant, the Investigator must contact the AbbVie Therapeutic Area Medical Director before enrolling the subject.

Subjects can have a repeat ECG at any time during the study as warranted, based on the opinion of the Investigator.

Due to a state of emergency or pandemic situation like COVID-19, subject visits may be conducted via phone or video conference. In these situations, if a visit requires completion of an ECG, the ECG will be performed at the next earliest feasible visit, unless the Investigator has determined, based on clinical judgement, that an ECG is required to ensure that it is safe to continue study drug administration. In this case, the ECG should be performed as soon as restrictions allow at the study site or local hospital/facility.

#### X-Rays of Hands and Feet

Detailed instructions for performing and transmitting the study related x-rays of hands and feet are provided in a separate Imaging Acquisition Guideline (IAG)/Site Operational Manual.

Handling of X-Rays of Hands and Feet at Screening

Screening x-rays of bilateral hands (posterior-anterior view) and bilateral feet (anteroposterior view) must be performed within the 35-day screening period.


Once a subject has been deemed eligible to participate and has had screening x-rays performed, the x-rays will be sent to the central imaging laboratory designated by the Sponsor. Digitalized images may be acceptable, provided that they meet the specifications outlined in the IAG/Site Operations Manual. X-rays not meeting the quality requirements must be repeated within the 35-day screening window. Subjects can receive the first dose of study drug if the x-rays have been determined to be of sufficient quality by the central imaging laboratory.

Screening x-rays of hands and feet will serve as baseline x-rays for scoring purposes.

Joint x-rays will be sent to the central imaging vendor designated by the Sponsor. The x-rays will only be assessed by the imaging vendor for erosions and joint space narrowing, and will not be assessed for any other clinically significant findings that may impact a subject's health.

Handling of X-Rays of Hands and Feet after Baseline

Handling of x-rays of hands and feet after baseline in Period 1 is illustrated in Figure 3.

All subjects (regardless of response) will receive Week 24 x-rays (Figure 3, box A) and Week 48 x-rays (Figure 3, box B).

If a subject prematurely discontinues from the study (withdrawal of informed consent), depending on the time of discontinuation, new x-rays might be needed.

- Subjects who prematurely discontinue before Week 12 will not get x-rays (Figure 3, box C)
- Subjects who prematurely discontinue from Week 12 to before Week 24 (≥ Week 12 and < Week 24), will have new x-rays performed (Figure 3, box D).
- Subjects who prematurely discontinue after Week 24 to before Week 36 (> Week 24 and < Week 36), will not have x-rays performed (Figure 3, box E).



• Subjects who prematurely discontinue from Week 36 to before Week 48 (≥ Week 36 and < Week 48), will have new x-rays performed (Figure 3, box F).

If a subject prematurely discontinues from study drug but continues to participate in the study, subject should follow the regular visit schedule as outlined in Appendix D and Appendix F, including performance of scheduled x-rays of hands and feet. However, depending on the time of study drug discontinuation in Period 1, new x-rays might be needed.

- Subjects who prematurely discontinue from study drug before Week 12 will not get new x-rays.
- Subjects who prematurely discontinue from study drug from Week 12 to Week 16 (≥ Week 12 and ≤ Week 16), will have new x-rays performed.
- Subjects who prematurely discontinue from study drug after Week 16 to Week 24 (> Week 16 and ≤ Week 24), will have x-rays performed at Week 24 (standard).
- Subjects who prematurely discontinue from study drug after Week 24 to Week 36 (> Week 24 and < Week 36), will not have new x-rays performed.
- Subjects who prematurely discontinue from study drug from Week 36 to Week 40 (≥ Week 36 and ≤ Week 40), will have new x-rays performed.
- Subjects who prematurely discontinue from study drug after Week 40 to Week 48 (> Week 40 and ≤ Week 48), will have x-rays performed at Week 48 (standard).

X-rays will be sent to the central imaging laboratory designated by the Sponsor. Digitalized images may be acceptable, provided that they meet the specifications outlined in the IAG/Site Operations Manual. X-rays not meeting the quality requirements must be repeated.

Overall in Period 1, each subject will undergo a maximum of 3 scheduled visits for x-ray examination of bilateral hands and feet (unless unscheduled repeat imaging is needed due



to failure to meet the quality requirements) at Screening, Week 24, and Week 48/PD. One additional x-ray examination of bilateral hands and feet may be needed depending on the time of premature study drug discontinuation for those subjects that continue the study.

In Period 2, a follow-up x-ray of hands and feet is planned at Week 96, Week 192, and Week 260. Subjects who prematurely discontinue from Period 2 will undergo an x-ray of hands and feet unless the previous x-ray was performed within the previous 24 weeks. Images will be sent to the central imaging laboratory designated by the Sponsor.

Due to a state of emergency or pandemic situation like COVID-19, subject visits may be conducted via phone or video conference. In these situations, if a visit by phone or video conference occurs at one of the designated study visits specified to complete x-rays of hands and feet, it will be performed at the next earliest feasible visit.

Upadacitinib 7.5 mg QD + MTX 10 mg/week (7.5 mg/week for Japan 2 only) Upadacitinib 7.5 mg QD+ optimized meds Upadacitinib 7.5 mg QD Upadacitinib 7.5 mg QD (n=75) randomization for subjects in Japan JAPAN ONLY Upadadtinib 15 mg QD 3 1:1:1-randomization globally MTX 10 mg/week (7.5 mg/week for Japan Upadadtinib 15 mg QD+ optimized meds Upadacitinib 15 mg QD Upadacitinib 15 mg QD GLOBAL JAPAN ONLY Upadacitinib 30 mg QD 3 + MTX 10 mg/week (7.5 mg/week for Japan Upadacitinib 30 mg QD + optimized meds Upadacitinib 30 mg QD 1 Upadacitinib 30 mg QD (n=37) GLOBAL JAPAN ONLY 3 MTX + Upadacitinib 7.5 mg, 15 mg, or 30 mg 2 덮 (2:1:1) (titrate to 20 mg) MTX + optimized meds (titrate to 15 mg) 1 (n=263) (n=37) MTX GLOBAL JAPAN ONLY W24 W26 Screen Baseline (B) Week 48 x-rays (A) Week 24 x-rays for ALL patients for ALL patients (C) No x-rays for PD (D) New x-rays for PD (E) No x-rays for PD (F) New x-rays for PD > W24 and < W36 ≥ W12 and < W24 hefore W12 > W36 and < W48

Figure 3. Handling of X-Rays of Hands and Feet after Baseline (Period 1)

MTX = methotrexate; n = number; PD = premature discontinuation; QD = once daily; SJC = swollen joint count; TJC = tender joint count; W = week

\* Subjects who prematurely discontinue from the study drug from Week 12 to Week 16 (≥ Week 12 and ≤ Week 16) or from Week 36 to Week 40 (≥ Week 36 and ≤ Week 40), but continue to participate in the study will have new x-rays performed.

#### **Height and Weight**

Height will be measured at the Screening Visit only (with shoes off). Body weight will be measured at all scheduled visits as specified in Appendix D and Appendix F. All measurements will be recorded in metric units where applicable.



Upadacitinib M13-545 Protocol Amendment 8 EudraCT 2015-003334-27

## Vital Signs

Vital sign determinations of systolic and diastolic blood pressure in sitting position, pulse rate, respiratory rate, and body temperature will be obtained at visits specified in Appendix D and Appendix F. Blood pressure, pulse rate, body temperature, and respiratory rate should be performed before blood draws are performed.

#### **Physical Examination**

A complete physical examination will be performed at the designated study visits as specified in Appendix D and Appendix F. The physical examination at the Baseline Visit will serve as the baseline physical examination for the entire study. Physical examination abnormalities noted by the Investigator at Baseline prior to the first dose of study drug will be recorded in the subject's medical history; abnormalities noted after the first dose of study drug will be evaluated and documented by the Investigator as to whether or not the abnormality is an AE (see Section 6.1.1.1 for AE definition). All findings whether related to an AE or part of each subject's medical history will be captured on the appropriate eCRF page.

Due to a state of emergency or pandemic situation like COVID-19, subject visits may be conducted via phone or video conference. In these situations, if a visit by phone or video conference occurs at one of the designated study visits specified to complete physical examination, the complete physical examination will be performed at the next feasible visit.

At any time, a symptom-directed physical examination can be performed as deemed necessary by the Investigator.

#### Physician Global Assessment of Disease Activity VAS

At visits specified in Appendix D and Appendix F, the Physician will rate global assessment of subject's current disease activity ranging from 0 to 100 independent of the subject's self-assessment using the VAS, which consists of a horizontal 100 mm line



anchored at either end by opposite adjectives reflecting the spectrum/severity of the parameters assessed (Appendix G).

Due to a state of emergency or pandemic situation like COVID-19, subject visits may be conducted via phone or video conference. In these situations, the Physician Global Assessment of Disease Activity will be completed by the physician at the next feasible visit.

## TJC and SJC Assessment

TJC Assessment

An assessment of 68 joints (Appendix H) will be done for tenderness by pressure manipulation on physical examination at visits specified in Appendix D and Appendix F. Joint pain/tenderness will be classified as: present ("1"), absent ("0"), replaced ("9") or no assessment ("NA").

SJC Assessment

An assessment of 66 joints (Appendix H) will be done by directed physical examination at visits specified in Appendix D and Appendix F. The joints to be examined for swelling are the same as those examined for tenderness, except the hip joints are excluded. Joint swelling will be classified as present ("1"), absent ("0"), replaced ("9") or no assessment ("NA").

Any injected joints will be considered as "not assessed" ("NA") for 3 months from the time of the intra-articular injection.

If possible, the TJC and SJC should be performed by an independent and blinded joint assessor who should not perform any other study related procedures.

In order to minimize variability, the same independent joint assessor should evaluate the subject at each visit for the duration of the trial as much as possible. A back-up independent joint assessor should be identified. The independent joint assessors should



be a qualified medical professional (e.g., nurse, physician's assistant, physician). Any other joint assessor must be trained and competent in performing such assessments. It is the responsibility of the Investigator to ensure that all assessors are qualified and trained to perform joint assessments. If the independent assessor is not available, the pre-identified back-up assessor should perform such assessments.

Due to a state of emergency or pandemic situation like COVID-19, subject visits may be conducted via phone or video conference. In these situations, the TJC and SJC will be performed at the next feasible visit by the independent joint assessor, if possible.

#### **CDAI**

The CDAI calculation is required to determine if a subject fails to achieve Clinical Remission at the Week 26 visit. An Interactive Response Technology (IRT) will calculate CDAI with input from site personnel on joint counts and the subject's and physician's Global Assessment of RA Disease Activity score. A worksheet will be provided to capture the components required for IRT entry to obtain the CDAI calculation.

The calculation used to determine CDAI score at Week 26 is as follows:

$$CDAI = TJC28 + SJC28 + PtGA + PhGA$$

NOTE: As described in the section pertaining to Rescue Therapy, the Investigator should optimize background RA therapies in subjects who fail to achieve a CDAI  $\leq$  2.8 at Week 26, but achieve at least 20% improvement in both TJC and SJC.

#### **Pregnancy Test**

A serum pregnancy test will be performed for all women of child bearing potential at the Screening Visit. The serum pregnancy test will be sent to and performed by the central laboratory. If the serum pregnancy test is positive the subject is considered a screen failure. If the serum pregnancy test is borderline, it should be repeated  $\geq 3$  days later to determine eligibility. If the repeat serum pregnancy test is:



- Positive, the subject is considered a screen failure;
- Negative, the subject can be enrolled into the trial;
- Still borderline,  $\geq 3$  days later, this will be considered documentation of continued lack of a positive result and the subject can be enrolled into the trial.

In Period 1, a urine pregnancy test will be performed for all women of childbearing potential at the Baseline Visit prior to the first dose of study drug and at all subsequent visits. More frequent pregnancy tests will be performed throughout the study if required per local/country requirements.

- If the baseline urine pregnancy test performed at the site is negative, then dosing with study drug may begin. If the baseline urine pregnancy test performed at the site is positive, dosing with study drug must be withheld and a serum pregnancy test is required. The serum pregnancy test will be sent to and performed by the central laboratory. If the serum pregnancy test is positive, study drug must be permanently discontinued. In the event a pregnancy test comes back borderline, a repeat test is required.
- If a urine pregnancy test post baseline is positive, study drug needs to be temporarily discontinued and a serum pregnancy test is required. The serum pregnancy test will be sent to and performed by the central laboratory. If the serum pregnancy test is negative, study drug may be restarted. If the serum pregnancy test is positive, study drug must be permanently discontinued.

In Period 2, for women of childbearing potential, a urine pregnancy test will be performed at all visits and monthly at home between scheduled study visits. The results of the monthly at home tests will be communicated to the site. If a urine pregnancy test is positive, the subject must stop dosing, return to the study site and have blood drawn for a serum pregnancy test that will be analyzed at the central laboratory.

In the event a urine pregnancy test may not be performed at the protocol specified visits due to study modifications related to a state of emergency or pandemic situation like COVID-19, it can be performed by subjects at a local laboratory or it is possible for the Investigator to arrange a shipment from the study site directly to the subject's home of



urine pregnancy test kits to have the urine pregnancy test done at home (see Section 5.3.1.1 - Sub-Section "Study Drug Dispensing, Dosing, and Compliance" for details). Home urine pregnancy test should be performed monthly, regardless of ability to obtain other laboratory samples.

At each visit, the study staff should review the pregnancy avoidance recommendations with each subject of childbearing potential and male subjects receiving MTX with a partner of childbearing potential, and document this discussion in the subject's source records.

If during the course of the study a woman becomes surgically sterile or post-menopausal and complete documentation as described in Section 5.2.4 is available, pregnancy testing is no longer required.

A pregnant or breastfeeding female will not be eligible for participation in this study or be allowed to continue study drug.

#### **Clinical Laboratory Tests**

Samples will be obtained for the clinical laboratory tests listed in Table 2. Unscheduled clinical labs may be obtained at any time during the study if deemed appropriate per Investigator's discretion. A certified central laboratory will be utilized to process and provide results for the clinical laboratory tests. All abnormal laboratory tests that are considered clinically significant by the Investigator will be followed to a satisfactory resolution.

The central laboratory chosen for this study will provide instructions regarding the collection, processing, and shipping of these samples.

If travel restrictions or other changes in local regulations due to state of emergency or pandemic situation like COVID-19 prevent the subject from having blood drawn for laboratory testing at the study site, it is possible for the Investigator to arrange for subjects to have laboratory work done at a local lab, hospital, or other facility to ensure the safety



assessments are conducted per protocol. Local lab results should be obtained along with reference ranges and kept within the subjects' source documentation. Local lab results should be reviewed by the investigator or designee as soon as possible and documented in the eCRF.

If laboratory samples cannot be obtained, study drug administration may be continued provided labs have been obtained within the prior 3 months, the investigator has reviewed the laboratory results and confirmed and discussed with the subject that there is no safety concern for the subject to continue use of the study drug in the absence of current lab results. The subject should be scheduled for laboratory draws as soon as feasible and no later than the next scheduled visit in order to continue the study drug administration.

If laboratory results are not available within the prior 3 months/two consecutive 12-week intervals, study drug dispensation is not allowed until the required laboratory tests are completed to ensure the safety assessments are conducted per protocol.

Blood samples will be obtained for the laboratory tests at visits specified in Appendix D and Appendix F. Blood draws should be performed only after all questionnaires (HAQ-DI, Patient's Assessment of Pain, etc.), clinical assessments, and vital sign determinations are obtained.

For clinic visits where samples for serum chemistry tests are collected, subjects should be fasting (a minimum 8-hour fast) whenever possible. If a subject is not able to fast when necessary, due to unforeseen circumstances, the non-fasting status will be recorded in study source documentation.

Urine samples will be obtained for urinalysis testing at visits specified in Appendix D and Appendix F. The central laboratory will be responsible for performing a macroscopic urinalysis (urine dipstick) on the collected urine specimens. Specified abnormal macroscopic urinalyses defined as leukocytes, nitrite, protein, ketones, or blood greater than negative, or glucose greater than normal will be followed up with a microscopic analysis at the central laboratory.



For any laboratory test value outside the reference range that the Investigator considers to be clinically significant, the Investigator should apply the standard of care for medical evaluation and treatment per local guidelines:

- The Investigator will repeat the test to verify the out-of-range value.
- The Investigator will follow the out-of-range value to a satisfactory clinical resolution.

A laboratory test value that requires a subject to be discontinued from study drug or requires a subject to receive treatment will be recorded as an AE.

Table 2. Clinical Laboratory Tests

| Hematology<br>(Central Lab) | Clinical Chemistry <sup>a</sup><br>(Central Lab) | Urinalysis <sup>b</sup><br>(Central Lab) | Other Laboratory Tests |
|---|---|---|---|
| Hematocrit Hemoglobin RBC count WBC count Neutrophils Bands Lymphocytes Monocytes Basophils Eosinophils Platelet count | BUN Creatinine Total bilirubin INR (reflex only) <sup>c</sup> ALT AST Alkaline phosphatase CPK Sodium Potassium Chloride Bicarbonate Calcium Inorganic phosphate Uric acid Cholesterol LDL-C HDL-C Total protein Glucose Triglycerides Albumin | Specific gravity Ketones pH Protein Blood Glucose Urobilinogen Bilirubin Leukocytes Nitrites Microscopic examination, if needed | Central Lab Tests: Serum pregnancy (bHCG) test <sup>d</sup> HBs Ag <sup>e</sup> HBs Ab <sup>e</sup> HBc Ab <sup>e</sup> HBV DNA PCR (reflex only) <sup>e</sup> HCV Ab <sup>e</sup> HCV RNA reflex only <sup>e</sup> QuantiFERON-TB Gold <sup>f</sup> Rheumatoid Factor <sup>e</sup> Anti-CCP autoantibodies <sup>e</sup> hs-CRP <sup>g</sup> IgG and IgM FSH <sup>h</sup> VZV specific IgG <sup>i</sup> Beta-D-Glucan <sup>i</sup> Local Lab Tests: Urine pregnancy test <sup>j</sup> ESR |
| | | | HIV (if required) <sup>k</sup> |



## Table 2. Clinical Laboratory Tests (Continued)

ALT = alanine aminotransferase; AST = aspartate aminotransferase; bHCG = beta human chorionic gonadotropin;

BUN = blood urea nitrogen; CCP = cyclic citrullinated peptide; CPK = creatine phosphokinase;

DNA = deoxyribonucleic acid; ESR = erythrocyte sedimentation rate; FSH = follicle stimulating hormone;

HBc Ab = hepatitis B core antibody; HBs Ab = hepatitis B surface antibody; HBs Ag = hepatitis B surface antigen;

HBV = hepatitis B virus; HCV Ab = hepatitis C virus antibody; HDL-C = high-density lipoprotein cholesterol;

HIV = human immunodeficiency virus; hsCRP = high-sensitivity C-reactive protein; IgG = immunoglobulin G;

IgM = immunoglobulin M; INR = international normalized ratio; LDL-C = low-density lipoprotein cholesterol;

PCR = polymerase chain reaction; RBC = red blood cell; RNA = ribonucleic acid; TB = tuberculosis; WBC = white blood cell; VZV = varicella zoster virus

- a. Minimum 8-hour fast. If a subject is not able to fast when necessary, due to unforeseen circumstances, the non-fasting status will be recorded in study source documentation.
- b. A urine dipstick macroscopic urinalysis will be completed by the central laboratory at all required visits. A microscopic analysis will be performed in the event the dipstick results show leukocytes, nitrite, protein, ketones, or blood greater than negative or glucose greater than normal.
- c. INR will only be measured with a separate blood sample at repeat testing if ALT and/or AST > 3 × ULN.
- d. A serum pregnancy test will be performed for all women of childbearing potential at the Screening Visit and if post baseline urine pregnancy test turns positive.
- e. HBV DNA testing is required for subjects who meet specific toxicity management criteria (See ALT/AST toxicity management criteria in Table 4).
- f. If PPD not performed.
- g. Central lab hsCRP results will remain blinded to the Sponsor, Investigator, study site personnel, and subject for all visits except Screening. Results of tests such as hsCRP may be blunted in subjects taking a JAK inhibitor, thereby limiting the clinical utility of these tests in the setting of a possible safety assessment or adverse event management. Any local hsCRP or local CRP tests should not be reported to the investigator until treatment allocation is unblinded.
- h. For more details, please refer to Section 5.2.4 (Contraception Recommendations).
- i. At Screening for subjects in Japan only.
- j. A urine pregnancy test will be performed for all women of childbearing potential at the Baseline Visit prior to the first dose of study drug and all subsequent visits. If the baseline urine pregnancy test performed at the site is negative, then dosing with study drug may begin. If the baseline urine pregnancy test performed at the site is positive, dosing with study drug must be withheld and a serum pregnancy test is required. The serum pregnancy test will be sent to and performed by the central laboratory. If the serum pregnancy test is positive, study drug must be permanently discontinued. In the event a pregnancy test comes back borderline, a repeat test is required. If a urine pregnancy test post baseline is positive, study drug needs to be temporarily discontinued and a serum pregnancy test is required. The serum pregnancy test will be sent to and performed by the central laboratory. If the serum pregnancy test is positive, study drug must be permanently discontinued.
- k. If required by country regulatory authorities to confirm eligibility, subjects will be tested for antibodies to HIV at Screening, and it should be documented that the test has been performed. This testing is to be done at a local lab. A subject will not be eligible for study participation if test results indicate a positive HIV infection. AbbVie will not receive results from the testing and will not be made aware of any positive result.



## **Hepatitis Screen**

All subjects will be tested for the presence of HBV and HCV at Screening.

Hepatitis B:

Subjects will be tested for the presence of HBV at Screening using the following tests:

- HBs Ag (Hepatitis B surface antigen)
- HBc Ab/anti-HBc (Hepatitis B core antibody)
- HBs Ab/anti-HBs (Hepatitis B surface antibody)

A positive result for HBs Ag will be exclusionary.

A negative result for HBs Ag will be tested (automatic reflex testing) for core antibodies (HBc Ab) and surface antibodies (HBs Ab).

- A negative test result for HBc Ab does **not** require HBV DNA PCR qualitative testing and the subject may be enrolled (Figure 4, Scenarios A and B).
- For a subject who has had a HBV vaccination (should document in the medical history), a positive test result for HBs Ab is expected and the subject may be enrolled (Figure 4, Scenario B).\*
- A positive test result for HBc Ab requires HBV DNA PCR testing (automatic reflex testing) (Figure 4, Scenarios C and D).
  - A positive result for HBV DNA or a result that exceeds detection sensitivity will be exclusionary.
  - A subject with a negative result for HBV DNA may be enrolled.
- For subjects in Japan only: A positive result for HBs Ab/anti-HBs requires HBV DNA PCR testing.
  - A positive result for HBV DNA or a result that exceeds detection sensitivity will be exclusionary.
  - A subject with a negative result for HBV DNA may be enrolled.

Figure 4. Criteria for HBV DNA PCR Qualitative Testing



\* For subjects who have had a HBV vaccination (should document in the medical history), a positive test result for HBs Ab is expected and these subjects may be enrolled.

## Hepatitis C:

Blood samples for Hepatitis C serology will be obtained at the Screening Visit. A subject will not be eligible for study participation if test results indicate active Hepatitis C (HCV RNA detectable in any subject with anti HCV Ab).

## **HIV**

Subjects with a known history of HIV infection are excluded from study participation. If required by country regulatory authorities to confirm eligibility, subjects will be tested for antibodies to HIV at Screening. This testing is to be done at a local lab. A subject will not be eligible for study participation if test results indicate a positive HIV infection. AbbVie will not receive results from the testing and will not be made aware of any positive result.



#### **VZV** (For Subjects in Japan Only)

Tests for varicella-zoster virus (VZV) will be performed at Screening to evaluate immunity of a subject to VZV for better understanding of the safety profile of upadacitinib.

To assess the cell-mediated immune status to VZV, a skin test using the VZV antigen will be performed. VZV antigen is injected intradermally into the forearm of each subject, and the longest diameters of erythema and edema will be measured in millimeters (mm) between 24 (recommended) and 48 hours after the injection and recorded on the appropriate eCRF page along with date and time of injection and measurement. The absence of erythema or edema will be recorded as "0 mm."

Blood samples will be used for measuring IgG-class antibodies specific to VZV to estimate the prior exposure to VZV of the subject.

## Randomization/Drug Assignment

All Screening laboratory results must be reviewed, signed, and dated by the Principal Investigator or Sub-investigator prior to the Baseline Visit. Subjects will not be enrolled into the study if laboratory or other Screening result abnormalities are deemed clinically significant by the Principal Investigator or Sub-investigator.

Subjects will be eligible for randomization if they continue to meet all of the selection criteria (Section 5.2) at Baseline and are willing to continue in the study.

Subjects will be randomized in a 1:1:1 ratio using interactive response technology (IRT) to treatment Groups 2, 3, and 4, below, except for subjects from Japan, who will be randomized in a 2:1:1:1 ratio to Groups 1, 2, 3, and 4:

- Group 1: Upadacitinib 7.5 mg QD monotherapy (subjects in Japan only; N = 75)
- Group 2: Upadacitinib 15 mg QD monotherapy (N = 300) (includes 37 subjects from Japan)



- Group 3: Upadacitinib 30 mg QD monotherapy (N = 300) (includes 37 subjects from Japan)
- Group 4: MTX monotherapy (N = 300) (includes 37 subjects from Japan)

Randomization will be stratified by geographic region.

See Section 5.5.3 for details.

#### Study Drug Dispensing, Dosing, and Compliance

Study drug(s) will be dispensed to subjects beginning at Baseline (Day 1) and as specified in Appendix D and Appendix F. The first dose of study drug(s) will be administered after all other Baseline (Day 1) procedures are completed. Subjects will maintain a dosing diary for all study drug(s) administered outside of the study visit (i.e., at home) to capture dosing dates and times. At visits specified in Appendix D and Appendix F, the site personnel will review and retain a copy of the dosing diary, returned study drug kits, and empty study drug packaging to verify compliance.

To maintain the blind in this study with two blinded investigational study drugs (MTX and upadacitinib), each subject will be instructed to take two capsules once weekly (MTX and/or matching placebo) and a tablet once daily (upadacitinib or matching placebo). MTX and matching placebo will be distributed as identical capsules to maintain blinding during the MTX titration and during the rest of the study. Starting with Amendment 6 subjects receiving MTX will receive open-label MTX tablets in quantities sufficient to cover their respective dose.

Determination of which subjects are assigned to receive MTX-placebo versus upadacitinib placebo will be via the IRT (Interactive Response Technology), which will randomly assign each subject to the appropriate treatment group in a blinded manner.

All relevant dosing information will be entered into the eCRF at each visit.

(Refer to Section 5.5 for additional information.)



Study drug may be shipped from the study site directly to the study subject's home due to study modifications related to a state of emergency or pandemic situation like COVID-19 if all the following criteria are met:

- Direct-to-patient (DTP) shipment of study drug is allowed by local regulations and the relevant ethics committee
- Subject agrees to have the study drug shipped directly to their home
- Shipments may also include other study supplies (e.g., drug dosing diaries, inhome urine pregnancy test kits). Instructions will be provided by AbbVie as to how a study site can initiate a DTP shipment using Marken, a global vendor selected by AbbVie to provide this service when necessary. Shipments of study drugs from the study site to a subject's home will be appropriately temperature controlled (qualified shipper or temperature monitoring) within the labeled storage conditions. Signature is required upon delivery; due to COVID-19 related social distancing, this may be provided by the courier after delivery. Documentation of the shipment is to be retained by the clinical site.
- AbbVie will not receive subject identifying information related to these shipments, as the site will work directly with the courier.

The study site is responsible for meeting IRB/IEC reporting requirements related to DTP shipments of study drug, and for obtaining consent to provide delivery information to the courier and documenting this consent in source documents.

# Optional Home Healthcare Service Due to State of Emergency or Pandemic Situation like COVID-19

Subjects may be offered the option of home healthcare visits provided by a study nurse or third-party vendor. Study procedures conducted in the home setting may include vital signs and body weight, physical exam, blood and urine samples collection, urine pregnancy test, adverse event and concomitant therapy assessment including compliance to contraception requirements if applicable, latent TB risk assessment form, review of subject dosing diary, TJC and SJC performed by the same independent joint assessor, if possible, to minimize variability.



This option can only be offered in countries and sites that comply with local regulatory and IRB/IEC requirements for homecare. Any pre-requisite submissions or notifications to the site IRB/IEC and local competent health authority should be made, and approvals must be obtained prior to implementation.

The investigator should be available via phone call if a consultation is necessary.

It is recommended that medical personnel entering a subject's home adhere to local health regulations during the COVID-19 pandemic, such as the use of Personal Protective Equipment (PPE), as required.

If the home visits will not be performed by site personnel, the site may be responsible for selecting a vendor, contracting with a vendor, and for ensuring continued compliance with the terms of the Clinical Study Agreement.

Individuals performing home visits need to be added to the delegation log.

# 5.3.1.2 Collection and Handling of Optional Samples for Exploratory Research and Validation Studies

In Period 1, subjects will have the option to provide samples for exploratory research and validation studies. Subjects may still participate in the study even if they decide not to participate in this optional exploratory research/validation study.

Exploratory research can help to improve our understanding of how individuals respond to drugs and our ability to predict which subjects would benefit from receiving specific therapies. In addition, exploratory research may help to improve our understanding of how to diagnose and assess/monitor RA by assessing associations between disease characteristics, outcomes data, and biomarkers of interest.

Validation studies, including those related to the development of potential in vitro diagnostic tests, may be carried out retrospectively in order to assess associations between events of interest (i.e., efficacy and/or safety events) and candidate biomarkers.



AbbVie (or people or companies working with AbbVie) will store the biomarker exploratory research/validation studies samples in a secure storage space with adequate measures to protect confidentiality. The samples will be retained while research on upadacitinib (or drugs of this class) or RA and related conditions continues, but for no longer than 20 years after the completion of Period 1.

## **DNA Samples for Pharmacogenetic or Epigenetic Analyses**

Whole blood samples for DNA isolation will be collected at the visits indicated in Appendix E from each subject who consents to provide samples for exploratory/validation research. The procedure for obtaining and documenting informed consent is discussed in Section 9.3.

Samples will be shipped frozen to AbbVie or a designated laboratory for DNA extraction and/or long-term storage or analyses. Instructions for the preparation and shipment of the pharmacogenetic and/or epigenetic research samples will be provided in a laboratory manual.

#### RNA Samples for Transcriptomic and/or Epigenetic Analyses

Whole blood samples for RNA isolation will be collected at the visits indicated in Appendix E from each subject who consents to provide samples for exploratory/validation research. The procedure for obtaining and documenting informed consent is discussed in Section 9.3.

Samples will be shipped to AbbVie or a designated laboratory for RNA extraction and/or long-term storage or analyses. Instructions for the preparation and shipment of the samples will be provided in a laboratory manual.

# Serum and Plasma Samples for Systemic Analyses, Including but Not Limited to Proteomic and Metabolomic

Serum and plasma samples will be collected at the visits indicated in Appendix E from each subject who consents to provide samples for exploratory/validation research. These



samples may be used for assay of study drugs if needed. The procedure for obtaining and documenting informed consent is discussed in Section 9.3.

Samples will be shipped to AbbVie or a designated laboratory for long-term storage and/or analyses. Instructions for the preparation and shipment of the samples will be provided in a laboratory manual.

## 5.3.2 Drug Concentration Measurements

## 5.3.2.1 Collection of Samples for Analysis

Blood samples for assay of upadacitinib and possibly other medications will be collected as follows:

- At Weeks 2 and 4 prior to dosing;
- At Weeks 12, 16, 20, 24, 32, 36, 40, and 48/PD at any time during the visit.

On Week 2 and Week 4 Visit days, if possible, subjects should take the study drug dose at the clinic after collecting the pharmacokinetic (PK) blood sample, except if the subjects regularly take the study drug dose at night. Those subjects who regularly take the study drug dose at night should continue to take study drug according to their normal schedule. For all other visits, subjects can take the study drug dose on visit days at their regular schedule and not necessarily at the clinic.

The date and accurate time of the PK sample collection will be recorded on the lab requisition form. The date and accurate time of the last two study drug doses will be recorded on the eCRF to the nearest minute.

Refer to the study specific laboratory manual for detailed instructions on sample collection, processing, and shipment.



#### 5.3.2.2 Measurement Methods

Plasma concentrations of upadacitinib will be determined by the Drug Analysis Department at AbbVie using a validated liquid chromatography/mass spectrometry method.

- 5.3.3 Efficacy Variables
- 5.3.3.1 Period 1 Variables

## 5.3.3.1.1 Primary Variables

The primary endpoint in Period 1 is the proportion of subjects achieving ACR50 response at Week 12 (US/FDA regulatory purposes) or the proportion of subjects achieving Clinical Remission (CR) (EU/EMA regulatory purposes) at Week 24. For Japan/PMDA regulatory purposes, the primary endpoints are the proportion of subjects achieving ACR20 response at Week 12 and change from baseline in modified Total Sharp Score (mTSS) at Week 24. Analyses will be conducted separately for US/FDA, EU/EMA and Japan/PMDA regulatory purposes; the primary endpoint is specified separately for each set of analyses.

ACR20/50 response rate will be determined based on 20%/50% or greater improvement in TJC and SJC and ≥ 3 of the 5 measures of Patient's Assessment of Pain (VAS), Patient's Global Assessment of Disease Activity (VAS), Physician's Global Assessment of Disease Activity (VAS), HAQ-DI, or hsCRP.

CR is defined as Disease Activity Score (DAS)28 (C-reactive protein [CRP]) < 2.6. DAS28 (CRP) score will be determined based on a continuous scale of combined measures of TJC, SJC, Patient's Global Assessment of Disease Activity (PtGA) (in mm), and hsCRP (in mg/L) at Week 24.

DAS28 (CRP) = 
$$0.56 \times \sqrt{\text{TJC28*}} + 0.28 \times \sqrt{\text{SJC28**}} + 0.36 \ln(\text{hsCRP*} + 1) + 0.014 \times \text{PtGA*} + 0.96$$

\* TJC28 refers to the Subject's total Tender Joint Count out of the provided 28 evaluated joints.



- \*\* SJC28 refers to the Subject's total Swollen Joint Count out of the provided 28 evaluated joints.
- & hsCRP refers to the high-sensitivity c-reactive protein lab value. hsCRP unit in the DAS28 (CRP) equation is expressed as mg/L.
- » PtGA refers to the Patient's Global Assessment of Disease Activity. where  $\sqrt{}$  is square root and ln is natural log.

Modified Total Sharp Score (mTSS) is the van der Heijde mTSS.

## 5.3.3.1.2 Key Secondary Variables

Ranked key secondary endpoints for US/FDA regulatory purposes are:

- 1. Change from baseline in DAS28 (CRP) at Week 12;
- 2. Change from baseline in HAQ-DI at Week 12;
- 3. Change from baseline in modified Total Sharp Score (mTSS) at Week 24;
- Proportion of subjects achieving Low Disease Activity (LDA) based on DAS28 (CRP) ≤ 3.2 at Week 12;
- 5. Proportion of subjects achieving CR based on DAS28 (CRP) < 2.6 at Week 24;
- 6. Change from baseline in Short Form-36 (SF-36) Physical Component Score (PCS) at Week 12.

Ranked key secondary endpoints at Week 24 for EU/EMA regulatory purposes are:

- 1. Change from baseline in DAS28 (CRP);
- 2. Change from baseline in HAQ-DI;
- 3. ACR50 response rate;
- 4. Change from baseline in modified Total Sharp Score (mTSS);
- 5. Proportion of subjects achieving LDA based on DAS28 (CRP)  $\leq$  3.2;
- 6. Change from baseline in SF-36 PCS;



7. Proportion of subjects with no radiographic progression (defined as change from baseline in mTSS ≤ 0) at Weeks 24.

Ranked key secondary endpoints for Japan/PMDA regulatory purposes are:

- 1. Change from baseline in DAS28 (CRP) at Week 12;
- 2. Change from baseline in HAQ-DI at Week 12;
- 3. Proportion of subjects achieving LDA based on DAS28 (CRP)  $\leq$  3.2 at Week 12;
- 4. Proportion of subjects achieving CR based on DAS28 (CRP) < 2.6 at Week 24;
- 5. Change from baseline in SF-36 PCS at Week 12.

Other key secondary endpoints for US/FDA regulatory purposes are:

- 1. ACR20 response rate at Week 12;
- 2. ACR70 response rate at Week 12;
- 3. Proportion of subjects with no radiographic progression at Week 24.

Other key secondary endpoints for EU/EMA regulatory purposes are:

- 1. ACR20 response rate at Week 24;
- 2. ACR70 response rate at Week 24.

Other key secondary endpoints for Japan/PMDA regulatory purposes are:

- 1. ACR50 response rate at Week 12;
- 2. ACR70 response rate at Week 12;
- 3. Proportion of subjects with no radiographic progression at Week 24.

ACR20/50/70 response rates will be determined based on 20%/50%/70% or greater improvement in TJC and SJC and ≥ 3 of the 5 measures of Patient's Assessment of Pain (VAS), Patient's Global Assessment of Disease Activity (VAS), Physician's Global Assessment of Disease Activity (VAS), HAQ-DI, and hsCRP.

#### 5.3.3.1.3 Additional Variables

Additional endpoints at all visits are:

- ACR20/50/70 response rates at all visits;
- Change from baseline in individual components of ACR response at all visits;
- Change from baseline in DAS28(CRP) and DAS28 (erythrocyte sedimentation rate [ESR]) at all visits;
- Change from baseline in CDAI and SDAI at all visits;
- Proportion of subjects achieving LDA or CR by DAS28(CRP), DAS28(ESR), Simplified Disease Activity Index (SDAI), and Clinical Disease Activity Index (CDAI) at all visits (see below);
- Change from baseline in morning stiffness (severity and duration) at all visits;
- Proportion of subjects with change from baseline in HAQ-DI ≤ -0.22 at all visits;
- Proportion of subjects with change from baseline in HAQ-DI  $\leq$  -0.3 at all visits;
- ACR/EULAR Boolean remission at all visits.

| | DAS28 (CRP) and DAS28 (ESR) | SDAI | CDAI |
|-----|-----------------------------|--------|-------|
| LDA | ≤ 3.2 | ≤ 11.0 | ≤ 10 |
| CR | < 2.6 | ≤ 3.3 | ≤ 2.8 |

Additional endpoints (at Weeks 12, 24, and 48) are:

- Change from baseline in EQ-5D-5L;
- Change from baseline in FACIT-F;
- Change from baseline in WPAI;



• Change from baseline in SF-36.

Additional endpoints (at Weeks 24 and 48) are:

- Change from baseline in mTSS;
- Proportion of subjects with no radiographic progression (defined as change from baseline in mTSS ≤ 0);
- Change from baseline in radiographic joint space narrowing and erosion scores.

#### 5.3.3.2 Period 2 Variables

Assessments to evaluate efficacy of treatment in Period 2 will be analyzed for the following measures at Weeks 60, 72, 84, 96, every 12 weeks through Week 240, and Week 260/PD:

- ACR20/50/70 response rates;
- Change from baseline in individual ACR components;
- Change from baseline in DAS28 (CRP);
- Change from baseline in DAS28 (ESR);
- Change from baseline in CDAI and SDAI;
- Proportion of subjects achieving LDA and proportion of subjects achieving CR based on DAS28 (CRP), DAS28 (ESR), SDAI, and CDAI criteria (as defined for Period 1);
- Change from baseline in morning stiffness (severity and duration);
- Proportion of subjects with change from baseline in HAQ-DI  $\leq$  -0.22;
- Proportion of subjects with change from baseline in HAQ-DI  $\leq$  -0.3;
- ACR/EULAR Boolean remission at all visits;
- Concomitant corticosteroid use.

Additionally, assessment for the evaluation of radiographic changes in Period 2 will occur at Week 96 and every 96 weeks thereafter (or Premature Discontinuation Visit):



- Change from baseline in mTSS;
- Proportion of subjects with no radiographic progression (defined as change from baseline mTSS of  $\leq 0$ );
- Change from baseline in radiographic joint space narrowing and erosion scores.

## 5.3.4 Safety Variables

Safety evaluations include AE monitoring, physical examinations, vital sign measurements, ECG, and clinical laboratory testing (hematology, chemistry, and urinalysis) as a measure of safety and tolerability for the entire study duration.

#### 5.3.5 Pharmacokinetic Variables

Plasma upadacitinib concentrations will be obtained at the times indicated in Appendix D. A non-linear mixed-effects modeling approach will be used to estimate the population central values and the empirical Bayesian estimates of the individual values of upadacitinib oral clearance (CL/F) and volume of distribution (V/F). Additional parameters may be estimated if useful in the interpretation of the data.

## 5.3.6 Exploratory Research Variables and Validation Studies

Optional samples may be collected to conduct exploratory investigations into known and novel biomarkers. The types of biomarkers to be analyzed may include, but are not limited to nucleic acids, proteins, lipids, or metabolites.

Biomarker assessments may be used to assess and generate prognostic, predictive, pharmacodynamic, or surrogate biomarker signatures. These assessments may be explored in the context of RA or related conditions and/or upadacitinib or drugs of similar classes. These results from these analyses are exploratory in nature and may not be included with the clinical study report (CSR).

The samples may also be used to develop new therapies, research methods or technologies. In addition, samples from this study may be stored for future use. Samples may then be



used to validate putative biomarker signatures obtained from a prospective study, leading to the development of diagnostic tests.

## 5.4 Removal of Subjects from Therapy or Assessment

## 5.4.1 Discontinuation of Individual Subjects

Subjects can request to be discontinued from participating in the study at any time for any reason, including but not limited to disease progression or lack of response to treatment. The Investigator may discontinue any subject's participation for any reason, including an AE, safety concerns, lack of efficacy, or failure to comply with the protocol. See Section 6.1.7 for toxicity management criteria.

Subjects will have study drug discontinued immediately if any of the following occur:

- Clinically significant abnormal laboratory results or AEs, which rule out continuation of the study drug, as determined by the Investigator or the AbbVie Therapeutic Area Medical Director.
- Serious infections (e.g., sepsis) which cannot be adequately controlled within 2 weeks by anti-infective treatment or would put the subject at risk for continued participation in the trial as determined by the Investigator.
- The Investigator believes it is in the best interest of the subject.
- The subject requests withdrawal from the study.
- Inclusion or exclusion criteria violation was noted after the subject started study drug, when continuation of the study drug would place the subject at risk as determined by the AbbVie Therapeutic Area Medical Director.
- Introduction of prohibited medications or dosages when continuation of the study drug would place the subject at risk, as determined by the AbbVie Therapeutic Area Medical Director.
- Subject is non-compliant with TB prophylaxis (if applicable) or develops active TB at any time during the study.
- The subject becomes pregnant while on study drug.
- Malignancy, except for localized NMSC or carcinoma in situ of the cervix.



- Subject is significantly non-compliant with study procedures which would put the subject at risk for continued participation as determined by the Investigator or the AbbVie Therapeutic Area Medical Director.
- Subject develops a gastrointestinal perforation (other than due to appendicitis or mechanical injury).
- Subject with disease progression or not responding to treatment as determined by the Investigator.
- Confirmed diagnosis of deep vein thrombosis, pulmonary embolus or non-cardiac, non-neurologic arterial thrombosis.
- Starting at Week 48, subjects who fail to show at least 20% improvement in both TJC and SJC compared to baseline at 2 consecutive visits, despite optimization of background RA therapies (see Section 5.2.3.1 for permitted background RA therapies), will be discontinued from study drug. Therefore, the earliest discontinuation would be at Week 60, after completion of all Week 60 study visit activities.

In order to minimize missing data for efficacy and safety assessments, subjects who prematurely discontinue study drug treatment or study participation should complete a Premature Discontinuation visit (PD visit) as described in Section 5.1.

All attempts must be made to determine the date of the last study drug dose and the primary reason for discontinuation of study drug or study participation. The information will be recorded on the appropriate eCRF page. However, these procedures should not interfere with the initiation of any new treatments or therapeutic modalities that the Investigator feels are necessary to treat the subject's condition. Following discontinuation of study drug, the subject will be treated in accordance with the Investigator's best clinical judgment, irrespective of whether the subject decides to continue participation in the study.

During the COVID-19 pandemic, it has been necessary to employ mitigation strategies to enable the investigator to ensure subject safety and continuity of care.

During a state of emergency or pandemic situation like COVID-19, the investigator should contact the sponsor medical contact before discontinuing a subject from the study



or study drug for a reason other than "planned per protocol," to ensure all acceptable mitigation steps have been explored.

## **Lost to Follow-Up**

For subjects to be considered lost to follow-up, reasonable attempts must be made to obtain information on the final status of the subject. At a minimum, two phone calls must be made and one certified letter must be sent and documented in the subject's source documentation.

## 5.4.2 Discontinuation of Entire Study

AbbVie may terminate this study prematurely, either in its entirety or at any study site, for reasonable cause provided that written notice is submitted in advance of the intended termination. The Investigator may also terminate the study at his/her site for reasonable cause, after providing written notice to AbbVie in advance of the intended termination. Advance notice is not required by either party if the study is stopped due to safety concerns. If AbbVie terminates the study for safety reasons, AbbVie will immediately notify the Investigator by telephone and subsequently provide written instructions for study termination.

#### 5.5 Treatments

#### 5.5.1 Treatments Administered

There are two active study drugs in this study. The first is daily upadacitinib and the second is weekly MTX.

Upadacitinib (or matching placebo) study drug will be taken orally once daily, beginning on Day 1 (Baseline), and should be taken at approximately the same time each day. The study drug can be taken with or without food.



MTX (or matching placebo) study drug will be taken orally once weekly, beginning on Day 1 (Baseline), and should be taken the same day and approximately the same time each week. The study drug can be taken with or without food.

Each subject will be instructed to take 2 capsules once weekly (MTX and/or matching placebo) and 1 tablet once daily (upadacitinib or matching placebo) to maintain blinding. MTX and matching placebo will be assigned via the Interactive Response Technology (IRT) system, and distributed as identical capsules in blister packs, to provide the correct total dose for each individual subject and to maintain blinding during and after MTX titration (Period 1 and Period 2). Detailed dosing instructions can be found in the Subject Dosing Diary and Instructions. Starting with Amendment 6 subjects receiving MTX will receive open-label MTX tablets in quantities sufficient to cover their respective dose.

Subjects should take a dietary supplement of oral folic acid beginning on Day 1 (Baseline) throughout study participation. Folic acid dosing and timing of regimen should be followed according to the Investigator's instructions.

When the last subject completes the Week 24 Visit of Period 1, the study conduct of Period 1 may be unblinded only to the sponsor for analysis. Subjects and sites will remain blinded to treatment assignment throughout Period 1. When the last subject completes the last visit of Period 1 (Week 48), study drug assignment in both periods may be unblinded to the Sponsor and sites, and subjects would then be dispensed study drug in an open-label fashion until the completion of Period 2. All subjects will continue study treatment to which they were assigned at the time of study unblinding. Dose changes of open-label study drugs are not permitted during unblinded Period 2. Background therapies may be adjusted as per the discretion of the investigator. Starting with Amendment 6, subjects receiving upadacitinib 15 mg and 30 mg QD will receive open-label upadacitinib 15 mg QD. Starting with Amendment 6 subjects receiving MTX will receive open-label MTX.

If a subject is unable to come to the study site to pick up their study drug due to state of emergency or any pandemic like COVID-19, a direct-to-patient (DTP) study drug



shipment can be made from the study site to the subject if allowed by local regulations. AbbVie will submit any required notifications to the regulatory authority as applicable. Refer to Section 5.3.1.1 for details on DTP shipment of study drug.

# 5.5.2 Identity of Investigational Product

The individual study drug information is presented in Table 3.

**Table 3.** Identity of Investigational Product

| Investigational<br>Product | Mode of Administration | Formulation | Strength | Manufacturer |
|---|---|---|---|---|
| Upadacitinib<br>(ABT-494) | oral | tablet | 7.5 mg<br>15 mg<br>30 mg | AbbVie |
| Upadacitinib<br>(ABT-494)<br>matching placebo | oral | tablet | NA | AbbVie |
| MTX | oral | 2.5 mg tablet<br>over-encapsulated<br>in hard gelatin<br>capsule | 7.5 mg<br>10 mg | Over-encapsulated MTX capsule: Fisher Clinical Services for AbbVie MTX: Dava Pharmaceuticals and/or Orion and/or Hexal AG and/or Goldshield and/or PAR Pharmaceuticals |
| MTX | oral | tablet | 2.5 mg | Dava Pharmaceuticals and/or<br>Orion and/or Hexal AG and/or<br>Goldshield and/or PAR<br>Pharmaceuticals and/or SUN<br>Pharmaceuticals and/or Mylan<br>and/or Hikma Pharmaceuticals |
| MTX matching placebo | oral | capsule | NA | Fisher Clinical Services and/or AbbVie |

Folic acid will be supplied by the subject, according to Investigator's instructions for dosing and timing of administration.



## 5.5.2.1 Packaging and Labeling

Upadacitinib and matching placebo will be packaged in bottles with quantities sufficient to accommodate study design. MTX and matching placebo will be packaged in blister packs and/or bottles and/or cartons with quantities sufficient to accommodate study design. Each kit label will contain a unique kit number. This kit number is assigned to a subject via IRT and encodes the appropriate study drug to be dispensed at the subject's corresponding study visit. Each kit will be labeled as required per country requirements. Labels must remain affixed to the kits. All blank spaces on the label will be completed by the site staff prior to dispensing to the subjects.

## 5.5.2.2 Storage and Disposition of Study Drugs

Study drugs must be stored at controlled room temperature (15° to 25°C/59° to 77°F). The investigational products are for investigational use only and are to be used only within the context of this study. The study drug supplied for this study must be maintained under adequate security and stored under the conditions specified on the label until dispensed for subject use or destroyed as appropriate.

## 5.5.3 Method of Assigning Subjects to Treatment Groups

All subjects will be randomized using IRT. Before the study is initiated, IRT directions will be provided to each site.

All subjects will be assigned a unique identification number by the IRT at the Screening Visit. For subjects that re-screen, the Screening number assigned by the IRT at the initial Screening Visit should be used; a new Screening number should not be requested.

Subjects will be eligible for randomization if they continue to meet all of the selection criteria (Section 5.2) at Baseline and are willing to continue in the study.

Subjects will be randomized in a 1:1:1 ratio using interactive response technology (IRT) to treatment Groups 2, 3, and 4, below, except for subjects from Japan, who will be randomized in a 2:1:1:1 ratio to Groups 1, 2, 3, and 4:



- Group 1: Upadacitinib 7.5 mg QD monotherapy (subjects in Japan only; N = 75)
- Group 2: Upadacitinib 15 mg QD monotherapy (N = 300) (includes 37 subjects from Japan)
- Group 3: Upadacitinib 30 mg QD monotherapy (N = 300) (includes 37 subjects from Japan)
- Group 4: MTX monotherapy (N = 300) (includes 37 subjects from Japan)

Randomization will be stratified by geographic region.

The IRT will assign a randomization number that will encode the subject's treatment group assignment according to the randomization schedule generated by the Statistics Department at AbbVie.

IRT will provide the appropriate study drug kit number(s) to dispense to each subject. Study drug will be administered at the study visits as summarized in Section 5.3.1.1. Returned study drug should not be re-dispensed to any subject.

Starting with Amendment 6, subjects receiving upadacitinib 15 mg and 30 mg QD will receive open-label upadacitinib 15 mg QD. Starting with Amendment 6 subjects receiving MTX will receive open-label MTX.

# 5.5.4 Selection and Timing of Dose for Each Subject

Subjects should take study drug as outlined in Section 5.5.1.

On dosing days that occur on study visit days, subjects should follow the regular dosing schedule (refer to Section 5.3.2.1 regarding Week 2 and Week 4 Visits).

Each subject's dosing schedule should be closely monitored by the site at each study visit by careful review of the subject's dosing diary. This will ensure that all subjects enrolled into the study maintain their original dosing schedule beginning with the first dose of study drug (Baseline/Day 1).



#### Upadacitinib/Placebo tablets (daily dosing):

- If a subject should forget to take his/her daily upadacitinib (or matching placebo) dose at his/her regularly scheduled dosing time, he/she should take the forgotten dose as soon as they remember the dose was missed as long as it is at least 10 hours before his/her next scheduled dose. If a subject only remembers the missed dose within 10 hours before next scheduled dose, the subject should skip the missed dose and take the next dose at the scheduled time.
- If the subject experiences a study drug interruption > 14 consecutive days during Period 1 or > 30 days during Period 2 (other than for reasons listed in Section 6.1.7), he/she should notify the Investigator, and the Investigator will determine if study drug should be restarted. If study drug treatment is interrupted or withdrawn in Periods 1 or 2, both daily and weekly study drug administration must be stopped. Period 2 may be unblinded after all subjects complete Period 1, at which time daily and weekly study drugs can be individually interrupted.

#### MTX/Placebo capsules or tablets (weekly dosing):

- Weekly MTX (or matching placebo) should be taken the same day and approximately the same time each week. If the subject should forget to take his/her oral MTX (or matching placebo) dose on his/her regularly scheduled dosing date, he/she should take the forgotten dose as soon as he/she remembers. If more than 72 hours has elapsed since the missed dose, the subject should contact the Investigator for further dosing instructions. The study drug can be taken with or without food.
- If the subject experiences a study drug interruption ≥ 3 consecutive missed doses in Period 1 or 2 (other than for reasons listed in Section 6.1.7), he/she should notify the Investigator, and the Investigator will determine if study drug should be restarted. If study drug treatment is interrupted or withdrawn in Periods 1 or 2, both daily and weekly study drug administration must be stopped. Period 2 may be unblinded after all subjects complete Period 1, at which time daily and weekly study drugs can be individually interrupted.



#### 5.5.5 Blinding

## 5.5.5.1 Blinding of Investigational Product

All AbbVie personnel with direct oversight conduct and management of the trial (with the exception of AbbVie Drug Supply Management Team), the Investigator, study site personnel, and the subject will remain blinded to each subject's treatment throughout Period 1.

In order to maintain the blind, the upadacitinib and placebo tablets along with MTX and placebo capsules provided for the study will be identical in appearance. The IRT will provide access to unblinded subject treatment information in the case of medical emergency.

In the event of a medical situation that requires unblinding of the study drug assignment, the Investigator is requested to contact the AbbVie Therapeutic Area Medical Director prior to breaking the blind. However, if an urgent therapeutic intervention is necessary which warrants breaking the blind prior to contacting the AbbVie Therapeutic Area Medical Director, the Investigator can directly access the IRT system to break the blind without AbbVie notification or agreement. Unblinding is available in the IRT system via the Unblind Subject transaction, which is available only to the Investigator. If the IRT system is unavailable, unblinding may occur by contacting EndPoint technical support via either phone (preferred) or email (support@endpointclinical.com). For country-specific phone numbers, please see the following website: http://www.endpointclinical.com/help-desk/. In the event that the blind is broken before notification to the AbbVie Therapeutic Area Medical Director, we request that the AbbVie Therapeutic Area Medical Director be notified within 24 hours of the blind being broken. The date and reason that the blind was broken must be conveyed to AbbVie and recorded on the appropriate eCRF.

When the last subject completes the last visit of Period 1 (Week 48), study drug assignment in both periods may be unblinded to the Sponsor and sites, and subjects would then be dispensed study drug in an open-label fashion until the completion of Period 2.



## 5.5.5.2 Blinding of Data for Data Monitoring Committee

An external Data Monitoring Committee (DMC) comprised of persons independent of AbbVie and with relevant expertise in their field will review unblinded safety data from the ongoing study. The primary responsibility of the DMC will be to protect the safety of the subjects participating in this study.

A separate DMC charter will be prepared outside of the protocol and will describe the roles and responsibilities of the DMC members, frequency of data reviews, and relevant safety data to be assessed.

Communications from the DMC to the Study Teams will not contain information that could potentially unblind the team to subject treatment assignments.

As of September 2018, with all subjects having reached the end of Period 1, and after final review of unblinded safety data, the DMC concluded its oversight of this study.

## 5.5.6 Treatment Compliance

The Investigator or his/her designated and qualified representatives will administer/dispense study drug only to subjects enrolled in the study in accordance with the protocol. The study drug must not be used for reasons other than that described in the protocol.

Subject dosing will be recorded on a subject dosing diary. Subjects will be instructed to return all drug containers (even if empty) to the study site personnel at each clinic visit. The study site personnel will document compliance in the study source documents.

## 5.5.7 Drug Accountability

The Investigator or his/her representative will verify that study drug supplies are received intact and in the correct amounts. This will be documented by signing and dating the Proof of Receipt or similar document and by registering the arrival of drug through the


IRT. The original Proof of Receipt Note and the IRT confirmation sheet will be kept in the site files as a record of what was received.

In addition, an IRT will be used to document investigational product accountability including but not limited to date received, the lot number, kit number(s), date dispensed, subject number, and the identification of the person dispensing the drug.

All empty/used study drug packaging will be inventoried by the site. Empty/used study drug packaging should be returned by the subject at each visit for accountability and compliance purposes and new packaging issued as necessary. Site staff will complete study drug accountability via IRT by using source documents, subject dosing diaries, and by visually inspecting the packaging whenever possible. After drug accountability and monitor reconciliation has been completed, used packaging and unused study drug will be destroyed on site according to local procedures or regulations or returned to the destruction depot (for those sites that do not meet AbbVie's documentation requirements for on-site destruction). The use of a third-party vendor for drug destruction must be preapproved by AbbVie. For sites performing on-site drug destruction or using a third-party vendor for drug destruction, a copy of the destruction methodology and date of destruction should be maintained at the site's facility.

Site monitors will reconcile the site's processes, source documents, subject's dosing diaries, IRT or site accountability records, and destruction records to assure site compliance.

# 5.6 Discussion and Justification of Study Design

# 5.6.1 Discussion of Study Design and Choice of Control Groups

This multicenter study includes two periods.

Period 1 is a 48-week randomized, double-blind, parallel-group, active comparator-controlled treatment period designed to compare the safety and efficacy of upadacitinib 7.5 mg QD monotherapy (for subjects in Japan only), 15 mg QD



monotherapy, and 30 mg QD monotherapy versus MTX monotherapy in adult MTX-naïve subjects with moderately to severely active RA. Period 1 is also designed to compare the efficacy of upadacitinib 15 mg QD monotherapy and 30 mg QD monotherapy versus MTX monotherapy for the prevention of structural progression. Period 1 is designed to test superiority of upadacitinib versus MTX for achieving the primary endpoint (the proportion of subjects achieving ACR50 response [US/FDA regulatory purposes] or the proportion of subjects achieving CR [EU/EMA regulatory purposes] or ACR20 and change from baseline in mTSS [Japan/PMDA regulatory purposes]) at Week 24, and other secondary efficacy parameters.

The purpose of Period 2 is to evaluate the long-term safety, tolerability, and efficacy of upadacitinib (7.5, 15, or 30 mg QD) in subjects with RA who have completed Period 1. All subjects will continue treatment to which they were assigned at the end of Period 1 in a blinded manner. This will allow unbiased assessments of long-term safety of upadacitinib without compromising the study conduct or results of ongoing Period 1. Dose reduction or escalation of upadacitinib during Period 2 is not permitted to allow unbiased assessments of long-term safety and efficacy of upadacitinib 30 mg QD versus 15 mg QD.

When the last subject completes the last visit of Period 1 (Week 48), study drug assignment in both periods may be unblinded to the Sponsor and sites, and subjects would then be dispensed study drug in an open-label fashion until the completion of Period 2.

Starting with Amendment 6, subjects receiving upadacitinib 15 mg and 30 mg QD will receive open-label upadacitinib 15 mg QD. Starting with Amendment 6 subjects receiving MTX will receive open-label MTX.

#### 5.6.2 Appropriateness of Measurements

Standard statistical, clinical, and laboratory procedures will be utilized in this study. All efficacy measurements in this study are standard for assessing disease activity in subjects



with RA. All clinical and laboratory procedures in this study are standard and generally accepted.

## 5.6.3 Suitability of Subject Population

The intended study population is moderately to severely active RA patients who are naïve to MTX treatment. Key entry criteria are to enroll adult female and male subjects who are at least 18 years of age with symptoms consistent with RA for  $\geq 6$  weeks who also fulfill the 2010 ACR/EULAR classification criteria for RA and no prior or limited MTX treatment. Eligible study subjects must have  $\geq 6$  swollen joints (based on 66 joint counts) and  $\geq 6$  tender joints (based on 68 joint counts) at Screening and Baseline Visits, and hsCRP  $\geq 5$  mg/L (central lab, ULN 2.87 mg/L) at Screening.

## 5.6.4 Selection of Doses in the Study

Three doses of the once-daily formulation of upadacitinib will be evaluated: upadacitinib 7.5 mg QD (subjects in Japan only), 15 mg QD, and 30 mg QD. The dose selection in this study is based on extrapolation of pre-clinical efficacy models and analyses of PK, pharmacodynamic, safety, and efficacy data from the Phase 1 studies in healthy volunteers (single and multiple ascending dose Studies M13-401 and M13-845, respectively) and Phase 2 studies in RA subjects (Studies M13-537 and M13-550). The doses selected for Study M13-545, upadacitinib 7.5 mg QD (for subjects in Japan only), 15 mg QD, and 30 mg QD, dosed up to 260 weeks, are expected to be efficacious with an acceptable safety profile.

Preliminary results from an ongoing relative bioavailability study demonstrated that single 15 mg and 30 mg doses of the once-daily formulation provide comparable AUC and significantly lower C<sub>max</sub> than single doses of 12 mg immediate release formulation (AUC equivalent to 6 mg BID dose tested in Phase 2) and 24 mg immediate release formulation (AUC equivalent to 12 mg BID dose tested in Phase 2), respectively, under fasting conditions. At steady-state, the once-daily dose of 15 mg QD is predicted to achieve comparable daily AUC and C<sub>max</sub>, and non-inferior C<sub>trough</sub> to 6 mg BID immediate release formulation. In the Phase 2 studies, the 6 mg BID dose was shown to achieve near



maximum efficacy. The once-daily dose of 30 mg QD is predicted to achieve comparable daily AUC and  $C_{max}$ , and non-inferior  $C_{trough}$  to 12 mg BID immediate release formulation. In the Phase 2 studies, the 12 mg BID dose was clearly shown to achieve the plateau of efficacy.

# 6.0 Complaints

A Complaint is any written, electronic, or oral communication that alleges deficiencies related to the physical characteristics, identity, quality, purity, potency, durability, reliability, safety, effectiveness, or performance of a product/device after it is released for distribution.

Complaints associated with any component of this investigational product must be reported to the Sponsor (Section 6.2.2). For AEs, please refer to Section 6.1. For product complaints, please refer to Section 6.2.

## 6.1 Medical Complaints

The Investigator will monitor each subject for clinical and laboratory evidence of AEs on a routine basis throughout the study. The Investigator will assess and record any AE in detail including the date of onset, event diagnosis (if known) or sign/symptom, severity, time course (end date, ongoing, intermittent), relationship of the AE to study drug, and any action(s) taken. For SAEs considered as having "no reasonable possibility" of being associated with study drug, the Investigator will provide other cause(s) of the event. For AEs to be considered intermittent, the events must be of similar nature and severity. AEs, whether in response to a query, observed by site personnel, or reported spontaneously by the subject will be recorded.

All AEs will be followed to a satisfactory conclusion.



#### 6.1.1 Definitions

#### 6.1.1.1 Adverse Event

An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not the event is considered causally related to the use of the product.

Such an event can result from use of the drug as stipulated in the protocol or labeling, as well as from accidental or intentional overdose, drug abuse, or drug withdrawal. Any worsening of a pre-existing condition or illness is considered an AE. Worsening in severity of a reported AE should be reported as a new AE. Laboratory abnormalities and changes in vital signs are considered to be AEs only if they result in discontinuation from study drug, necessitate therapeutic medical intervention, and/or if the investigator considers them to be AEs.

An elective surgery/procedure scheduled to occur during the study will not be considered an AE if the surgery/procedure is being performed for a pre-existing condition and the surgery/procedure has been pre-planned prior to study entry. However, if the pre-existing condition deteriorates unexpectedly during the study (e.g., surgery performed earlier than planned), then the deterioration of the condition for which the elective surgery/procedure is being done will be considered an AE.

#### 6.1.1.2 Serious Adverse Events

If an adverse event meets any of the following criteria, it is to be reported to AbbVie as a SAE within 24 hours of the site being made aware of the SAE.

**Death of Subject** An event that results in the death of a subject.



**Life-Threatening** An event that, in the opinion of the investigator, would have

resulted in immediate fatality if medical intervention had not been taken. This does not include an event that would have

been fatal if it had occurred in a more severe form.

Hospitalization or Prolongation of Hospitalization An event that results in an admission to the hospital for any length of time or prolongs the subject's hospital stay. This does not include an emergency room visit or admission to an

outpatient facility.

**Congenital Anomaly** An anomaly detected at or after birth, or any anomaly that

result in fetal loss.

Persistent or Significant Disability/Incapacity An event that results in a condition that substantially interferes with the activities of daily living of a study subject. Disability is not intended to include experiences of relatively minor medical significance such as headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (e.g., sprained ankle).

Important Medical Event Requiring Medical or Surgical Intervention to Prevent Serious Outcome An important medical event that may not be immediately life-threatening or result in death or hospitalization, but based on medical judgment may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above (i.e., death of subject, life-threatening, hospitalization, prolongation of hospitalization, congenital anomaly, or persistent or significant disability/incapacity). Additionally, any elective or spontaneous abortion or stillbirth is considered an important medical event. Examples of such events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.

For SAEs with the outcome of death, the date and cause of death will be recorded on the appropriate case report form.



#### 6.1.1.3 Adverse Events of Special Interest

The following AEs of special interest will be monitored during the study (see detailed toxicity management in Section 6.1.7):

- Serious infections, opportunistic infections, herpes zoster, and TB;
- Malignancy (all types);
- Adjudicated gastrointestinal perforations;
- Adjudicated cardiovascular events (e.g., major adverse cardiovascular event [MACE]);
- Anemia;
- Decreased neutrophil counts;
- Decreased lymphocyte counts;
- Increased serum creatinine and renal dysfunction;
- Hepatic events and increased hepatic transaminases;
- Increased creatine phosphokinase (CPK);
- Adjudicated embolic and thrombotic events (non-cardiac, non-CNS).

#### 6.1.2 Adverse Event Severity

The Investigator will classify adverse events according to the Rheumatology Common Toxicity Criteria v.2.0 (Appendix R).<sup>22</sup>

#### 6.1.3 Relationship to Study Drug

The Investigator will use the following definitions to assess the relationship of the adverse event to the use of study drug:



Upadacitinib M13-545 Protocol Amendment 8 EudraCT 2015-003334-27

**Reasonable** After consideration of factors including timing of the event, biologic plausibility, clinical judgment, and potential alternat

biologic plausibility, clinical judgment, and potential alternative causes, there is **sufficient** evidence (information) to suggest a

causal relationship.

No Reasonable After consideration of factors including timing of the event, biologic plausibility, clinical judgment, and potential alternation of factors including timing of the event, biologic plausibility, clinical judgment, and potential alternation of factors including timing of the event, biologic plausibility and potential alternation of factors including timing of the event, biologic plausibility and potential alternation of factors including timing of the event, biologic plausibility and potential alternation of factors including timing of the event, biologic plausibility and potential alternation of factors including timing of the event, biologic plausibility and potential alternation of factors including timing of the event, and potential alternation of factors including timing of the event, and potential alternation of factors including timing of the event, and potential alternation of factors including timing of the event, and potential alternation of factors including timing of the event, and potential alternation of factors including the event of the ev

biologic plausibility, clinical judgment, and potential alternative causes, there is **insufficient** evidence (information) to suggest a

causal relationship.

For causality assessments, events assessed as having a reasonable possibility of being related to the study drug will be considered "associated." Events assessed as having no reasonable possibility of being related to study drug will be considered "not associated." In addition, when the Investigator has not reported a causality or deemed it not assessable, AbbVie will consider the event associated.

If an investigator's opinion of no reasonable possibility of being related to study drug is given, an Other cause of event must be provided by the investigator for the Serious Adverse Event.

#### 6.1.4 Adverse Event Collection Period

All AEs reported from the time of study drug administration until 30 days following discontinuation of study drug administration have elapsed will be collected, whether solicited or spontaneously reported by the subject. Subjects who discontinue study drug treatment but continue to participate in the study will have SAEs and nonserious AEs collected for the remainder of study participation. In addition, SAEs and protocol-related nonserious AEs will be collected from the time the subject signed the study-specific informed consent.

Adverse event information will be collected as shown in Figure 5.



Figure 5. Adverse Event Collection



Additionally, in order to assist the adjudication process, additional information on any potential cardiovascular events including thromboembolic events will be collected, if applicable.

In case of any of the following reported events, an appropriate supplemental eCRF should be completed:

- Cardiac events;
- Myocardial infarction or unstable angina;
- Heart failure;
- Cerebral vascular accident and transient ischemic attack;
- Cardiovascular procedures (SAE Supplemental Procedure eCRF);
- Embolic and thrombotic events (non-cardiac, non-CNS);
- Hepatic;
- Renal;
- Herpes Zoster Infection;
- CPK increase considered by the investigator to be an AE.
- COVID-19.

Supplemental study case report forms should be completed in the event of COVID-19 related missed/virtual visits, study drug interruptions or discontinuations, or adverse



events (including documentation of specific signs/symptoms of infection and testing results).

COVID-19 infections should be captured as adverse events. If the event meets the criteria for a serious adverse event (SAE), then follow the SAE reporting directions per the protocol and above.

The following COVID-19 related supplemental eCRFs should be completed (for both serious and non-serious events):

- COVID-19 Supplemental Signs/Symptoms
- COVID-19 Status Form

## 6.1.5 Serious Adverse Event Reporting

In the event of an SAE, whether associated with study drug or not, the Investigator will notify Clinical Pharmacovigilance within 24 hours of the site being made aware of the SAE by entering the SAE data into the electronic data capture (EDC) system (RAVE®). SAEs that occur prior to the site having access to the RAVE system, or if RAVE is not operable, should be documented on the SAE Non-CRF forms and emailed (preferred route) or faxed to Clinical Pharmacovigilance within 24 hours of the site being made aware of the SAE.

Email: PPDINDPharmacovigilance@abbvie.com

FAX to: +1 (847) 938-0660

For safety concerns, contact the Immunology Safety Team at:



M13-545 Protocol Amendment 8 EudraCT 2015-003334-27

Immunology Safety Team 1 North Waukegan Road North Chicago, IL 60064

Toll Free: +1 (833) 942-2226

Email: GPRD\_SafetyManagement\_Immunology@abbvie.com

For any subject safety concerns, please contact the physician listed below:

Primary Therapeutic Area Medical Director:

| MD |
|-------------------------|
| Medical Director |
| AbbVie Inc. |
| 1 North Waukegan Road |
| North Chicago, IL 60064 |
| _ |
| Contact Information: |
| Office: |
| Mobile: |
| Fax: |
| Email: |

In emergency situations involving study subjects when the primary Therapeutic Area Medical Director is not available by phone, please contact the 24-hour AbbVie Medical Escalation Hotline where your call will be re-directed to a designated backup AbbVie Therapeutic Area Medical Director:

Phone: +1 (973) 784-6402

The sponsor will be responsible for Suspected Unexpected Serious Adverse Reactions (SUSAR) reporting for the Investigational Medicinal Product (IMP) in accordance with Global and Local Regulations. The reference document used for SUSAR reporting in the European Union countries will be the most current version of the Investigator's Brochure



for upadacitinib and/or the Summary of Product Characteristics (SmPC) for MTX, as applicable.

In Japan, the Principal Investigator will provide documentation of all SAEs to the Director of the investigative site and the Sponsor.

#### 6.1.6 Pregnancy

Pregnancy in a study subject must be reported to AbbVie within 24 hours after the site becomes aware of the pregnancy. Subjects who become pregnant during the study must be discontinued from study drug (Section 5.4.1).

Information regarding a pregnancy occurrence in a study subject and the outcome of the pregnancy will be collected. Pregnancies in study subjects will be collected from the date of the first dose through 180 days following the last dose of study drug.

Pregnancy in a study subject is not considered an AE. However, the medical outcome of an elective or spontaneous abortion, stillbirth, or congenital anomaly is considered an SAE and must be reported to AbbVie within 24 hours of the site becoming aware of the event.

Subjects and partners of subjects receiving MTX should avoid pregnancy throughout the course of the study, starting with the Screening Visit through 180 days after the last study drug administration for female subjects and male subjects receiving MTX. Male subjects receiving MTX should also refrain from donating sperm for up to 180 days post last dose of study drug. Results of a positive pregnancy test or confirmation of a pregnancy will be assessed starting with the Screening Visit through the final study visit.

# 6.1.7 Toxicity Management

The toxicity management of the AEs including AEs of special interest consists of safety monitoring (review of AEs on an ongoing basis, and periodical/ad hoc review of safety issues by a safety data monitoring committee), interruption of study drug dosing with appropriate clinical management if applicable, and discontinuation of the subjects from



the study drug. The management of specific AEs and laboratory parameters is described below.

For subjects who discontinued study drug, but continued study participation and are instead on standard of care therapies, these toxicity management requirements do not apply (including alerts from the central lab) and any intolerability to standard of care therapies should be managed by the prescribing physician.

Serious Infections: Subjects should be closely monitored for the development of signs and symptoms of infection during and after treatment with study drug. Study drug should be interrupted if a subject develops a serious infection or an opportunistic infection. A subject who develops a new infection during treatment with study drug should undergo prompt diagnostic testing appropriate for an immunocompromised subject. As appropriate, antimicrobial therapy should be initiated, and the subject should be closely monitored. Re-challenge with study drug may occur once the infection has been successfully treated. Subjects who develop active TB must be discontinued from study drug.

**COVID-19:** Interrupt study drug in subjects with a confirmed diagnosis of COVID-19. Consider interrupting study drug in subjects with signs and/or symptoms and suspicion of COVID-19. The COVID-19 eCRF must be completed.

**Herpes zoster:** If a subject develops herpes zoster, consider temporarily interrupting study drug until the episode resolves.

**Gastrointestinal Perforation:** If a diagnosis of gastrointestinal perforation is confirmed (other than appendicitis or penetrating injury), the subject must be permanently discontinued from study drug.

**Cardiovascular Events (MACE):** Subjects presenting with potential cardiovascular events should be carefully monitored. These events will be reviewed and adjudicated by an independent Cardiovascular Adjudication Committee in a blinded manner.



**Thrombosis Events:** Subjects who develop symptoms of thrombosis should be promptly evaluated and treated appropriately. If the diagnosis of deep vein thrombosis, pulmonary embolus or non-cardiac, non-neurologic arterial thrombosis is confirmed, the subject must be discontinued from study drug.

**Malignancy:** Subjects who develop malignancy other than NMSC or carcinoma in situ of the cervix must be discontinued from study drug. Information including histopathological results should be queried for the confirmation of the diagnosis. Periodic skin examination is recommended for subjects who are at increased risk for skin cancer.

**ECG Abnormality:** Subjects must be discontinued from study drug for an ECG change considered clinically significant and with reasonable possibility of relationship to study drug OR a confirmed absolute QTcF value > 500 msec.

Management of Select Laboratory Abnormalities: For any given laboratory abnormality, the Investigator should assess the subject, apply the standard of care for medical evaluation and treatment following any local guidelines. Specific toxicity management guidelines for abnormal laboratory values are described in Table 4, and may require an appropriate supplemental eCRF to be completed. All abnormal laboratory tests that are considered clinically significant by the Investigator will be followed to a satisfactory resolution. If a repeat test is required per Table 4, the repeat testing must occur as soon as possible.



# Table 4. Specific Toxicity Management Guidelines for Abnormal Laboratory Values

| Laboratory Parameter | Toxicity Management Guideline |
|---|---|
| Hemoglobin | If hemoglobin < 8 g/dL interrupt study drug dosing and confirm by repeat testing with new sample. |
| | • If hemoglobin decreases ≥ 3.0 g/dL from baseline without an alternative etiology, interrupt study dosing and confirm by repeat testing with new sample. |
| | • If hemoglobin decreases ≥ 3.0 g/dL from baseline and an alternative etiology is known, the subject may remain on study drug at the investigator's discretion. |
| | If confirmed, continue to withhold study drug until hemoglobin value returns to normal reference range or its baseline value. |
| Absolute neutrophil count (ANC) | • If confirmed < 1000 cells/µL by repeat testing with new sample, interrupt study drug dosing until ANC value returns to normal reference range or its baseline value. |
| | • Discontinue study drug if confirmed < 500 cells/μL by repeat testing with new sample. |
| Absolute lymphocyte counts (ALC) | • If confirmed < 500 cells/µL by repeat testing with new sample, interrupt study drug dosing until ALC returns to normal reference range or its baseline value. |
| Total white blood cell count | • If confirmed < 2000 cells/μL by repeat testing with new sample, interrupt study drug dosing until white blood cell count returns to normal reference range or its baseline value. |
| Platelet count | • If confirmed < 50,000 cells/µL by repeat testing with new sample, interrupt study drug dosing until platelet count returns to normal reference range or its baseline value. |



Table 4. Specific Toxicity Management Guidelines for Abnormal Laboratory Values (Continued)

| <b>Laboratory Parameter</b> | Toxicity Management Guideline |
|---|---|
| AST or ALT | • Interrupt study drug immediately if confirmed ALT or AST > 3 × ULN by repeat testing with new sample and either a total bilirubin > 2 × ULN or an international normalized ratio > 1.5. |
| | <ul> <li>A separate blood sample for INR testing will be needed to measure INR at the<br/>time of repeat testing for ALT or AST. A repeat test of INR is not needed for<br/>determination if above toxicity management criteria are met.</li> </ul> |
| | • Interrupt study drug immediately if confirmed ALT or AST > 3 × ULN by repeat testing with new sample along with appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (> 5%). |
| | • Interrupt study drug immediately if confirmed ALT or AST > 5 × ULN by repeat testing with new sample for more than 2 weeks. |
| | • If ALT or AST > 8 × ULN, interrupt study drug immediately, confirm by repeat testing with new sample, and contact the TA MD. |
| | Subjects who meet any of the above criteria should be evaluated for an alternative etiology of the ALT or AST elevation and managed as medically appropriate. If applicable, the alternative etiology should be documented in the eCRF. If ALT or AST values return to the normal reference range or its Baseline value, study drug may be restarted. If restarting study drug, documentation should include reason that rechallenge is expected to be safe. If after clinically appropriate evaluation, no alternative etiology for ALT or AST elevation is found or the ALT or AST elevation has not resolved or is not trending down toward normal, the subject should be discontinued from study drug. |
| | For any confirmed ALT or AST elevations > 3 ULN, complete supplemental hepatic eCRF. |
| | Subjects with HBc Ab+ (irrespective of HBs Ab status) and negative HBV DNA at screening who develop the following should have HBV DNA by PCR testing performed within 1 week: |
| | $\circ ALT > 5 \times ULN \underline{OR}$ |
| | o ALT or AST > 3 × ULN if an alternative cause is not readily identified |
| | <ul> <li>A separate blood sample for HBV DNA PCR testing will be needed at the<br/>time of repeat testing for ALT or AST.</li> </ul> |
| | A positive result for HBV DNA PCR testing in these subjects will require immediate interruption of study drug and a hepatologist consultation should occur within 1 week for recommendation regarding subsequent treatment. |
| Serum Creatinine | <ul> <li>If serum creatinine is &gt; 1.5 × the baseline value and &gt; ULN, repeat the test for serum creatinine (with subject in an euvolemic state) to confirm the results. If the results of the repeat testing still meet this criterion, then interrupt study drug and restart study drug once serum creatinine returns to ≤ 1.5 × baseline value and ≤ ULN.</li> <li>If confirmed serum creatinine ≥ 2 mg/dL, interrupt study drug and re-start study</li> </ul> |
| | drug once serum creatinine elevation scenarios, complete supplemental renal eCRF. |



Table 4. Specific Toxicity Management Guidelines for Abnormal Laboratory Values (Continued)

| Laboratory Parameter | Toxicity Management Guideline |
|---|---|
| Creatine Phosphokinase | • If confirmed CPK value ≥ 4 × ULN and there are no symptoms suggestive of myositis or rhabdomyolysis, the subject may continue study drug at the investigator's discretion. |
| | <ul> <li>If CPK ≥ 4 × ULN accompanied by symptoms suggestive of myositis or<br/>rhabdomyolysis, interrupt study drug and contact AbbVie TA MD.</li> <li>For the above CPK elevation scenarios, complete supplemental CPK eCRF.</li> </ul> |

For allowed study drug interruption, the following rules apply:

#### Period 1

- Upadacitinib/Placebo tablet (daily dosing):
  - Allow study drug interruption  $\leq$  14 consecutive days for AEs and emergency surgery during the first 24 weeks;
  - After Week 24, study drug interruption due to AEs/ surgery is allowed ≤ 21 days.
- MTX/Placebo capsules (weekly dosing):
  - Allow study drug interruption  $\leq 2$  consecutive missed doses for AEs and emergency surgery during the first 24 weeks;
  - After Week 24, study drug interruption due to AEs/surgery is allowed
     ≤ 3 consecutive doses.
- If the subject must undergo emergency surgery, the study drug should be interrupted at the time of the surgery.
- Elective surgery during the first 24 weeks is discouraged and needs to be
  discussed with the AbbVie Therapeutic Area Medical Director. If the subject
  undergoes elective surgery, the study drugs should be interrupted one week
  prior to the planned surgery.
- After surgery, allow reintroduction of study drugs once the physician has examined the surgical site and determined that it has healed and there is no sign of infection.



#### Period 2

- Upadacitinib/Placebo tablet (daily dosing):
  - Up to 30 consecutive days of oral study drug interruption is allowed. The Investigator will make determination if study drug should be restarted for interruptions > 30 days.
- MTX/Placebo capsules or tablets (weekly dosing):
  - Study drug interruption due to AEs/surgery is allowed for ≤ 3 consecutive doses. The Investigator will make determination if study drug should be restarted for interruptions > 30 days.
- If the subject undergoes elective surgery, the study drug should be interrupted 1 week prior to the planned surgery. Allow reintroduction of study drug once the physician has examined the surgical site and determined that it has healed and there is no sign of infection.
- If the subject must undergo emergency surgery, the study drug should be interrupted at the time of surgery. Allow reintroduction of study drug once the physician has examined the surgical site and determined that it has healed and there is no sign of infection.

#### 6.1.8 Data Monitoring Committee

An external DMC will review unblinded safety data. See Section 5.5.5.2 for details.

#### 6.1.9 Cardiovascular Adjudication Committee

An independent committee of physician experts in cardiovascular adjudication will be utilized to assess potential cardiovascular AEs in a blinded manner as defined by the Cardiovascular Adjudication Committee charter.

#### 6.2 Product Complaint

#### 6.2.1 Definition

A Product Complaint is any Complaint (see Section 6.0 for the definition) related to the biologic or drug component of the product.



For a product this may include, but is not limited to, damaged/broken product or packaging, product appearance whose color/markings do not match the labeling, labeling discrepancies/inadequacies in the labeling/instructions (example: printing illegible), missing components/product, or packaging issues.

Any information available to help in the determination of causality to the events outlined directly above should be captured.

# 6.2.2 Reporting

Product Complaints concerning the investigational product must be reported to the Sponsor within 24 hours of the study site's knowledge of the event via the Product Complaint form. Product Complaints occurring during the study will be followed-up to a satisfactory conclusion. All follow-up information is to be reported to the Sponsor (or an authorized representative) and documented in source as required by the Sponsor. Product Complaints associated with AEs will be reported in the study summary. All other complaints will be monitored on an ongoing basis.

Product Complaints may require return of the product with the alleged complaint condition. In instances where a return is requested, every effort should be made by the Investigator to return the product within 30 days. If returns cannot be accommodated within 30 days, the site will need to provide justification and an estimated date of return.

The description of the complaint is important for AbbVie in order to enable AbbVie to investigate and determine if any corrective actions are required.

#### 7.0 Protocol Deviations

AbbVie does not allow intentional/prospective deviations from the protocol unless when necessary to eliminate an immediate hazard to study subjects. The Principal Investigator is responsible for complying with all protocol requirements, and applicable global and local laws regarding protocol deviations. If a protocol deviation occurs (or is identified, including those that may be due to the COVID-19 or any pandemic or any state of



emergency situation) after a subject has been enrolled, the Principal Investigator is responsible for notifying IEC/IRB regulatory authorities (as applicable), and the following AbbVie Clinical Contacts:

Primary Contact: Alternate Contact: Study Project Manager II Study Management Associate III AbbVie S.r.l AbbVie Inc. Via dell'Arte 25 00144 Roma 1 North Waukegan Road North Chicago, IL 60064 Italy Office: Office: Fax: Fax: Email: Email:

Such contact must be made as soon as possible to permit a review by AbbVie to determine the impact of the deviation on the subject and/or the study.

Examples of protocol deviations include the following:

- Subject entered into the study even though she/he did not satisfy entry criteria;
- Subject who developed withdrawal criteria during the study and was not withdrawn;
- Subject who received wrong treatment or incorrect dose;
- Subject who received excluded or prohibited concomitant treatment.

In Japan, the Investigator will record all protocol deviations in the appropriate medical records at site.



# 8.0 Statistical Methods and Determination of Sample Size

#### 8.1 Statistical and Analytical Plans

A global analysis will be conducted for the comparisons of upadacitinib 15 mg QD and 30 mg QD treatment groups versus the MTX treatment group for all subjects (excluding the Japan specific upadacitinib 7.5 mg treatment group). A separate Japan sub-study analysis will be conducted for the comparisons of upadacitinib 7.5 mg QD, 15 mg QD, and 30 mg QD treatment groups versus the MTX treatment group for subjects enrolled in Japan only.

An unblinded analysis will be conducted after all subjects have completed Week 24 for the purpose of regulatory submission. To maintain integrity of the trial and avoid introduction of bias, study sites and subjects will remain blinded for the duration of Period 1. Additional unblinded analyses may be conducted after the Week 24 analysis.

Completed and specific details of the statistical analysis will be described and fully documented in the Statistical Analysis Plan (SAP). The SAP will be finalized prior to the database lock for the primary analysis at Week 24. The statistical analyses will be performed using SAS (SAS Institute Inc., Cary, NC, USA).

Starting with Amendment 6, subjects receiving upadacitinib 15 mg and 30 mg QD will receive open-label upadacitinib 15 mg QD. Starting with Amendment 6 subjects receiving MTX will receive open-label MTX. The details for handling the change in dose in analysis will be described in the Statistical Analysis Plan (SAP) for final reporting.

#### 8.1.1 Analysis Populations

#### 8.1.1.1 Full Analysis Set

The Full Analysis Set (FAS) includes all randomized subjects who received at least one dose of study drug. The FAS will be used for all efficacy and baseline analyses.



#### 8.1.1.2 Per Protocol Analysis Set

The Per Protocol Analysis Set represents a subset of the FAS and consists of all FAS subjects who did not meet any major protocol violations during the study. Definitions of major protocol violations will be detailed in the SAP. Additional analysis may be conducted on the Per Protocol analysis set, in order to evaluate the impact of major protocol violations.

# 8.1.1.3 Safety Analysis Set

The Safety Analysis Set consists of all subjects who received at least one dose of study drug. For the Safety Analysis Set, subjects are assigned to a treatment group based on the treatment actually received, regardless of the treatment randomized.

# 8.1.2 Subject Accountability, Disposition and Study Drug Exposure

# 8.1.2.1 Subject Accountability

The following will be summarized by site and by treatment group as well as overall, separately for Period 1 and Period 2: number of subjects randomized, the number of subjects who received at least one dose of study drug, the number of subjects who completed, the number of subjects who prematurely discontinued study drug, and the number of subjects who prematurely discontinued study participation.

#### 8.1.2.2 Subject Disposition

Separately for Period 1 and Period 2, the number and percentage of subjects who are randomized, received at least one dose of study drug, prematurely discontinued study participation, and completed will be summarized by treatment group and overall. Reasons for premature discontinuation of study drug and study participation will be summarized separately for all randomized subjects by treatment group and overall, with frequencies and percentages by reason for discontinuation.



## 8.1.2.3 Study Drug Exposure

Exposure to study drug will be summarized for the Safety Analysis Set for Period 1 alone as well as for Period 1 and Period 2 combined. The exposure to study drug (days) will be summarized with the mean, standard deviation, median, and range for each treatment group.

Study drug compliance will be summarized for each treatment group for Period 1. The compliance is defined as the number of tablets/capsules taken (i.e., the difference between the number of tablets/capsules dispensed and the number of tablets/capsules returned) during the subject's participation in Period 1 divided by the number of tablets/capsules a subject is supposed to take each day/week times the length of time that the subject was in the Treatment Phase of Period 1.

# 8.1.3 Analysis of Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized by treatment group and overall for the FAS. For the purpose of this analysis, baseline data for each subject will be the data collected immediately prior to the first dose of study drug in Period 1.

Summary statistics for continuous variables will include the number of observations, mean, standard deviation, median, and range. For discrete variables, frequencies and percentages for each category will be summarized.

Medical history will be presented by counts and percentages of subjects, broken down by Body System and Diagnosis.

Prior therapy and medication will be summarized by treatment group. Prior therapy and medication will include all therapies and medications with a start date prior to the date of first dose of study drug.

Concomitant medications will also be summarized with frequencies and percentages for each treatment group. All medications administered during study drug exposure will be included.



#### 8.1.4 Efficacy Analysis

All efficacy analyses will be carried out using the FAS population, which includes all randomized subjects who receive at least one dose of study drug.

## 8.1.4.1 Efficacy Analysis for Period 1

# 8.1.4.1.1 Primary Efficacy Variables

The primary endpoints for US/FDA, EU/EMA, and Japan/PMDA regulatory purposes are listed in Section 5.3.3.1.1. Analyses will be conducted separately for US/FDA, EU/EMA and Japan/PMDA regulatory purposes; for each set of analyses, only the specified primary endpoint is applicable.

The analysis of the primary efficacy endpoint will be conducted on the FAS based on treatment as randomized. Supportive analysis will also be conducted on the Per Protocol Analysis Set. For the analysis of ACR20, ACR50 and CR, the comparisons will be made between each upadacitinib dose and the MTX group using the Cochran-Mantel-Haenszel test adjusting for main stratification factors. Non-Responder Imputation (NRI) will be used as the primary analysis. For the analysis of change from baseline in mTSS, between-group comparisons for each upadacitinib treatment group and the MTX treatment group will be performed using the analysis of covariance model with treatment group as the fixed factor, and the corresponding baseline value and the main stratification factors as the covariates. Both linear extrapolation analysis and as observed analysis will be conducted.

The primary efficacy analyses will be performed in demographic subgroups including age, gender, weight, body mass index, race, and geographical region to assess the consistency of the treatment effect. Additional subgroup analyses based on baseline disease characteristics and stratification factors will also be conducted.

# 8.1.4.1.2 Key Secondary Efficacy Variables

Key secondary endpoints for US/FDA, EU/EMA, and Japan/PMDA regulatory purposes regulatory purposes are listed in Section 5.3.3.1.2.



For binary endpoints, frequencies and percentages will be reported for each treatment group. Similar analyses as for the primary endpoint will be conducted.

For continuous endpoints, the mean, standard deviation, median, and range will be reported for each treatment group. Between-group comparisons for each upadacitinib treatment group and the MTX treatment group will be performed using the analysis of covariance model with treatment groups as the fixed factor, and the corresponding baseline value and the main stratification factors as the covariates.

See Section 8.1.4.1.5 for imputation methods.

#### 8.1.4.1.3 Other Efficacy Variables

Additional efficacy variables are listed in Section 5.3.3.1.3 and will be summarized for all visits, including visits beyond Week 24. For binary endpoints, frequencies and percentages will be reported for each treatment group. For continuous endpoints, the change from baseline mean, standard deviation, median, and range will be reported for each treatment group.

# 8.1.4.1.4 Multiplicity Control for the Primary and Ranked Key Secondary Endpoints

For the global analysis of upadacitinib 15 mg QD and 30 mg QD compared to MTX (excluding the Japan specific upadacitinib 7.5 mg treatment group), the overall type I error rate of the primary and ranked key secondary endpoints for the two doses will be strongly controlled using a graphical multiple testing procedure. Specifically, the testing will utilize the endpoint sequence of primary endpoint(s) followed by the ranked key secondary endpoints in the order as specified in Section 5.3.3.1.2, and will begin with testing the primary endpoint using  $\alpha$  of 0.025 for each dose. Continued testing will follow a pre-specified  $\alpha$  transfer path which includes downstream transfer along the endpoint sequence within each dose as well as cross-dose transfer. More details of the graphical procedure will be specified in the SAP.



#### 8.1.4.1.5 Imputation Methods

The following methods will be used for missing data imputation:

**Observed Cases (OC):** The OC analysis will not impute values for missing evaluations, and thus a subject who does not have an evaluation on a scheduled visit will be excluded from the OC analysis for that visit.

**Multiple Imputation (MI):** The MI analysis imputes missing data multiple times under appropriate random variation and thus generate multiple imputed "pseudo-complete" datasets. Results will be aggregated across the multiple imputed datasets, overcoming drawbacks of the single imputation methods.

**Non-Responder Imputation (NRI):** NRI applies to binary endpoints only. In NRI analysis, subjects who prematurely discontinue study drug will be considered non-responders after discontinuation.

**Linear Extrapolation for Radiographic Data:** For radiographic data (i.e., mTSS-based endpoints), if a subject receives rescue therapy or prematurely discontinued, the radiographic data at time points after rescue or discontinuation will be imputed assuming a linear relationship between baseline and previous time point when X-ray should be collected.

For non-radiographic data, the NRI approach will serve as the primary analysis approach for key binary endpoints. The MI approach will serve as the primary analysis approach for key continuous endpoints. Sensitivity analysis based on OC will also be conducted for key endpoints. For radiographic data, analysis based on both linear extrapolation and an as-observed analysis (where the as-observed Week 24/48 assessments for all subjects are used) will be conducted.

# 8.1.4.2 Long-Term Efficacy for Period 1 and Period 2 Combined

The efficacy endpoints of long-term efficacy analysis are listed in Section 5.3.3.2 and will be summarized for all visits.



Long-term efficacy by time point will be summarized using descriptive statistics. For binary endpoints, frequencies and percentages will be summarized. For continuous endpoints, the mean and standard deviation will be reported.

#### 8.1.5 Safety Analysis

#### 8.1.5.1 General Considerations

Safety analyses will be carried out using the Safety Analysis Set. Analyses will be conducted for Period 1 alone, as well as for Period 1 and Period 2 combined.

Safety analyses are based on treatments actually received. Safety will be assessed by AEs, physical examination, laboratory assessments, ECG, and vital signs. Frequency tables and lists of subjects with treatment-emergent AEs by preferred term as in the Medical Dictionary for Regulatory Activities (MedDRA) dictionary, by system organ class, by severity, and by relationship to the study drug as assessed by the Investigator will be provided. The changes from baseline in vital signs, physical examination results, and clinical laboratory values will be analyzed in a descriptive manner. Shift of laboratory values from baseline to defined time points will be tabulated.

Missing safety data will not be imputed.

#### 8.1.5.2 Analysis of Adverse Events

Unless otherwise specified, the following conventions apply for both the Period 1 safety analysis and the combined safety analysis of Period 1 and Period 2.

# 8.1.5.2.1 Treatment-Emergent Adverse Events (TEAE)

AEs will be coded using MedDRA. A TEAE is defined as AE that began or worsened in severity after initiation of study drug.

AEs starting more than 30 days following the last dose of study drug will not be included in summaries of TEAEs. For subjects who continued into Period 2, AEs that are reported in Period 2 will be summarized in the combined safety analysis of Period 1 and Period 2.



As a general safety summary, the number and percentage of subjects experiencing TEAEs will be summarized for each treatment group for the following AE categories:

- All AEs;
- All severe AEs;
- All reasonably possibly related AEs;
- All SAEs;
- Frequent AEs (reported in 2% of subjects or more in any treatment group);
- Frequent reasonably possibly related AEs (reported in 5% of subjects or more in any treatment group);
- Discontinuations due to AEs;
- Death.

Additional AEs may be considered for tabulation/summary based on recommendations from Clinical and Safety as deemed appropriate.

TEAEs will be summarized and presented by system organ classes (SOCs) and preferred terms (PTs) using MedDRA. The SOCs will be presented in alphabetical order, and the PTs will be presented in alphabetical order within each SOC.

TEAE will also be summarized by maximum severity and by maximum relationship.

The AEs of special interest (including but not limited to serious infection, opportunistic infection, herpes zoster, TB, gastrointestinal perforations, malignancies, MACE, renal dysfunction, anemia, increased CPK, drug-related hepatic disorders, and embolic and thrombotic events (non-cardiac, non-CNS)) will be summarized. Event rate (per 100 patient years) for AEs of special interest will also be summarized for the combined safety analysis of Period 1 and Period 2.

All AEs leading to discontinuation of study drug will be presented in listing format. A listing by treatment group of TEAEs grouped by SOC and MedDRA preferred term with subject identification numbers will be generated.



#### 8.1.5.2.2 Serious Adverse Events and Death

All treatment-emergent SAEs and AEs leading to death will also be presented in listing format. In addition, SAEs will be summarized by SOC and MedDRA PT.

## 8.1.5.3 Analysis of Laboratory, Vital Sign, and ECG Data

Changes from baseline by visit, and changes from baseline to minimum value, maximum value, and final values in continuous laboratory data, and vital signs will be summarized by treatment group.

Baseline values are defined as the last non-missing measurements recorded on or before the date of the first dose of study drug in Period 1.

The laboratory data will be categorized as Grade 1, Grade 2, Grade 3, and Grade 4 according to OMERACT criteria (Rheumatology Common Toxicity Criteria v.2.0). For creatine phosphokinase, and serum creatinine, NCI CTC criteria will be used. The shift tables will tabulate the number and percentage of subjects with baseline and post-baseline values by grade level.

Listings will be provided for potentially clinically significant laboratory values and vital signs.

# 8.1.6 Pharmacokinetic and Exposure-Response Analyses

Individual upadacitinib plasma concentrations at each study visit will be tabulated and summarized with appropriate statistical methods.

Data from this study may be combined with data from other studies for the population PK and exposure-response analyses. Population PK and exposure-response analyses of only data from this study may not be conducted. The following general methodology will be used for the population PK and exposure-response analyses.

Population PK analyses will be performed using the actual sampling time relative to dosing. PK models will be built using a non-linear mixed-effects modeling approach with



NONMEM software (Version 7, or a higher version). The structure of the starting PK model will be based on the PK analysis of data from previous studies. The CL/F and V/F of upadacitinib will be the PK parameters of major interest in the analyses. If necessary, other parameters, including the parameters describing absorption characteristics, may be fixed if useful in the analysis.

The evaluation criteria described below will be used to examine the performance of different models.

- 1. The objective function of the best model is significantly smaller than the alternative model(s).
- 2. The observed and predicted concentrations from the preferred model are more randomly distributed across the line of unity (a straight line with zero intercept and a slope of one) than the alternative model(s).
- 3. Visual inspection of model fits standard errors of model parameters and change in inter-subject and intra-subject error.

Once an appropriate base PK model (including inter- and intra-subject error structure) is developed, empirical Bayesian estimates of individual model parameters will be calculated by the posterior conditional estimation technique using non-linear mixed-effects modeling. The relationship between these conditional estimates CL/F and V/F values with only potentially physiologically relevant or clinically meaningful covariates (such as subject age, sex, body weight, concomitant medications, laboratory markers of hepatic of renal function, etc.) will be explored using stepwise forward selection method, or another suitable regression/smoothing method at a significance level of 0.05. After identification of all relevant covariates, a stepwise backward elimination of covariates from the full model will be employed to evaluate the significance (at P < 0.005, corresponding to a decrease in objective function > 7.88 for one degree of freedom) of each covariate in the full model.



Linear or non-linear relationships of primary PK parameters with various covariates will be explored.

Relationships between upadacitinib exposure and clinical observations (primary efficacy variable) will be explored. Exposure-response relationships for secondary efficacy variables and/or some safety measures of interest may also be explored. The relationship between exposure (e.g., population PK model predicted average concentrations, area under the curve, trough concentrations, the individual model-predicted PK profiles, or some other appropriate measure of exposure) and drug effect will be explored. Several classes of models (e.g., linear, log-linear, exponential,  $E_{max}$ , sigmoid  $E_{max}$ , etc.) will be evaluated to characterize the exposure-response relationship based on observed data. Results of the PK and exposure-response analyses may be summarized in a separate report prior to regulatory filing of upadacitinib for the treatment of RA, rather than in the CSR.

Additional analyses will be performed if useful and appropriate.

## 8.2 Determination of Sample Size

The planned sample size of 900 (not including the Japan specific upadacitinib 7.5 mg QD treatment group) provides at least 90% power for a 20% difference in ACR50 response rate (assuming a Week 12 MTX ACR50 rate of 20%). This sample size also provides at least 90% power for a 16% difference in DAS28 CR response rate (assuming a Week 24 MTX CR rate of 24%), and for a 20% difference in ACR20 response rate (assuming a Week 12 MTX ACR20 rate of 50%). With this sample size, there is approximately 80% power to detect a difference of 0.58 in change from baseline in mTSS (assuming a standard deviation of 2.2). This sample size will also provide at least 90% power for other ranked key secondary endpoints including change from baseline in DAS28 (CRP), change from baseline in HAQ-DI, ACR70, and SF-36. The above power calculations are all based on a two-sided significance level of 0.025 and accounting for a 10% dropout rate. An additional 75 Japanese subjects will be enrolled into the Japan specific upadacitinib 7.5 mg QD treatment arm for Japan/PMDA regulatory purposes.



#### 8.3 Randomization Methods

Subjects will be randomly assigned in a 1:1:1 ratio to treatment Groups 2, 3, and 4, below, except for subjects from Japan, who will be randomized in a 2:1:1:1 ratio to Groups 1, 2, 3, and 4:

- Group 1: Upadacitinib 7.5 mg QD monotherapy (subjects in Japan only; N = 75)
- Group 2: Upadacitinib 15 mg QD monotherapy (N = 300) (includes 37 subjects from Japan)
- Group 3: Upadacitinib 30 mg QD monotherapy (N = 300) (includes 37 subjects from Japan)
- Group 4: MTX monotherapy (N = 300) (includes 37 subjects from Japan)

Randomization will be stratified by geographic region.

See Section 5.5.3 for details.

#### 9.0 Ethics

# 9.1 Independent Ethics Committee (IEC) or Institutional Review Board (IRB)

Good Clinical Practice requires that the clinical protocol, any protocol amendments, the Investigator's Brochure, the informed consent, and all other forms of subject information related to the study (e.g., advertisements used to recruit subjects) and any other necessary documents be reviewed by an IEC/IRB. The IEC/IRB will review the ethical, scientific and medical appropriateness of the study before it is conducted. IEC/IRB approval of the protocol, informed consent, and subject information and/or advertising, as relevant, will be obtained prior to the authorization of drug shipment to a study site.

Any amendments to the protocol will require IEC/IRB approval prior to implementation of any changes made to the study design. The investigator will be required to submit,



maintain and archive study essential documents according to International Conference on Harmonization (ICH) GCP.

Any SAEs that meet the reporting criteria, as dictated by local regulations, will be reported to both responsible Ethics Committees and Regulatory Agencies, as required by local regulations. During the conduct of the study, the Investigator should promptly provide written reports (e.g., ICH Expedited Reports, and any additional reports required by local regulations) to the IEC/IRB of any changes that affect the conduct of the study and/or increase the risk to subjects. Written documentation of the submission to the IEC/IRB should also be provided to AbbVie.

## 9.2 Ethical Conduct of the Study

The study will be conducted in accordance with the protocol, ICH guidelines, applicable regulations and guidelines governing clinical study conduct and the ethical principles that have their origin in the Declaration of Helsinki. Responsibilities of the clinical investigator are specified in Appendix A.

In the event a significant disaster/crisis (e.g., epidemic/pandemic, natural disaster, conflict/combat) occurs leading to difficulties in performing protocol-specified procedures, AbbVie may engage with study site personnel in efforts to ensure the safety of subjects, maintain protocol compliance, and minimize risks to the integrity of the study while trying to best manage subject continuity of care. This may include alternative methods for assessments (e.g., virtual site visits), alternative locations for data collection (e.g., use of a local lab instead of a central lab), and shipping investigational product and/or supplies direct to subjects to ensure continuity of treatment where allowed. In all cases, these alternative measures must be allowed by local regulations and permitted by IRB/IEC. Investigators should notify AbbVie if any urgent safety measures are taken to protect the subjects against any immediate hazard.



#### 9.3 Subject Information and Consent

The Investigator or his/her representative will explain the nature of the study to the subject, and answer all questions regarding this study. Prior to any study-related screening procedures being performed on the subject, the informed consent statement will be reviewed and signed and dated by the subject, the person who administered the informed consent, and any other signatories according to local requirements. A copy of the informed consent will be given to the subject and the original will be placed in the subject's medical record. An entry must also be made in the subject's dated source documents to confirm that informed consent was obtained prior to any study-related procedures and that the subject received a signed copy.

Information regarding incentives for subjects and information regarding provisions for treating and/or compensating subjects who are harmed as a consequence of participation in the study can be found in the informed consent.

Samples for exploratory research/validation studies will only be collected if the subject has voluntarily signed and dated the separate written consent for exploratory research/validation studies, approved by an IRB/IEC, after the nature of the testing has been explained and the subject has had an opportunity to ask questions. The separate written consent must be signed before the exploratory research/validation studies samples are collected and testing is performed. The separate written consent may be part of the main consent form. If the subject does not consent to the exploratory research/validation studies, it will not impact the subject's participation in the study.

In the event a subject withdraws from the main study, optional exploratory research samples will continue to be stored and analyzed unless the subject specifically withdraws consent for the optional samples. If consent is withdrawn for the optional sampling, the subject must inform their study doctor, and once AbbVie is informed, the optional samples will be destroyed. However, if the subject withdraws his/her consent and the samples have already been tested, those results will still remain as part of the overall research data.



Due to a pandemic situation like COVID-19 or state of emergency, it is possible that additional protocol modifications not outlined in this protocol may become necessary. If this situation arises, in addition to the study informed consent, additional verbal consent may be obtained prior to these adaptations or substantial changes in study conduct in accordance with local regulations.

# 9.3.1 Informed Consent Form and Explanatory Material

In Japan, the Principal Investigator will prepare the informed consent and explanatory material required to obtain subject's consent to participate in the study with the cooperation of the sponsor and will revise these documents as required. The prepared or revised consent forms and explanatory material will be submitted to the sponsor. Approval of the IRB will be obtained prior to use in the study.

## 9.3.2 Revision of the Consent Form and Explanatory Material

In Japan, when important new information related to the subject's consent becomes available, the Principal Investigator will revise the informed consent and explanatory material based on the information without delay and will obtain the approval of the IRB prior to use in the study. The Investigator will provide the information, without delay, to each subject already participating in the study, and will confirm the intention of each subject to continue the study or not. The Investigator shall also provide a further explanation using the revised form and explanatory material and shall obtain written consent from each subject of their own free will to continue participating in the study.

# 10.0 Source Documents and Case Report Form Completion

#### 10.1 Source Documents

Source documents are defined as original documents, data and records. This may include joint evaluation form, hospital records, clinical and office charts, laboratory data/information, subjects' diaries or evaluation checklists, pharmacy dispensing and other records, recorded data from automated instruments, microfiches, photographic negatives,



microfilm or magnetic media, and/or x-rays. Data collected during this study must be recorded on the appropriate source documents.

The Investigator(s)/Institution(s) will permit study-related monitoring, audits, IEC/IRB review, and regulatory inspection(s), providing direct access to source data documents.

During the COVID-19 pandemic or any pandemic/state of emergency, remote monitoring of data may be employed if allowed by the local regulatory authority, IRB/IEC, and the study site.

#### 10.2 Case Report Forms

Case report forms (CRFs) must be completed for each subject screened/enrolled in this study. These forms will be used to transmit information collected during the study to AbbVie and regulatory authorities, as applicable. The CRF data for this study are being collected with an EDC system called Rave® provided by the technology vendor Medidata Solutions Incorporated, NY, USA. The EDC system and the study-specific eCRFs will comply with Title 21 CFR Part 11. The documentation related to the validation of the EDC system is available through the vendor, Medidata, while the validation of the study-specific eCRFs will be conducted by AbbVie and will be maintained in the Trial Master File at AbbVie.

The Investigator will document subject data in his/her own subject files. These subject files will serve as source data for the study. All eCRF data required by this protocol will be recorded by investigative site personnel in the EDC system. All data entered into the eCRF will be supported by source documentation.

The Investigator or an authorized member of the investigator's staff will make any necessary corrections to the eCRF. All change information, including the date and person performing the corrections, will be available via the audit trail, which is part of the EDC system. For any correction, a reason for the alteration will be provided. The eCRFs will be reviewed periodically for completeness, legibility, and acceptability by AbbVie personnel (or their representatives). AbbVie (or their representatives) will also be allowed


access to all source documents pertinent to the study in order to verify eCRF entries. The Principal Investigator will review the eCRFs for completeness and accuracy and provide his or her electronic signature and date to eCRFs as evidence thereof.

Medidata will provide access to the EDC system for the duration of the study through a password-protected method of internet access. Such access will be removed from investigator sites at the end of the site's participation in the study. Data from the EDC system will be archived on appropriate data media (CD-ROM, etc.) and provided to the Investigator at that time as a durable record of the site's eCRF data. It will be possible for the Investigator to make paper printouts from that media.

Patient and site reported data must be completed for each subject screened/enrolled in this study.

- The following data are being collected with an Electronic Patient-Reported Outcome (ePRO) system called Trialmax, provided by the technology vendor CRF Health of Plymouth Meeting, PA, USA:
  - o Completed by Patient:
    - Patient Global Assessment of Disease Activity VAS
    - Patient's Assessment of Pain VAS
    - HAQ-DI
    - SF-36
    - FACIT-F
    - WPAI
    - EQ-5D-5L
  - Completed by Site:
    - Physician Global Assessment of Disease Activity VAS
- The following data will be completed by the patient on paper and entered into the EDC system:
  - Patient's Assessment of Severity and Duration of Morning Stiffness



The ePRO system is in compliance with Title 21 CFR Part 11. The documentation related to the system validation of the ePRO system is available through the vendor, CRF Health, while the user acceptance testing of the study-specific PRO design will be conducted and maintained at AbbVie.

The subject will be entering the data on an electronic device; these data will be uploaded to a server. The data on the server will be considered source and will be maintained and managed by CRF Health.

Internet access to the ePRO data will be provided by CRF Health for the duration of the trial. This access will be available for the duration of the trial to the site investigator, as well as delegated personnel. Such access will be removed from investigator sites following the receipt of the study archive. Data from the ePRO system will be archived on appropriate data media (CD-ROM, etc.) and provided to the investigator at that time as a durable record of the site's ePRO data. It will be possible for the investigator to make paper print-outs from that media.

The ePRO data will be collected by the following method:

#### Tablet Based

• The instrument/scale will be collected electronically via a tablet device into which the subject will directly enter the required pieces of information. The electronic device will be programmed to allow data entry for only the visits specified in the protocol and will not allow for subjects to complete more than one of the same assessment at any one visit. All data entered on the device will be immediately stored to the device itself and automatically uploaded to a central server administrated by CRF Health. The Investigator and delegated staff will be able to access all uploaded subject entered data via a password protected website, up until the generation, receipt and confirmation of the study archive.



### 11.0 Data Quality Assurance

Prior to the initiation of the study, a meeting may be held with AbbVie personnel, the investigators and appropriate site personnel. This meeting may include a detailed discussion of the protocol, performance of study procedures, CRF, subject dosing diary, and specimen collection methods. Another alternative of site training may include module training via a study portal.

The AbbVie monitor will monitor each site throughout the study. Source document review will be performed against entries on the CRF and a quality assurance check will be performed to ensure that the Investigator is complying with the protocol and regulations.

Data hand entered in the database will be verified at AbbVie. Any discrepancies will be reviewed against the CRF and corrected on-line. After completion of the entry process, computer logic and manual checks will be created by AbbVie to identify items such as inconsistent study dates. Any necessary corrections will be made by the site to the eCRF.

Routine hematology, serum chemistry and serology, and urinalysis, and other tests such as rheumatoid factor, anti-CCP, and HBV/HCV testing, will be conducted using a central laboratory (refer to Appendix D and Appendix F). The data from these analyses will be electronically transferred from the central laboratory to the study database.

Laboratory tests including, but not limited to, urine pregnancy testing and ESR, will be conducted locally by each study site (refer to Appendix D and Appendix F). Sites will provide AbbVie with laboratory certifications and normal ranges for each local laboratory used. The full name, address, phone number and fax number for each local laboratory will also be included.

#### 12.0 Use of Information

Any research that may be done using exploratory research/validation studies samples from this study will be experimental in nature and the results will not be suitable for clinical decision making or patient management. Hence, the subject will not be informed of



individual results, should analyses be performed, nor will anyone not directly involved in this research. Correspondingly, researchers will have no access to subject identifiers. Individual results will not be reported to anyone not directly involved in this research other than for regulatory purposes. Aggregate data from exploratory research/validation studies may be provided to investigators and used in scientific publications or presented at medical conventions. Exploratory research/validation studies information will be published or presented only in a way that does not identify any individual subject.

### 13.0 Completion of the Study

The Investigator will conduct the study in compliance with the protocol and complete the study within the timeframe specified in the contract between the Investigator (Director of the Site in Japan) and AbbVie. Continuation of this study beyond this date must be mutually agreed upon in writing by both the Investigator (Director of the Site in Japan) and AbbVie. The Investigator will provide a final report to the IEC/IRB following conclusion of the study, and will forward a copy of this report to AbbVie or their representative.

The Investigator (Director of the Site in Japan) must retain any records related to the study according to local requirements. If the Investigator (Director of the Site in Japan) is not able to retain the records, he/she must notify AbbVie to arrange alternative archiving options.

AbbVie will select the signatory Investigator from the Investigators who participate in the study. Selection criteria for this Investigator will include level of participation as well as significant knowledge of the clinical research, investigational drug, and study protocol. The signatory Investigator for the study will review and sign the final study report in accordance with the European Agency for the Evaluation of Medicinal Products Guidance on Investigator's Signature for Study Reports.

The end-of-study is defined as the date of the last subject's last visit.



# 14.0 Investigator's Agreement

- 1. I have received and reviewed the Investigator's Brochure for upadacitinib.
- 2. I have read this protocol and agree that the study is ethical.
- 3. I agree to conduct the study as outlined and in accordance with all applicable regulations and guidelines.
- 4. I agree to maintain the confidentiality of all information received or developed in connection with this protocol.
- 5. I agree that all electronic signatures will be considered the equivalent of a handwritten signature and will be legally binding.

Protocol Title: A Phase 3, Randomized, Double-Blind Study Comparing

Upadacitinib (ABT-494) Once Daily Monotherapy to MTX

Monotherapy in MTX-Naïve Subjects with Moderately to Severely

Active Rheumatoid Arthritis

Protocol Date: 03 December 2020

| Signature of Principal Investigator | Date |
|---------------------------------------------------|------|
| Name of Principal Investigator (printed or typed) | |



#### 15.0 Reference List

- 1. Grigor C, Capell H, Stirling A, et al. Effect of treatment strategy of tight control for rheumatoid arthritis (the TICORA study): a single-blind randomised controlled trial. Lancet. 2004;364(9430):263-9.
- 2. Vermeer M, Kuper HH, Bernelot Moens HJ, et al. Adherence to a treat-to-target strategy in early rheumatoid arthritis: results of the DREAM remission induction cohort. Arthritis Res Ther. 2012;14(6):R254.
- 3. Verstappen SM, Jacobs JW, van der Veen MJ, et al. Intensive treatment with methotrexate in early rheumatoid arthritis: aiming for remission. Computer Assisted Management in Early Rheumatoid Arthritis (CAMERA, an open-label strategy trial). Ann Rheum Dis. 2007;66:1143-9.
- 4. Aletaha D, Neogi T, Silman AJ, et al. 2010 rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Ann Rheum Dis. 2010;69(9):1580-8.
- 5. Burmester GR, Feist E, and Dorner T. Emerging cells and cytokine targets in rheumatoid arthritis. Nat Rev Rheumatol. 2014;10(2):77-88.
- 6. Emery P. Why is there persistent disease despite biological therapy? Importance and early intervention. Arthritis Res Ther. 2014;16(3):115.
- 7. Meier FM, McInnes IB. Small-molecule therapeutics in rheumatoid arthritis: scientific rationale, efficacy and safety. Best Pract Res Clin Rheumatol. 2014;28(4):605-24.
- 8. Vaddi K, Luchi M. JAK inhibition for the treatment of rheumatoid arthritis: a new era in oral DMARD therapy. Expert Opin Investig Drugs. 2012;21(7):961-73.
- 9. Murray PJ. The Jak-STAT signaling pathway: input and output integration. J Immunol. 2007;178(5):2623-9.
- 10. Xeljanz® (tofacitinib) [package insert] New York, NY; Pfizer Labs, 2015.



- 11. Nawendy N, Krishnaswai S, Wang R, et al. Effect of CP-690,550, an orally active janus kinase inhibitor, on renal function in healthy adult volunteers. J Clin Pharmacol. 2009;49(4):423-9.
- 12. Greenwald MK, Fidelus-Gort R, Levy R, et al. A randomized dose-ranging, placebo-controlled study of INCB028050, a selective JAK1 and JAK2 inhibitor in subjects with active rheumatoid arthritis [abstract]. Arthritis Rheum. 2010;62 (Suppl 10):2172.
- 13. Dougados M, van der Heijde D, Chen YC, et al. Baricitinib, an oral janus kinase (JAK)1/JAK2 inhibitor, in patients with active rheumatoid arthritis (RA) and an inadequate response to CDMARD therapy: results of the phase 3 RA-build study. Ann Rheum Dis. 2015;74 (Suppl 2):79.
- 14. Genovese MC, Kremer J, Zamani O, et al. Baricitinib, an oral janus kinase (JAK)1/JAK2 inhibitor, in patients with active rheumatoid arthritis (RA) and an inadequate response to TNF inhibitors: results of the phase 3 RA-beacon study. Ann Rheum Dis. 2015;74 (Suppl 2):75.
- 15. Fleischmann R, Kremer J, Cush J, et al. Placebo-controlled trial of tofacitinib monotherapy in rheumatoid arthritis. N Engl J. Med. 2012;367(6):495-507.
- 16. van Vollenhoven RF, Fleischmann R, Cohen S, et al. Tofacitinib or adalimumab versus placebo in rheumatoid arthritis. N Engl J Med. 2012;367(6):508-19.
- 17. Burmester GR, Blanco R, Charles-Schoeman C, et al. Tofacitinib (CP-690,550) in combination with methotrexate in patients with active rheumatoid arthritis with an inadequate response to tumour necrosis factor inhibitors: a randomized phase 3 trial. Lancet. 2013;381(9865):451-60.
- 18. Kremer J, Li Z-G, Hall S, et al. Tofacitinib in combination with nonbiologic disease-modifying antirheumatic drugs in patients with active rheumatoid arthritis. Ann Intern Med. 2013;159(4):253-61.



- 19. van der Heijde D, Tanaka Y, Fleischmann R, et al. Tofacitinib (CP-690,550) in patients with rheumatoid arthritis receiving methotrexate: twelve month data from a twenty-four-month phase III randomized radiographic study. Arthritis Rheum. 2013;65(3):559-70.
- 20. Galapagos [press release]. 14 April 2015. Available from: http://www.glpg.com/files/1314/2904/2940/PR\_Darwin1\_April\_14\_2015\_FINAL. pdf. Accessed on: 02 September 2015.
- 21. Galapagos [press release]. 27 April 2015. Available from: http://www.glpg.com/files/3514/3016/6234/PR\_Darwin2\_FINAL.pdf. Accessed on: 02 September 2015.
- 22. Woodworth T, Furst DE, Alten R, et al. Standardizing assessment and reporting of adverse effects in rheumatology clinical trials II: the Rheumatology Common Toxicity Criteria v.2.0. J Rheumatol. 2007;34(6):1401-14.
- 23. Bretz F, Maurer W, Brannath W, et al. A graphical approach to sequentially rejective multiple test procedures. Stat Med. 2009;28(4):586-604.



#### **Appendix A.** Responsibilities of the Clinical Investigator

Clinical research studies sponsored by AbbVie are subject to the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) Good Clinical Practices (GCP) and local regulations and guidelines governing the study at the site location. In signing the Investigator Agreement in Section 14.0 of this protocol, the investigator is agreeing to the following:

- 1. Conducting the study in accordance with the relevant, current protocol, making changes in a protocol only after notifying AbbVie, except when necessary to protect the safety, rights or welfare of subjects.
- 2. Personally conducting or supervising the described investigation(s).
- 3. Informing all subjects, or persons used as controls, that the drugs are being used for investigational purposes and complying with the requirements relating to informed consent and ethics committees (e.g., independent ethics committee [IEC] or institutional review board [IRB]) review and approval of the protocol and amendments.
- 4. Reporting adverse experiences that occur in the course of the investigation(s) to AbbVie and the site director.
- 5. Reading the information in the Investigator's Brochure/safety material provided, including the instructions for use and the potential risks and side effects of the investigational product(s).
- 6. Informing all associates, colleagues, and employees assisting in the conduct of the study about their obligations in meeting the above commitments.
- 7. Maintaining adequate and accurate records of the conduct of the study, making those records available for inspection by representatives of AbbVie and/or the appropriate regulatory agency, and retaining all study-related documents until notification from AbbVie.



- 8. Maintaining records demonstrating that an ethics committee reviewed and approved the initial clinical investigation and all amendments.
- 9. Reporting promptly, all changes in the research activity and all unanticipated problems involving risks to human subjects or others, to the appropriate individuals (e.g., coordinating investigator, institution director) and/or directly to the ethics committees and AbbVie.
- 10. Following the protocol and not make any changes in the research without ethics committee approval, except where necessary to eliminate apparent immediate hazards to human subjects.



# **Appendix B.** List of Protocol Signatories

| Name | Title | Functional Area |
|---|---|---|
| | Executive Medical Director | Immunology Clinical Development |
| | Medical Director | Therapeutic Area |
| | Senior Medical Director | Pharmacovigilance and Patient Safety |
| | Director, Statistics | Statistics |
| | Senior Director, Immunology<br>Therapeutic Area Head | Statistics |
| | Assistant Director, Clinical Pharmacology | Clinical Pharmacokinetics and Pharmacodynamics |
| | Study Project Manager | Clinical Program Development |



#### **Appendix C.** Local Requirements

#### Canada

Section 5.2.1 Inclusion Criteria

- 10. If female of childbearing potential, subject must be practicing two forms of contraception (one highly effective method combined with one effective method, refer to Contraception Recommendations for Females below) that are effective from Study Day 1 through at least 180 days after the last dose of study drug.
- 11. Male subjects who are sexually active with female partner(s) of childbearing potential must agree from Study Day 1 through 180 days after the last dose of study drug to practice the protocol-specified contraception (refer to Contraception Recommendations for Males below).

Section 5.2.4 Contraception Recommendations

#### **Contraception Recommendation for Females**

A woman who is postmenopausal or permanently surgically sterile (bilateral oophorectomy, bilateral salpingectomy or hysterectomy) is not considered to be a woman of childbearing potential and is not required to follow contraception recommendations. Postmenopausal is defined as:

- Age ≥ 55 years with no menses for 12 or more months without an alternative medical cause; or
- Age < 55 years with no menses for 12 or more months without an alternative medical cause AND an FSH level > 40 mIU/mL.

If the female subject is < 55 years of age:

AND has had no menses for  $\geq 12$  months AND has no history of permanent surgical sterilization (defined above), FSH should be tested at Screening.



- If FSH is not tested, it is assumed that the subject is of childbearing potential and protocol-specified contraception is required.
- If the FSH is tested and the result is consistent with post-menopausal status, contraception is not required.
- If the FSH is tested and the result is consistent with pre-menopausal status, contraception is required and a serum pregnancy test must be performed (see Section 5.3.1.1 pregnancy test).

#### For a female subject at any age:

- Female subjects with menses within the past 12 months are of childbearing potential and FSH is therefore not required but contraception is required.
- Female subjects who are surgically sterile (defined above) are not of childbearing potential and therefore no FSH testing or contraception is required.

A woman who does not meet the definition of postmenopausal or permanently surgically sterile is considered of childbearing potential and is required to use two forms of contraception. This includes one form of highly effective contraception and one effective method of contraception that are effective from Study Day 1 (or earlier) through at least 180 days after the last dose of study drug.

- Highly effective methods:
  - Hormonal contraceptives started at least 2 months prior to randomization (e.g., combined [estrogen and progestogen containing] oral contraceptives, patch, vaginal ring, injectables, and implants);
  - Intrauterine device (IUD) or intrauterine system (IUS);
  - Vasectomy and tubal ligation.
- Effective methods:
  - O Barrier methods of contraception (e.g., male condom, female condom, cervical cap, diaphragm, contraceptive sponge).



Note: The proper use of diaphragm or cervical cap includes use of spermicide and is considered one barrier method. The cervical cap and contraceptive sponge are less effective in parous women. The use of spermicide alone is not considered a suitable barrier method for contraception. When used consistently and correctly, "double barrier" methods of contraception (e.g., male condom with diaphragm, male condom with cervical cap) can be used as an effective alternative to the highly effective contraception methods described above. Male and female condoms should not be used together as they can tear of become damaged.

#### **Contraception Recommendation for Males**

There are no contraception requirements for male subjects receiving upadacitinib only, or their female partner(s).

For a male subject receiving MTX who has a female partner who is postmenopausal or permanently sterile, no contraception is required.

A male subject receiving MTX who is sexually active with female partner(s) of childbearing potential must agree from Study Day 1 through 180 days after the last dose of MTX study drug to practice contraception with:

• Condom use and female partner(s) using at least one of the highly effective contraceptive methods as defined in the protocol for female study subjects of childbearing potential.

Additionally, male subjects receiving MTX must agree not to donate sperm from Study Day 1 through 180 days after the last dose of MTX study drug.

Male subjects receiving MTX are responsible for informing his partner(s) of the risk of becoming pregnant and for reporting any pregnancy to the study doctor.

#### Colombia

Section 5.2.1 Inclusion Criteria



- 10. If female of childbearing potential, subject must be practicing two forms of contraception (one highly effective method combined with one effective method, refer to Contraception Recommendations for Females below) that are effective from Study Day 1 through at least 180 days after the last dose of study drug.
- 11. Male subjects who are sexually active with female partner(s) of childbearing potential must agree from Study Day 1 through 180 days after the last dose of study drug to practice the protocol-specified contraception (refer to Contraception Recommendations for Males below).

#### Section 5.2.4 Contraception Recommendations

#### **Contraception Recommendation for Females**

A woman who is postmenopausal or permanently surgically sterile (bilateral oophorectomy, bilateral salpingectomy or hysterectomy) is not considered to be a woman of childbearing potential and is not required to follow contraception recommendations.

#### Postmenopausal is defined as:

- Age  $\geq$  55 years with no menses for 12 or more months without an alternative medical cause; or
- Age < 55 years with no menses for 12 or more months without an alternative medical cause AND an FSH level > 40 mIU/mL.

A woman who does not meet the definition of postmenopausal or permanently surgically sterile is considered of childbearing potential and is required to practice at least one of the following highly effective methods of birth control that is effective from Study Day 1 (or earlier) through at least 180 days after the last dose of study drug.

• Combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal, injectable) associated with the inhibition of ovulation, initiated at least 30 days prior to Study Day 1.



- Progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation, initiated at least 30 days prior to Study Day 1.
- Bilateral tubal occlusion/ligation.
- Vasectomized partner(s), provided the vasectomized partner has received medical confirmation of the surgical success and is the sole sexual partner of the women of childbearing potential trial participant.
- Intrauterine device (IUD).
- Intrauterine hormone-releasing system (IUS).

A second form of contraception (barrier) such as a male or female condom with or without spermicide OR cap, diaphragm or sponge with spermicide should be used in addition to one of the highly effective birth control methods listed above.

#### **Contraception Recommendation for Males**

There are no contraception requirements for male subjects receiving upadacitinib only, or their female partner(s).

For a male subject receiving MTX who has a female partner who is postmenopausal or permanently sterile, no contraception is required.

A male subject receiving MTX who is sexually active with female partner(s) of childbearing potential must agree from Study Day 1 through 180 days after the last dose of MTX study drug to practice contraception with:

• Condom use and female partner(s) using at least one of the contraceptive measures (as defined in the protocol for female study subjects of childbearing potential).

Additionally, male subjects receiving MTX must agree not to donate sperm from Study Day 1 through 180 days after the last dose of MTX study drug.



Obbvie Upadacitinib
M13-545 Protocol Amendment 8 EudraCT 2015-003334-27

Male subjects receiving MTX are responsible for informing his partner(s) of the risk of becoming pregnant and for reporting any pregnancy to the study doctor.



# **Appendix D.** Study Activities (Period 1)

| | Screening | BL | Wk<br>2 | Wk<br>4 | Wk<br>8 | Wk<br>12 | Wk<br>16 | Wk<br>20 | Wk<br>24 | Wk<br>26 | Wk<br>28 | Wk<br>32 | Wk<br>36 | Wk<br>40 | Wk 48/<br>PD <sup>a</sup> | 30-Day |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Activity | D -35 to<br>D -1 | D1 <sup>b</sup> | D15 | D29 | D57 | D85 | D113 | D141 | D169 | D183 | D197 | D225 | D253 | D281 | D337 | F/U<br>Visit <sup>c</sup> |
| Informed consent <sup>d</sup> | X | | | | | | | | | | | | | | | |
| Inclusion/exclusion criteria | X | X | | | | | | | | | | | | | | |
| Medical/surgical history <sup>e</sup> | X | X | | | | | | | | | | | | | | |
| Alcohol and nicotine use | X | | | | | | | | | | | | | | | |
| Adverse event assessment <sup>f</sup> | Only<br>SAEs and<br>protocol-<br>related<br>nonserious<br>AEs | X | X | X | X | X | X | X | X | X | X | X | X | X | X | Х |
| Prior/concomitant therapy | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X <sup>g</sup> | X |
| Patient questionnaires <sup>h</sup> PtGA Pain (VAS) HAQ-DI Morning Stiffness (severity and duration) | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Patient questionnaires <sup>h</sup> EQ-5D-5L FACIT-F WPAI SF-36 | | X | | | | X | | | X | | | | | | X | |



# Obbie Upadacitinib M13-545 Protocol Amendment 8 EudraCT 2015-003334-27

| | Screening D -35 to | BL | Wk<br>2 | Wk<br>4 | Wk<br>8 | Wk<br>12 | Wk<br>16 | Wk<br>20 | Wk<br>24 | Wk<br>26 | Wk<br>28 | Wk<br>32 | Wk<br>36 | Wk<br>40 | Wk 48/<br>PD <sup>a</sup> | <b>30-Day</b><br>F/U |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Activity | D -1 | D1 <sup>b</sup> | D15 | D29 | D57 | D85 | D113 | D141 | D169 | D183 | D197 | D225 | D253 | D281 | D337 | Visit <sup>c</sup> |
| Latent TB risk assessment form <sup>i</sup> | X | | | | | | | | | | | | | | X | |
| Central lab QuantiFERON-TB Gold test <sup>i</sup> (and/or local PPD skin test) | X | | | | | | | | | | | | | | X <sup>i</sup> | |
| Chest x-ray <sup>j</sup> | X | | | | | | | | | | | | | | X <sup>j</sup> | |
| 12-lead ECG <sup>k</sup> | X | | | | | | | | | | | | | | $X^k$ | |
| X-rays (bilateral hands/feet) | X <sup>l</sup> | | | | | | | | X <sup>m</sup> | | | | | | X <sup>m</sup> | |
| Height (screening only) and weight | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Vital signs <sup>n</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Physical exam <sup>o</sup> | X | X | | | | | | | | | | | | | X | |
| Physician Global<br>Assessment (PhGA) | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| TJC68/SJC66 | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Serum pregnancy test at central lab <sup>p</sup> | X | | | | | | | | | | | | | | | |
| Local urine pregnancy test <sup>q</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Central Lab Tests hsCRP <sup>r</sup> Blood chemistry <sup>s</sup> Hematology (CBC) Urinalysis <sup>t</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |



Obbie Upadacitinib M13-545 Protocol Amendment 8 EudraCT 2015-003334-27

| | Screening | BL | Wk<br>2 | Wk<br>4 | Wk<br>8 | Wk<br>12 | Wk<br>16 | Wk<br>20 | Wk<br>24 | Wk<br>26 | Wk<br>28 | Wk<br>32 | Wk<br>36 | Wk<br>40 | Wk 48/<br>PD <sup>a</sup> | 30-Day |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Activity | D -35 to<br>D -1 | D1 <sup>b</sup> | D15 | D29 | D57 | D85 | D113 | D141 | D169 | D183 | D197 | D225 | D253 | D281 | D337 | F/U<br>Visit <sup>c</sup> |
| ESR (local lab) | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Other Central Lab Tests Rheumatoid factor Anti-CCP autoantibodies HBV/HCV screening | X | | | | | | | | | | | | | | | |
| HIV local lab (if required) <sup>u</sup> | X <sup>u</sup> | | | | | | | | | | | | | | | |
| VZV skin test <sup>v</sup> and VZV specific IgG <sup>w</sup> | X | | | | | | | | | | | | | | | |
| IgG and IgM (central lab) | | X | | | X | | | | X | | | | | | X | |
| Blood samples for upadacitinib PK assay | | | X <sup>x</sup> | X <sup>x</sup> | | X <sup>y</sup> | X <sup>y</sup> | X <sup>y</sup> | X <sup>y</sup> | | | X <sup>y</sup> | X <sup>y</sup> | X <sup>y</sup> | X <sup>y</sup> | |
| Blood samples for<br>exploratory research and<br>validation studies (optional<br>– see Appendix E) <sup>z</sup> | | X | X | | X | | | | X | | | | | | X | |
| Randomization/Drug assignment | | X | | | | | | | | | | | | | | |
| Calculation for rescue based on TJC/SJC | | | | | | X <sup>aa</sup> | X <sup>aa</sup> | X <sup>aa</sup> | X <sup>aa</sup> | | | | X <sup>aa</sup> | X <sup>aa</sup> | | |
| Calculation for drug<br>assignment based on<br>TJC/SJC and CDAI | | | | | | | | | | X <sup>bb</sup> | | | | | | |
| Dispense study drug and subject dosing diary | | X | | X | X | X | X | X | X | X | X | X | X | X | X <sup>cc</sup> | |



| | Screening | BL | Wk<br>2 | Wk<br>4 | Wk<br>8 | Wk<br>12 | Wk<br>16 | Wk<br>20 | Wk<br>24 | Wk<br>26 | Wk<br>28 | Wk<br>32 | Wk<br>36 | Wk<br>40 | Wk 48/<br>PD <sup>a</sup> | 30-Day |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Activity | D -35 to<br>D -1 | D1 <sup>b</sup> | D15 | D29 | D57 | D85 | D113 | D141 | D169 | D183 | D197 | D225 | D253 | D281 | D337 | F/U<br>Visit <sup>c</sup> |
| Review and copy subject<br>dosing diary and perform<br>drug reconciliation | | | | X | X | X | X | X | X | X | X | X | X | X | X | |

BL = Baseline Visit; CBC = complete blood count; CCP = cyclic citrullinated peptide; D = Day; ECG = electrocardiogram; EQ-5D-5L = EuroQoL-5D; ESR = erythrocyte sedimentation rate; FACIT-F = Functional Assessment of Chronic Illness Therapy – Fatigue; F/U = Follow-up; HAQ-DI = Health Assessment Questionnaire – Disability Index; HBV = hepatitis B virus; HCV = hepatitis C virus; HIV = human immunodeficiency virus; hsCRP = high-sensitivity C-reactive protein; NRS = numerical rating scale; PD = Premature Discontinuation (completely from study [withdrawal of consent]); PhGA = Physician's Global Disease Activity; PK = pharmacokinetics; PPD = purified protein derivative; PtGA = Patient's Global Assessment of Disease Activity; SAE = serious adverse event; SF-36 = 36-Item Short Form Health Survey; SJC = Swollen Joint Count; TB = tuberculosis; TJC = Tender Joint Count; VAS = visual analog scale; VZV = varicella zoster virus; Wk = Week; WPAI = Work Productivity and Activity Impairment

- a. Subjects may withdraw from the study completely (withdrawal of informed consent) or may discontinue study drug treatment, but may choose to continue to participate in the study (refer to Section 5.4.1 for additional details). If a subject is prematurely discontinued from study drug, the procedures outlined for the Premature Discontinuation visit (PD visit) should be completed as soon as possible, preferably within 2 weeks of study drug discontinuation.
- b. The Baseline Visit procedures will serve as the reference for all subsequent visits with the exception of the ECG and x-rays of hands and feet, which will be obtained at Screening only and used as the baseline reference (see also footnote l regarding x-rays of the hands and feet at Screening).
- c. This visit is 30 days after last dose of study drug for those subjects who prematurely discontinue from study drug and study participation. A 30-day follow-up phone call may occur for subjects who prematurely discontinued from study drug and study participation to determine the status of any ongoing AEs/SAEs or the occurrence of any new AEs/SAEs.
- d. Informed consent should be obtained at Screening prior to performing any study related procedures.
- e. Also note herpes zoster and hepatitis B vaccination status in medical history.
- f. Collect serious adverse events and protocol-related nonserious AEs that occur after a subject signs the informed consent, prior to the first dose of study drug.
- g. At Week 48 (after Week 48 assessments have been performed), per Investigator judgment, may add csDMARDs (concomitant use of up to 2 csDMARDs, except the combination of MTX and leflunomide), or increasing csDMARD dose.
- h. Prior to other procedures. For morning stiffness, duration will be captured only if NRS rating is > 0.
- i. Refer to Section 5.3.1.1 Study Procedures TB Testing for specific requirements for TB testing and TB prophylaxis. QuantiFERON-TB Gold test (and/or PPD skin test) is not required at the PD visit.



- j. The screening chest x-ray will not be required if a subject had a previous normal chest-x-ray within 90 days of Screening, provided that all source documentation is available at the site (refer to Section 5.3.1.1 Chest X-Ray for specific requirements). At Week 48, obtain chest x-ray for subjects with TB risk factors as identified by the TB risk assessment form or for subjects living in areas endemic for TB or for subjects with a newly positive QuantiFERON-TB Gold test (and/or PPD skin test) after baseline. A chest x-ray is not required at the PD visit.
- k. For subjects with a normal ECG taken within 90 days of Screening, a repeat ECG at Screening will not be required, provided all source documentation is available. Refer to Section 5.3.1.1 12-Lead ECG for additional details. All subjects will have an ECG at Week 48 and PD visit as applicable.
- 1. X-rays of hands and feet must be performed during the screening process. Subjects are eligible for the study if the locally read screening x-rays confirms the presence of ≥ 1 bone erosion OR in the absence of the documented bone erosion, both positive RF and positive anti-CCP autoantibodies are required. Screening x-rays will serve as baseline x-rays for scoring purposes. Refer to Section 5.3.1.1 Study Procedures X-Rays of Hands and Feet for additional details.
- m. For handling of x-rays during the study, please refer to Section 5.3.1.1.
- n. Blood pressure, pulse rate, body temperature, and respiratory rate should be performed before blood draws are performed.
- o. A full physical exam is required at the visits indicated. A symptom-directed physical exam may be performed when necessary.
- p. For all women of childbearing potential, collect serum for pregnancy test at screening. If serum pregnancy test comes back borderline, a repeat test is necessary (pregnancy is an exclusion criterion). Refer to Section 5.3.1.1 Study Procedures Pregnancy Test for additional details.
- q. For all women of childbearing potential, collect urine for pregnancy test at Baseline and all subsequent visits. If urine pregnancy test (which is performed at the site) is negative, begin or continue dosing. If urine pregnancy test is positive, withhold dosing and perform a serum pregnancy test. Pregnant subjects must permanently discontinue study drug. Refer to Section 5.3.1.1 Study Procedures Pregnancy Test for additional details.
- r. Central lab hsCRP results will remain blinded to the Sponsor, Investigator, study site personnel, and subject for all visits except Screening. Results of tests such as hsCRP may be blunted in subjects taking a JAK inhibitor, thereby limiting the clinical utility of these tests in the setting of a possible safety assessment or adverse event management. Any local hsCRP or local CRP tests should not be reported to the investigator until treatment allocation is unblinded.
- s. Minimum 8-hour fast. If a subject is not able to fast when necessary, due to unforeseen circumstances, the non-fasting status will be recorded in study source documentation.
- t. A urine dipstick macroscopic urinalysis will be completed by the central laboratory at all required visits. A microscopic analysis will be performed in the event the dipstick results show leukocytes, nitrite, protein, ketones, or blood greater than negative or glucose greater than normal.
- u. If required by country regulatory authorities to confirm eligibility, subjects will be tested for antibodies to HIV at Screening, and it should be documented that the test has been performed. This testing is to be done at a local lab. A subject will not be eligible for study participation if test results indicate a positive HIV infection. AbbVie will not receive results from the testing and will not be made aware of any positive result.
- v. For subjects in Japan only, VZV skin test will be performed locally at Screening.
- w. For subjects in Japan only, VZV specific IgG will be measured centrally at Screening.



Upadacitinib M13-545 Protocol Amendment 8 EudraCT 2015-003334-27

- x. At Week 2 and Week 4 Visits, PK samples should be collected prior to dosing and the subjects should take the study drug dose at the clinic after collecting the PK blood sample. However, if the subject normally takes the study drug dose at a time that is after the time of the scheduled study visit, the subject should follow the regular dosing schedule and the PK sample should be collected at any time during the visit.
- y. PK samples should be collected at any time during the visit. Subject should follow the regular dosing schedule.
- z. Samples only collected if subject provides written consent.
- aa. Rescue therapy is clearly outlined for subjects who meet the criteria described in Section 5.2.3.3.
- bb. Rescue therapy for those subjects who meet the following criteria at Week 26 is described in Section 5.2.3.3.
- cc. For subjects entering Period 2.

Note: Visit window is ± 3 days for the first 32 weeks and ± 7 days for the remainder of Period 1. Any of the procedures may be performed at an unscheduled visit at the discretion of the Investigator. Subjects who choose to discontinue study drug treatment, but continue to participate in the study, should complete a Premature Discontinuation Visit (PD Visit) as soon as possible, preferably within 2 weeks. Refer to Section 5.1 Discontinuation of Study Drug and Continuation of Study Participation (Period 1 and Period 2) for additional details.



#### Appendix E. Study Activities – Optional Samples for Exploratory Research and Validation Studies (Period 1 Only)

| | Screening | BL | Wk<br>2 | Wk<br>4 | Wk<br>8 | Wk<br>12 | Wk<br>16 | Wk<br>20 | Wk<br>24 | Wk<br>26 | Wk<br>28 | Wk<br>32 | Wk<br>36 | Wk<br>40 | Wk<br>48/PD |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Activity | D -35 to<br>D -1 | D1 | D15 | D29 | D57 | D85 | D113 | D141 | D169 | D183 | D197 | D225 | D253 | D281 | D337 |
| Pharmacogenetic samples <sup>a,b</sup> | | X | | | | | | | | | | | | | |
| Epigenetic samples <sup>b</sup> | | X | X | | X | | | | X | | | | | | X |
| Transcriptomic and epigenetic samples <sup>b</sup> | | X | X | | X | | | | X | | | | | | X |
| Plasma samples for proteomic and targeted protein investigations <sup>b</sup> | | X | X | | X | | | | X | | | | | | X |
| Serum samples for proteomic and targeted protein investigations <sup>b</sup> | | X | X | 1 | X | | - | | X | | | | | - | X |

BL = Baseline Visit; D = Day; PD = Premature Discontinuation; Wk = Week

Note: Collections to be performed only if subject provides separate written consent to collect the exploratory research/validation studies samples; if the separate consent is not signed, no samples can be collected. The separate written consent may be part of the main consent form.

a. The sample is preferred to be collected at BL, but can be drawn at any time during the subject's participation.

b. Based on the value of the different technologies, samples may also be used to assess other biomarker signatures, including but not limited to metabolomics, lipidomics, and other approaches. Samples may be used for assay of study drugs if needed.



# **Appendix F.** Study Activities (Period 2)

| Activity | Wk<br>60 | Wk<br>72 | Wk<br>84 | Wk<br>96 | Every<br>12 Weeks <sup>a</sup> | Monthly | Every<br>24 Weeks <sup>a</sup> | Every<br>48 Weeks <sup>a</sup> | Wk<br>192 | Final<br>(Wk 260)/<br>PD Visit <sup>o</sup> | 30-Day<br>F/U<br>Visit <sup>b</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Adverse event assessment | X | X | X | X | X | | | | | X | X |
| Concomitant therapy | X | X | X | X | X | | | | | X | X |
| Patient questionnaires <sup>c</sup> PtGA Pain (VAS) HAQ-DI Morning stiffness (severity and duration) | X | X | X | X | X | | | | | X | |
| Latent TB risk assessment form <sup>d</sup> | | | | X <sup>d</sup> | | | | X <sup>d</sup> | | | |
| Central lab QuantiFERON-TB<br>Gold test <sup>d</sup> (and/or local PPD skin<br>test) | | | | X <sup>d</sup> | | | | X <sup>d</sup> | | | |
| Chest x-ray <sup>e</sup> | | | | Xe | | | | Xe | | | |
| 12-lead ECG <sup>f</sup> | | | | Xf | | | | X <sup>f</sup> | | X | |
| X-rays (bilateral hands/feet) | | | | X | | | | | X | $X^g$ | |
| Vital signs and body weight <sup>h</sup> | X | X | X | X | X | | | | | X | X |
| Physical exam <sup>i</sup> | | X | | X | | | Xi | | | X | |
| Physician Global Assessment (PhGA) | X | X | X | X | X | | | | | X | |
| TJC68/SJC66 | X | X | X | X | X | | | | | X | |
| Local urine pregnancy test <sup>j</sup> | X | X | X | X | X | | | | | X | X |



| Activity | Wk<br>60 | Wk<br>72 | Wk<br>84 | Wk<br>96 | Every<br>12 Weeks <sup>a</sup> | Monthly | Every<br>24 Weeks <sup>a</sup> | Every<br>48 Weeks <sup>a</sup> | Wk<br>192 | Final<br>(Wk 260)/<br>PD Visit <sup>o</sup> | 30-Day<br>F/U<br>Visit <sup>b</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|
| At-home urine pregnancy test <sup>j</sup> | | | | | | X | | | | | |
| Central lab tests hsCRP <sup>k</sup> Blood chemistry <sup>l</sup> Hematology (CBC) Urinalysis <sup>m</sup> | X | X | X | X | X | | | | | X | X |
| ESR (local lab) | X | X | X | X | X | | | | | X | |
| Calculation for drug assignment based on TJC/SJC and CDAI | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | X <sup>n</sup> | | | | | | |
| Dispense study drug and subject dosing diary | X | X | X | X | X | | | | | | |
| Review and copy subject dosing diary and perform drug reconciliation | X | X | X | X | X | | | | | X | |

CBC = complete blood count; ECG = electrocardiogram; ESR = erythrocyte sedimentation rate; F/U = Follow-up; HAQ-DI = Health Assessment Questionnaire – Disability Index; hsCRP = high-sensitivity C-reactive protein; PD = Premature Discontinuation; PhGA = Physician's Global Disease Activity; PPD = purified protein derivative; PtGA = Patient's Global Assessment of Disease Activity; SJC = Swollen Joint Count; TB = tuberculosis; TJC = Tender Joint Count; VAS = visual analog scale; Wk = Week

- a. Every 12, 24, or 48 weeks, from the Week 96 Visit through Week 240.
- b. This visit is 30 days after last dose of study drug for those subjects who complete Period 2. A 30-day follow-up phone call may occur for subjects who prematurely discontinue from study drug and study participation to determine the status of any ongoing AEs/SAEs or the occurrence of any new AEs/SAEs.
- c. Prior to other procedures. For morning stiffness, duration will be captured only if NRS rating is > 0.
- d. TB testing should be performed every 48 weeks after Week 96 in subjects with previous negative QuantiFERON-TB Gold and/or PPD tests. Subjects with new evidence of latent TB should initiate prophylactic treatment immediately per local guidelines. Refer to Section 5.3.1.1 TB Testing/TB Prophylaxis for additional details. Study drug(s) should not be withheld at the time of the first positive TB test.



Upadacitinib M13-545 Protocol Amendment 8 EudraCT 2015-003334-27

- e. Obtain chest x-ray every 48 weeks after Week 96 for subjects with TB risk factors as identified by the TB risk assessment form, or for subjects living in areas endemic for TB, or for subjects with a newly positive QuantiFERON-TB Gold test (and/or PPD skin test) after baseline.
- f. ECGs will be performed every 48 weeks after Week 96. An ECG may be performed at any visit if deemed necessary by the Investigator.
- g. Subjects who prematurely discontinue from Period 2 will undergo an x-ray of hands and feet unless the previous x-ray was performed within the previous 24 weeks.
- h. Blood pressure, pulse rate, body temperature, and respiratory rate should be performed before blood draws are performed.
- i. A full physical exam is required every 24 weeks after Week 96. A symptom-directed physical exam may be performed when necessary.
- j. For women of childbearing potential, a urine pregnancy test will be performed at all visits and monthly at home between scheduled study visits. The results of the monthly at home tests will be communicated to the site. If a urine pregnancy test is positive, the subject must stop dosing, come in to the clinic and have blood drawn for a serum pregnancy test that will be analyzed at the central laboratory. Pregnant subjects must discontinue from study drug treatment. Refer to Section 5.3.1.1 Study Procedures Pregnancy Test for additional details.
- k. hsCRP results will remain blinded to Sponsor, Investigator, study site personnel, and the subject for all visits until the last subject reaches the end of Period 1.
- 1. Minimum 8-hour fast. If a subject is not able to fast when necessary, due to unforeseen circumstances, the non-fasting status will be recorded in study source documentation.
- m. Dipstick urinalysis will be completed by the central lab at all required visits. Specified abnormal macroscopic urinalyses defined as leukocytes, nitrite, protein, ketones, or blood greater than negative, or glucose greater than normal will be followed up with a microscopic analysis at the central laboratory.
- n. Starting at Week 48, subjects who fail to show at least 20% improvement in both TJC and SJC compared to baseline at 2 consecutive visits, despite optimization of background RA therapies, will be discontinued from study drug. Refer to Section 5.1.
- o. Subjects may withdraw from the study completely (withdrawal of informed consent) or may discontinue study drug treatment, but may choose to continue to participate in the study (refer to Section 5.4.1 for additional details).

Note: Visit window is ± 7 days for Period 2. Any of the procedures may be performed at an unscheduled visit at the discretion of the Investigator. Subjects who choose to discontinue study drug treatment, but continue to participate in the study, should complete a Premature Discontinuation Visit (PD Visit) as soon as possible, preferably within 2 weeks. Refer to Section 5.1 Discontinuation of Study Drug and Continuation of Study Participation (Period 1 and Period 2) for additional details.



# Appendix G. Physician's Global Assessment of Disease Activity Example Visual Analog Scale (VAS)

VAS will be used to assess the physician's global assessment of disease activity. The VAS consists of a horizontal 100 mm line anchored at either end by opposite adjectives reflecting the spectrum/severity of the parameters assessed:

• Physician's global assessment of disease activity (current status)

The Physician will rate global assessment of subject's current disease activity ranging from 0 to 100 (see example below)

| Mark the line below to indicate the subject's rheur | natoid arthritis disease activity |
|---|---|
| (independent of the subject's self-assessment). | |
| 0 | 100 |
| U | 100 |
| Very Low | Very High |



# Appendix H. Joint Evaluation Worksheet Example

| | | J | OINT | EVA | LUAT | ION | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 5 | Subjec | t Rigl | ıt | | | | Subje | ct Lef | t | |
| JOINT | Pa | 0 = Ab<br>1 = Pre | | | Rep<br>NA | ) =<br>laced<br>= No<br>ssment | Pa | 0 = Ab<br>1 = Pre | | | Rep<br>NA | =<br>laced<br>= No<br>ssment |
| (Tick Correct Answer) | Tend | erness | Swe | lling | Jo | int | Tend | erness | Swe | lling | Jo | int |
| Temporomandibular | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 2. Sternoclavicular | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 3. Acromio-clavicular | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 4. Shoulder | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 5. Elbow | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 6. Wrist | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 7. Metacarpophalangeal I | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 8. Metacarpophalangeal II | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 9. Metacarpophalangeal III | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 10. Metacarpophalangeal IV | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 11. Metacarpophalangeal V | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 12. Thumb Interphalangeal | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 13. Prox. Interphalangeal II | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 14. Prox. Interphalangeal III | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 15. Prox. Interphalangeal IV | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 16. Prox. Interphalangeal V | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 17. Distal Interphalangeal II | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 18. Distal Interphalangeal III | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 19. Distal Interphalangeal IV | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 20. Distal Interphalangeal V | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 21. Hip | 0 | 1 | | | 9 | NA | 0 | 1 | | | 9 | NA |
| 22. Knee | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 23. Ankle | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 24. Tarsus | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 25. Metatarsophalangeal I | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 26. Metatarsophalangeal II | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |



| JOINT EVALUATION | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 5 | Subjec | t Rigl | ht | | | | Subje | ct Lef | t | |
| | | 0 = Absent<br>1 = Present | | | | ) =<br>laced<br>= No<br>ssment | | 0 = Ab<br>1 = Pre | | | Rep<br>NA | =<br>laced<br>= No<br>ssment |
| JOINT<br>(Tick Correct Answer) | | nin/<br>erness | Swelling | | Joint | | Pain/<br>Tenderness | | Swe | lling | Joint | |
| 27. Metatarsophalangeal III | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 28. Metatarsophalangeal IV | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 29. Metatarsophalangeal V | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 30. Interphalangeal I | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 31. Interphalangeal II | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 32. Interphalangeal III | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 33. Interphalangeal IV | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 34. Interphalangeal V | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| TOTAL Joint Count | | | | | | | | | | | | |



#### **Appendix I.** Latent TB Risk Assessment Form Example

- 1. Have you or an immediate family member or other close contact ever been diagnosed or treated for tuberculosis?
- 2. Have you lived in or had prolonged travels to countries in the following regions:
  - Sub-Saharan Africa
  - India
  - China
  - Mexico
  - Southeast Asia or Micronesia
  - The former Soviet Union
- 3. Have you lived or worked in a prison, homeless shelter, immigration center, or nursing home?
- 4. Have you, or an immediate family member, had any of the following problems for the past 3 weeks or longer:
  - Chronic Cough
  - Production of Sputum
  - Blood-Streaked Sputum
  - Unexplained Weight Loss
  - Fever
  - Fatigue/Tiredness
  - Night Sweats
  - Shortness of Breath

 $From: http://www mayoclinic.com/health/tuberculosis/DS00372/DSECTION=risk-factors \\ http://www.in.gov/fssa/files/Tuberculosis\_Questionnaire.pdf$ 



#### Appendix J. Patient's Global Assessment of Disease Activity Example

#### Visual Analog Scale (VAS)

VAS will be used to assess the subject's global assessment of disease activity. Each VAS consists of a horizontal 100 mm line anchored at either end by opposite adjectives reflecting the spectrum/severity of the parameters assessed:

• Subject's global assessment of disease activity (within last 24 hours)

The subject will rate the severity of the RA symptoms and how he/she is doing from 0 to 100. This assessment will be used for the DAS28 (CRP) calculation in this study (see example below):

Please place a vertical mark on the line below to indicate how well your rheumatoid arthritis has been doing during THE LAST 24 HOURS:

| 0 | 100 |
|-----------|-------------|
| Very Well | Very Poorly |



#### **Appendix K.** Patient's Assessment of Pain Example

#### **Visual Analog Scale (VAS)**

VAS will be used to assess the subject's assessment of pain. Each VAS consists of a horizontal 100 mm line anchored at either end by opposite adjectives reflecting the spectrum/severity of the parameters assessed:

How much pain have you had because of your condition within the previous week?

Place a mark on the line below to indicate how severe your pain has been.

| NO | WORST |
|------|----------|
| | POSSIBLE |
| PAIN | PAIN |



#### Appendix L. Health Assessment Questionnaire (HAQ-DI) Example

## **HEALTH ASSESSMENT QUESTIONNAIRE**

In this section we are interested in learning how your illness affects your ability to function in daily life.

Please check the response which best describes your usual abilities OVER THE PAST WEEK:

WITHOUT ANY WITH SOME WITH MUCH UNABLE DIFFICULTY DIFFICULTY TO DO

DRESSING AND GROOMING

| <b>DRESSING AND GROOMING</b> | |
|---|---|
| Are you able to: | |
| Dress yourself, including tying shoelaces and doing buttons? | |
| Shampoo your hair? | |
| ARISING | |
| Are you able to: | |
| Stand up from a straight chair? | |
| Get in and out of bed? | |
| <b>EATING</b> | |
| Are you able to: | |
| Cut your own meat? | |
| Lift a full cup or glass to your mouth? | |
| Open a new milk carton? | |
| WALKING | |
| Are you able to: | |
| Walk outdoors on flat ground? | |
| Climb up five steps? | |
| Please check any AIDS OR DEVICES that you usually use for any of these activities: | |
| Cane | Devices used for dressing (button hook, zipper pull, long handled shoe horn, etc.) |
| ☐ Walker | ☐ Built up or special utensils |
| ☐ Crutches | ☐ Special or built up chair |
| Wheelchair Other (Specify:) | |



Upadacitinib
M13-545 Protocol Amendment 8
EudraCT 2015-003334-27

| Please check any categories for which you usually need HELP FROM ANOTHER PERSON: | | | | |
|---|---|---|---|---|
| Dressing and Grooming | Eating | | | |
| ☐ Arising | ☐ Walkin | g | | |
| Please check the response which best describes your usual abilities OVER THE PAST WEEK: | | | | |
| | WITHOUT ANY | WITH SOME | WITH MUCH | UNABLE |
| | DIFFICULTY | DIFFICULTY | DIFFICULTY | TO DO |
| <u>HYGIENE</u> | | | | |
| Are you able to: | | | | |
| Wash and dry your body? | | | | |
| Take a tub bath? | | | | |
| Get on and off the toilet? | | | | |
| <u>REACH</u> | | | | |
| Are you able to: | | | | |
| Reach and get down a 5-pound object (such as a bag of sugar) from just above your head? | | | | |
| Bend down to pick up clothing from the floor? | | | | |
| <u>GRIP</u> | | | | |
| Are you able to: | | | | |
| Open car doors? | | | | |
| Open jars which have been previously opened? | | | | |
| Turn faucets on and off? | | | | |
| <u>ACTIVITIES</u> | | | | |
| Are you able to: | | | | |
| Run errands and shop? | | | | |
| Get in and out of a car? | | | | |
| Do chores such as vacuuming or yard work? | | | | |
| Please check any AIDS OR DE | VICES that you usi | ially use for any of | these activities: | |
| ☐ Raised toilet seat | | ☐ Bathtub bar | | |
| ☐ Bathtub seat | | ☐ Long-handled appliances for reach | | |
| ☐ Jar opener (for jars previousl | y opened) | ☐ Long-handled appliances in bathroom | | |
| | | Other (Specify: _ | | _) |



# Upadacitinib M13-545 Protocol Amendment 8 EudraCT 2015-003334-27

| Please check any categories for which you usually need HELP FROM ANOTHER PERSON: | |
|---|---|
| Hygiene | ☐ Gripping and opening things |
| Reach | ☐ Errands and chores |
| HAQ – United States/English | |
| HAO-DL AUI 0-eng-USori doc © Stanford University | V |


EudraCT 2015-003334-27

# Appendix M. Patient's Assessment of Severity and Duration of Morning Stiffness Example

#### **Instructions:**

Please clearly mark an 'x' in the box  $(\boxtimes)$  that best describes your experience with morning stiffness on awakening in the past 7 days.

| No morning stiffness | g | | | | | | | | | ossible m<br>stiffness | orning |
|---|---|---|---|---|---|---|---|---|---|---|---|
| ▼ | | | | | | | | | | ▼ | |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |

When you experience morning stiffness, how long does it take to get as limber as possible: \_\_\_ hours \_\_\_ minutes



### Appendix N. EuroQoL-5D Example

Under each heading, please check the ONE box that best describes your health TODAY:

| Mobility | |
|---|---|
| I have no problems walking | |
| I have slight problems walking | |
| I have moderate problems walking | |
| I have severe problems walking | |
| I am unable to walk | |
| Self-Care | |
| I have no problems washing or dressing myself | |
| I have slight problems washing or dressing myself | |
| I have moderate problems washing or dressing myself | |
| I have severe problems washing or dressing myself | |
| I am unable to wash or dress myself | |
| Usual Activities (e.g., work, study, housework, family or leisure | e activities) |
| I have no problems with doing my usual activities | |
| I have slight problems with doing my usual activities | |
| I have moderate problems with doing my usual activities | |
| I have severe problems with doing my usual activities | |
| I am unable to do my usual activities | |



Pain/Discomfort I have no pain or discomfort I have slight pain or discomfort I have moderate pain or discomfort I have severe pain or discomfort I have extreme pain or discomfort **Anxiety/Depression** I am not anxious or depressed I am slightly anxious or depressed I am moderately anxious or depressed I am severely anxious or depressed I am extremely anxious or depressed 

- We would like to know how good or bad your health is TODAY.
- This scale is numbered from 0 to 100.
- 100 means the <u>best</u> health you can imagine.
   0 means the <u>worst</u> health you can imagine.
- Mark an X on the scale to indicate how your health is TODAY.
- Now, please write the number you marked on the scale in the box below.

YOUR HEALTH TODAY =

# The best health you can imagine



The worst health you can imagine



# Appendix O. Functional Assessment of Chronic Illness Therapy – Fatigue (FACIT-F) Scale Example

Below is a list of statements that other people with your illness have said are important. Please circle or mark one number per line to indicate your response as it applies to the <u>past 7 days</u>.

| | | | A little<br>bit | Some-<br>what | Quite<br>a bit | Very<br>much |
|---|---|---|---|---|---|---|
| HI7 | I feel fatigued | 0 | 1 | 2 | 3 | 4 |
| HI12 | I feel weak all over | 0 | 1 | 2 | 3 | 4 |
| Anl | I feel listless ("washed out") | 0 | 1 | 2 | 3 | 4 |
| An2 | I feel tired | 0 | 1 | 2 | 3 | 4 |
| An3 | I have trouble starting things because I am tired | 0 | 1 | 2 | 3 | 4 |
| As4 | I have trouble <u>finishing</u> things because I am tired. | 0 | 1 | 2 | 3 | 4 |
| An5 | I have energy | 0 | 1 | 2 | 3 | 4 |
| An7 | I am able to do my usual activities | 0 | 1 | 2 | 3 | 4 |
| Aa8 | I need to sleep during the day | 0 | 1 | 2 | 3 | 4 |
| An12 | I am too tired to eat | 0 | 1 | 2 | 3 | 4 |
| Anl4 | I need help doing my usual activities | 0 | 1 | 2 | 3 | 4 |
| Anl5 | I am frustrated by being too tired to do the things<br>I want to | 0 | 1 | 2 | 3 | 4 |
| Anl6 | I have to limit my social activity because I am tired | 0 | 1 | 2 | 3 | 4 |

English (Universal)

Copyright 1987, 1997

16 November 2007

Page 1 of 1



#### Appendix P. Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI:SHP) Questionnaire Example

### Work Productivity and Activity Impairment Questionnaire: Specific Health Problem V2.0 (WPAI:SHP)

The following questions ask about the effect of your PROBLEM on your ability to work a

| ınd po | erform regular activities. Please fill in the blanks or circle a number, as indicated. |
|---|---|
| 1. | Are you currently employed (working for pay)? NO YES If NO, check "NO" and skip to question 6. |
| Γhe n | ext questions are about the past 7 days, not including today. |
| 2. | During the past 7 days, how many hours did you miss from work because of problems associated with your PROBLEM? Include hours you missed on sick days, times you went in late, left early, etc., because of your PROBLEM. Do not include time you missed to participate in this study. |
| | HOURS |
| 3. | During the past 7 days, how many hours did you miss from work because of any other reason, such as vacation, holidays, time off to participate in this study? |
| | HOURS |
| 4. | During the past 7 days, how many hours did you actually work? |
| | HOURS (If "0," skip to question 6.) |



5. During the past seven days, how much did your PROBLEM affect your productivity while you were working?

Think about days you were limited in the amount or kind of work you could do, days you accomplished less than you would like, or days you could not do your work as carefully as usual. If PROBLEM affected your work only a little, choose a low number. Choose a high number if PROBLEM affected your work a great deal.

Consider only how much <u>PROBLEM</u> affected productivity <u>while you were working</u>.

| PROBLEM | | | | | | | | | | | | PROBLEM |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| had no | | | | | | | | | | | | completely |
| effect on<br>my work | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | <ul><li>prevented me from working</li></ul> |

#### CIRCLE A NUMBER

6. During the past 7 days, how much did your PROBLEM affect your ability to do your regular daily activities, other than work at a job?

By regular activities, we mean the usual activities you do, such as work around the house, shopping, childcare, exercising, studying, etc. Think about times you were limited in the amount or kind of activities you could do and times you accomplished less than you would like. If PROBLEM affected your activities only a little, choose a low number. Choose a high number if PROBLEM affected your activities a great deal.

Consider only how much <u>PROBLEM</u> affected your ability to do your regular daily activities, other than work at a job.





#### CIRCLE A NUMBER

#### WPAI:SHP V2.0 (US English)

Reilly MC, Zbrozek AS, Dukes E: The validity and reproducibility of a work productivity and activity impairment measure. PharmacoEconomics 1993; 4(5):353-365.



Appendix Q. Short Form-36 (SF-36<sup>TM</sup>) Health Status Survey Questionnaire Example

## Your Health and Well-Being

This survey asks for your views about your health. This information will help keep track of how you feel and how well you are able to do your usual activities. *Thank you for completing this survey!* 

For each of the following questions, please mark an  $\boxtimes$  in the box that best describes your answer.

1. In general, would you say your health is:

| | Excellent | Very good | Good | Fair | Poor |
|---|--------------|-----------|--------------|--------------|--------------|
| I | lacktriangle | ▼ | lacktriangle | lacktriangle | lacktriangle |
| | <u></u> 1 | <u>2</u> | <u>3</u> | <u></u> 4 | <u></u> 5 |

2. <u>Compared to 1 year ago</u>, how would you rate your health in general <u>now</u>?

| Much better now than one year ago | Somewhat better<br>now than one year<br>ago | About the same as one year ago | Somewhat worse<br>now than one year<br>ago | Much worse now than one year ago |
|---|---|---|---|---|
| lacktriangle | lacktriangle | lacktriangle | lacktriangle | lacktriangle |
| <u></u> 1 | <u>2</u> | <u>3</u> | <u></u> 4 | <u></u> 5 |

3. The following questions are about activities you might do during a typical day. Does your health now limit you in these activities? If so, how much?

| | | Yes,<br>limited<br>a lot | Yes,<br>limited<br>a little | No, not<br>limited<br>at all |
|---|---|---|---|---|
| ı | <u>Vigorous activities</u> , such as running, lifting heavy objects, participating in strenuous sports | □1 | □2 | □3 |
| ) | Moderate activities, such as moving a table, pushing a vacuum cleaner, bowling, or playing gol | f 🔲1 | <u> </u> | <u></u> 3 |
| : | Lifting or carrying groceries | <u> </u> | <u>2</u> | <u></u> 3 |
| ł | Climbing several flights of stairs | <u></u> 1 | <u>2</u> | <u></u> 3 |
| • | Climbing one flight of stairs | <u>1</u> | $\square 2$ | <u></u> 3 |
| Ĩ | Bending, kneeling, or stooping | <u> </u> | $\square 2$ | <u>3</u> |
| 3 | Walking more than a mile | <u> </u> | $\square 2$ | <u></u> 3 |
| 1 | Walking several hundred yards | <u> </u> | $\square 2$ | <u></u> 3 |
| | Walking one hundred yards | <u> </u> | $\square 2$ | <u>3</u> |
| | Bathing or dressing yourself | <u></u> 1 | $\square 2$ | <b>3</b> |



4. During the <u>past 4 weeks</u>, how much of the time have you had any of the following problems with your work or other regular daily activities <u>as a result of your physical health?</u>

| | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
|---|---|---|---|---|---|
| <sup>a</sup> Cut down on the <u>amount of time</u> you spent on work or other activities | <u></u> 1 | <u></u> | <u>3</u> | <u></u> 4 | <u></u> 5 |
| Accomplished less than you would like | <u> </u> | <u></u> | <u></u> 3 | <u></u> 4 | <u></u> 5 |
| Were limited in the <u>kind</u> of work or other activities | <u></u> 1 | <u></u> | <u></u> 3 | <u></u> 4 | <u></u> 5 |
| Had <u>difficulty</u> performing the work or other activities (for example, it took extra effort) | | <u></u> | <b>□</b> 3 | <u></u> 4 | <u></u> 5 |



| problen | the <u>past 4 weeks</u> , hons with your work on all problems (such a | r other regu | ılar daily | activities | as a resi | | llowing |
|---|---|---|---|---|---|---|---|
| | | | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
| <sup>a</sup> Cut down on<br>on work or othe | the <u>amount of time</u> you er activities | spent | <u> </u> | 2 | <u></u> 3 | <u></u> 4 | <u></u> |
| b Accomplishe | ed less than you would li | ke | <u> </u> | <u></u> | <u></u> 3 | <u>4</u> | <u></u> 5 |
| ° Did work or o | other activities <u>less care</u> | <u>fully</u> | | <u></u> 2 | 3 | <u></u> 4 | <u></u> 5 |
| problen | the past 4 weeks, to<br>ns interfered with yours, or groups? | | - | | | | |
| Not at all | Slightly | Mode | rately | Quite | a bit | Extre | mely |
| <u> </u> | <u> </u> | | ]3 | | ]4 | | ]5 |
| 7. How m | uch <u>bodily</u> pain hav | e you had d | luring the | e past 4 w | eeks? | | |
| None | Very mild | Mild | Moder | rate | Severe | Very | Severe |
| <b>▼</b> | <b>▼</b> | <b>▼</b> | <b>▼</b> | 1 | <b>▼</b> | | <b>▼</b><br>□6 |

i Did you feel tired?

| 8. | | past 4 weeks, how<br>both work outside | _ | | = | normal w | ork |
|---|---|---|---|---|---|---|---|
| | Not at all | A little bit | Moderately | Qu | ite a bit | Extr | emely |
| | <b>▼</b> | <b>▼</b> | <u>3</u> | | <b>V</b> □4 | | <b>▼</b><br>]5 |
| 9. | the past 4 w | tions are about how<br>veeks. For each qu<br>you have been feel | uestion, please g | ive the or | ne answer | that come | es closes |
| | | | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
| a D | oid you feel full of | f life? | _1 | <u></u> | <u>3</u> | <u></u> 4 | <u></u> 5 |
| b H | lave you been ver | y nervous? | _1 | <u>2</u> | <u></u> 3 | <u>4</u> | <u></u> 5 |
| с Н | ave you felt so do<br>that nothing coul | | | <u>2</u> | <u>3</u> | <u></u> 4 | <u></u> 5 |
| <sup>d</sup> H | lave you felt calm | and peaceful? | <u></u> 1 | <u>2</u> | <b>□</b> 3 | <u>4</u> | <u></u> 5 |
| e D | oid you have a lot | of energy? | <u></u> 1 | <u>2</u> | <b>□</b> 3 | <u>4</u> | <u></u> 5 |
| f H | ave you felt dowr depressed? | nhearted and | | <u>2</u> | 3 | <u></u> 4 | <u></u> 5 |
| g D | oid you feel worn | out? | _1 | <u>2</u> | <u>3</u> | <u></u> 4 | <b>□</b> 5 |
| h H | Iave you been hap | ру? | _1 | <u>2</u> | <u>3</u> | <u></u> 4 | <u></u> 5 |

 $\square 1$ 

 $\square 2$ 

**□**3

<u>\_\_\_4</u>

<u>\_\_\_\_</u>5

10. During the <u>past 4 weeks</u>, how much of the time has your <u>physical health or emotional problems</u> interfered with your social activities (like visiting friends, relatives, etc.)?

| All of the time | Most of the time | Some of the time | A little of the time | None of the time |
|---|---|---|---|---|
| <u> </u> | <u>2</u> | <u>3</u> | <b>_</b> 4 | <u></u> 5 |

11. How TRUE or FALSE is <u>each</u> of the following statements for you?

| | Definitely true | Mostly true | Don't<br>know | Mostly<br>false | Definitely false |
|---|---|---|---|---|---|
| <sup>a</sup> I seem to get sick a little easier than other people | <u></u> 1 | <u></u> | <u>3</u> | <u>4</u> | <u></u> 5 |
| <sup>b</sup> I am as healthy as anybody I know | <u> </u> | <u>2</u> | <b>□</b> 3 | <u></u> 4 | <u></u> 5 |
| <sup>c</sup> I expect my health to get worse | <u> </u> | <u>2</u> | <u></u> 3 | <u>4</u> | <u></u> 5 |
| <sup>d</sup> My health is excellent | <u> </u> | <u>2</u> | <b>□</b> 3 | <u>4</u> | <u></u> 5 |

#### THANK YOU FOR COMPLETING THESE QUESTIONS

 $SF-36v2^{TM}$  Health  $Survey^{\mathbb{C}}$  1996, 2000 by QualityMetric Incorporated and Medical Outcomes Trust. All Rights Reserved.

SF-36 $^{\$}$  is a registered trademark of Medical Outcomes Trust (SF-36v2 Standard, US Version 2.0)



### Appendix R. Rheumatology Common Toxicity Criteria v.2.0 Example

For designation of adverse event terms not shown in the Rheumatology Common Toxicity Criteria v.2.0 table, the approach described in Row 1 should be used.



#### Rheumatology Common Toxicity Criteria v.2.0

Based on Woodworth TG, et al. Standardizing assessment of adverse effects in rheumatology clinical trials II. Status of OMERACT Drug Safety Working Group May 2006: OMERACT 8. Standardizing Assessment and Reporting of Adverse Effects in Rheumatology Clinical Trials: Enabling Description of Comparative Safety Profiles for Anti-Rheumatic Therapies

| Safety Profiles for An | ti-Rheumatic Therapies | | | |
|---|---|---|---|---|
| | 1 – Mild | 2 – Moderate | 3 – Severe | 4 – Includes Life Threatening |
| | Asymptomatic, or transient<br>Short duration (< 1 week)<br>No change in life style<br>No medication or OTC | Symptomatic Duration (1 – 2 weeks) Alter lifestyle occasionally Meds relieve. (may be prescription) Study drug continued | Prolonged symptoms, reversible, major functional impairment Prescription meds/partial relief May be hospitalized < 24 hr Temporary study drug discontinuation, or/and dose reduced | At risk of death Substantial disability, especially if permanent. Multiple meds Hospitalised > 24 hr Study drug discontinued |
| A. Allergic/Immunol | ogic | | | |
| A1. Allergic reaction/ hypersensitivity (includes drug fever) | Transient rash: drug fever < 38°C: transient, asymptomatic bronchospasm | Generalised urticaria responsive to meds; or drug fever > 38°C, or reversible bronchospasm | Symptomatic bronchospasm requiring meds; symptomatic urticaria persisting with meds, allergy related oedema/angioedema | Anaphylaxis, laryngeal/pharyngeal oedema, requiring resuscitation |
| A2. Autoimmune reaction | Seriologic or other evidence of<br>autoimmune reaction, but patient<br>asymptomatic: all organ function<br>normal and no treatment is<br>required (e.g., vitiligo) | Evidence of autoimmune reaction involving a non-essential organ or functions, requiring treatment other than immunosuppressive drugs (e.g., hypothyroidism) | Reversible autoimmune reaction involving function of a major organ or toxicity requiring short term immunosuppressive treatment (e.g., transient colitis or anaemia) | Causes major organ dysfunction, or<br>progressive, not reversible, or<br>requires long term administration<br>of high dose immunosuppressive<br>therapy |
| A3. Rhinitis<br>(includes sneezing,<br>nasal stuffiness, post<br>nasal discharge) | Transient, non-prescription meds relieve | Prescription med. required, slow | Corticosteroids or other prescription med. with persistent disabling symptoms such as impaired exercise tolerance | NA |
| A4. Serum sickness | Transient, non-prescription meds relieve | Symptomatic, slow response to meds (e.g., oral corticosteroids) | Prolonged; symptoms only partially relieved by meds; parenteral corticosteroids required | Major organ dysfunction, requires long-term high-dose immunosuppressive therapy |



| A. Allergic/Immunole | ogic (continued) | | | |
|---|---|---|---|---|
| A5. Vasculitis | Localised, not requiring treatment; or rapid response to meds; cutaneous | Symptomatic, slow response to meds (e.g., oral corticosteroids) | Generalised, parenteral corticosteroids required or/and short duration hospitalisation | Prolonged, hospitalisation, ischemic changes, amputation |
| B. Cardiac | | | | |
| B1. Arrhythmia | Transient, asymptomatic | Transient, but symptomatic or recurrent, responds to meds | Recurrent/persistent; maintenance prescription | Unstable, hospitalisation required, parenteral meds |
| B2. Cardiac function decreased | Asymptomatic decline in resting ejection fraction by > 10%, but < 20% of baseline value | Asymptomatic decline of resting ejection fraction ≥ 20% of baseline value | CHF responsive to treatment | Severe or refractory CHF |
| B3. Edema | Asymptomatic (e.g., 1 + feet/calves), self-limited, no therapy required | Symptomatic (e.g., 2 + feet/calves), requires therapy | Symptoms limiting function (e.g., 3 + feet/calves, 2 + thighs), partial relief with treatment prolonged | Anasarca; no response to treatment |
| B4. Hypertension<br>(new onset or<br>worsening) | Asymptomatic, transient increase<br>by > 20 mmHg (diastolic) or to<br>> 150/100 if previously normal,<br>no therapy required | Recurrent or persistent increase > 150/100 or by > 10 mmHg (diastolic), requiring and responding readily to treatment | Symptomatic increase > 150/100,<br>> 20 mmHg, persistent, requiring<br>multi agency therapy, difficult to<br>control | Hypertensive crisis |
| B5. Hypotension<br>(without underlying<br>diagnosis) | Transient, intermittent,<br>asymptomatic, orthostatic<br>decrease in blood pressure<br>> 20 mmHg | Symptomatic, without interference with function, recurrent or persistent > 20 mmHg decrease, responds to treatment | Syncope or symptomatic, interferes with function, requiring therapy and sustained medical attention, dose adjustment or drug discontinuation | Shock |
| B6. Myocardial ischaemia | Transient chest pain/ECG changes; rapid relief with nitro | Recurring chest pain, transient<br>ECG ST-T changes; treatment<br>relieves | Angina with infarction, no or minimal functional compromise, reduce dose or discontinue study drug | Acute myocardial infarction, arrhythmia or/and CHF |



| B. Cardiac (continue | d) | | | |
|---|---|---|---|---|
| B7. Pericarditis/<br>pericardial effusion | Rub heard, asymptomatic | Detectable effusion by<br>echocardiogram, symptomatic<br>NSAID required | Detectable on chest x-ray,<br>dyspnoea; or pericardiocentesis;<br>requires corticosteroids | Pulsus alternates with low cardiac output; requires surgery |
| B8.<br>Phlebitis/thrombosis/<br>Embolism (excludes<br>injection sites) | Asymptomatic, superficial, transient, local, or no treatment required | Symptomatic, recurrent, deep vein thrombosis, no anticoagulant therapy required | Deep vein thrombosis requiring anticoagulant therapy | Pulmonary embolism |
| C. General (Constitu | tional) | | | |
| C1. Fatigue/malaise (asthenia) | Increase over baseline; most usual daily functions maintained, short term | Limits daily function intermittently over time | Interferes with basic ADL, persistent | Unable to care for self, bed or wheelchair bound > 50% of day debilitating, hospitalisation |
| C2. Fever (pyrexia) (note: fever due to drug allergy should be coded as allergy) | Transient, few symptoms 37.7 – 38.5°C | Symptomatic, recurrent 38.6 – 39.9°C. Relieved by meds | $\geq$ 40°C; $\leq$ 24 h, persistent symptoms; partial response to meds. | ≥ 40°C, debilitating, > 24 h, hospitalisation; no relief with meds |
| C3. Headache | Transient or intermittent, no meds or relieved with OTC | Persistent, recurring, non-narcotic analgesics relieve | Prolonged with limited response to narcotic medicine | Intractable, debilitating, requires parenteral meds. |
| C4. Insomnia | Difficulty sleeping, short term, no interfering with function | Difficulty sleeping interfering with function, use of prescription med. | Prolonged symptoms, with limited response to narcotic meds | Debilitating, hospitalisation; no relief with meds |
| C5. Rigors, chills | Asymptomatic, transient, no meds, or non-narcotic meds relieve | Symptomatic, narcotic meds relieve. | Prolonged symptoms, with limited response to narcotic meds | Debilitating, hospitalisation; no relief with meds |
| C6. Sweating (diaphoresis) | Episodic, transient | Frequent, short term | Frequent, drenching, disabling | Dehydration, requiring IV fluids/hospitalization > 24 hrs |
| C7. Weight gain | 5% – 9.9% | 10% – 19.9% | 20% – 30% | NA |
| C8. Weight loss | 5% - 9.9% | 10% – 19.9% | 20% – 30% | NA |



| D. Dermatologic | | | | |
|---|---|---|---|---|
| D1. Alopecia | Subjective, transient | Objective, fully reversible | Patchy, wig used, partly reversible | Complete, or irreversible even if patchy |
| D2. Bullous eruption | Localised, asymptomatic | Localised, symptomatic, requiring treatment | Generalised, responsive to treatment; reversible | Prolonged, generalised, or requiring hospitalisation for treatment |
| D3. Dry skin | Asymptomatic, controlled with emollients | Symptoms eventually (1 – 2 wks) controlled with emollients | Generalised, interfering with ADL > 2 wks, persistent pruritis, partially responsive to treatment | Disabling for extended period,<br>unresponsive to ancillary therapy<br>and requiring study drug<br>discontinuation for relief |
| D4. Injection site reaction | Local erythema, pain, pruritis,<br>< few days | Erythema, pain, oedema, may include superficial phlebitis, 1 – 2 wks | Prolonged induration, superficial ulceration; includes thrombosis | Major ulceration necrosis requiring surgery |
| D5. Petechiae (without vasculitis) | Few, transient asymptomatic | Dependent areas, persistent up to 2 wks | Generalised, responsive to treatment; reversible | Prolonged, irreversible, disabling |
| D6. Photosensitivity | Transient erythema | Painful erythema and oedema requiring topical treatment | Blistering or desquamation, requires systematic corticosteroids | Generalised exfoliation or hospitalisation |
| D7. Pruritis | Localised, asymptomatic, transient, local treatment | Intense, or generalised, relieved by systematic medication | Intense or generalised; poorly controlled despite treatment | Disabling, irreversible |
| D8. Rash (not bullous) | Erythema, scattered<br>macular/popular eruption; pruritis<br>transient; TOC or no meds | Diffuse macular/popular eruption<br>or erythema with pruritus; dry<br>desquamation; treatment required | Generalised, moist desquamation, requires systemic corticosteroids; responsive to treatment; reversible | Exfoliative or ulcerating; or requires hospitalisation; or parenteral corticosteroids |
| D9. Indurartion/<br>fibrosis/Thickening<br>(not sclerodermal) | Localized, high density on palpation, reversible, no effect on ADL and not disfiguring | Local areas < 50% body surface,<br>not disfiguring, transient<br>interference with ADL, reversible | Generalized, disfiguring, interferes with ADL, reversible | Disabling, irreversible, systemic symptoms |
| E. Ear/Nose/Throat | | | | |
| E1. Hearing loss | Transient, intermittent, no interference with function | Symptomatic, treatment required, reversible | Interferes with function; incomplete response to treatment | Irreversible deafness |
| E2. Sense of smell | Slightly altered | Markedly altered | Complete loss, reversible | Complete loss, without recovery |



EudraCT 2015-003334-27

| E3. Stomatitis | Asymptomatic | Painful, multiple, can eat | Interferes with nutrition, slowly reversible | Requires enteral support; residual dysfunction |
|---|---|---|---|---|
| E4. Taste<br>disturbance<br>(dysgeusia) | Transiently altered; metallic | Persistently altered; limited effect on eating | Disabling, effect on nutrition | NA |
| E5. Tinnitus | Intermittent, transient, no interference with function | Requires treatment, reversible | Disabling, or associated with hearing loss | Irreversible deafness |
| E6. Voice changes<br>(includes hoarseness,<br>loss of voice,<br>laryngitis) | Intermittent hoarseness, able to vocalise | Persistent hoarseness, able to vocalise | Whispered speech, slow return of ability to vocalise | Unable to vocalize for extended |
| E7. Xerostomia (dry mouth) | Transient dryness | Relief with meds | Interferes with nutrition, slowly reversible | Extended duration interference with nutrition, requires parenteral nutrition |
| F. Eye/Ophthalmolog | gic | | | |
| F1. Cataract | Asymptomatic, no change in vision, non-progressive | Symptomatic, partial visual loss, progressive | Symptoms impairing function, vision loss requiring treatment, including surgery | NA |
| F2. Conjunctivitis | Asymptomatic, transient, rapid response to treatment | Symptomatic, responds to treatment, changes not interfering with function | Symptoms prolonged, partial response to treatment, interferes with function | NA |
| F3. Lacrimation increased (tearing, watery eyes) | Symptoms not requiring treatment, transient | Symptomatic, treatment required, reversible | Unresponsive to treatment with major effect on function | NA |
| F4. Retinopathy | Asymptomatic, non-progressive, no treatment | Reversible change in vision; readily responsive to treatment | Disabling change in vision ophthalmological findings reversible, sight improves over time | Loss of sight |



| F. Eye/Ophthalmolo | gic (continued) | | | |
|---|---|---|---|---|
| F5. Vision changes<br>(e.g., blurred,<br>photophobia, night<br>blindness, vitreous<br>floaters) | Asymptomatic, transient, no treatment required | Symptomatic, vision changes not interfering with function, reversible | Symptomatic, vision changes interfering with function | Loss of sight |
| F6. Xerophtalmia (dry eyes) | Mild scratchiness | Symptomatic without interfering with function, requires artificial tears | Interferes with vision/function, corneal ulceration | Loss of sight |
| G. Gastrointestinal | | | | |
| G1. Anorexia | Adequate food intake, minimal weight loss | Symptoms requiring oral nutritional supplementation | Prolonged, requiring iv support | Requires hospitalization for nutritional support |
| G2. Constipation | Asymptomatic, transient, responds to stool softener, OTC laxatives | Symptomatic, requiring prescription laxatives, reversible | Obstipation requiring medical intervention | Bowel obstruction. Surgery required. |
| G3. Diarrhea | Transient, increase of 2 – 3 stools/day over pre-treatment (no blood or mucus), OTC agents relieve | Symptomatic, increase 4 – 6 stools/day, nocturnal stools, cramping, requires treatment with prescription meds. | Increase > 6 stools/day, associated with disabling symptoms, e.g., incontinence, severe cramping, partial response to treatment. | Prolonged, dehydration,<br>unresponsive to treatment, requires<br>hospitalization. |
| G4. Dyspepsia (heartburn) | Transient, intermittent, responds to OTC antacids, H-2 blockers | Prolonged, recurrent, requires prescription meds, relieved by meds | Persistent despite treatment,<br>interferes with function, associated<br>with GI bleeding | NA |
| G5. GI bleed<br>(gastritis, gastric or<br>duodenal ulcer<br>diagnosed-define<br>aetiology) | Asymptomatic, endoscopic finding, haemocult + stools, no transfusion, responds rapidly to treatment | Symptomatic, transfusion ≤ 2 units needed; responds to treatment | Haematemesis, transfusion 3 – 4 units, prolonged interference with function | Recurrent, transfusion > 4 units, perforation, requiring surgery, hospitalisation |
| G6. Haematochezia (rectal bleeding) | Haemorrhodial, asymptomatic, no transfusion | Symptomatic, transfusion ≤ 2 units, reversible | Recurrent, transfusion > 3 - 4 units | > 4 units, hypotension, requiring hospitalization |



| G. Gastrointestinal ( | continued) | | | |
|---|---|---|---|---|
| G7. Hepatitis | Laboratory abnormalities, asymptomatic, reversible | Symptomatic laboratory<br>abnormalities, not interfering with<br>function, slowly reversible | Laboratory abnormalities persistent > 2 wks, symptoms interfere with function | Progressive, hepato-renal, anasarca, pre-coma or coma |
| G8. Nausea, or<br>nausea/vomiting (use<br>diagnostic term) | Transient, intermittent, minimal interference with intake, rapid response to meds. | Persistent, recurrent, requires prescription meds, intake maintained | Prolonged, interferes with daily function and nutritional intake, periodic iv fluids | Hypotensive, hospitalization, parenteral nutrition, unresponsive to out-patient management |
| G9. Pancreatitis | Anylase elevation, intermittent nausea/vomiting, transient, responds rapidly to treatment | Amylase elevation with abdominal pain, nausea, occasional vomiting, responsive to treatment | Severe, persistent abdominal pain<br>with pancreatitic enzyme elevation,<br>incomplete or slow response to<br>treatment | Complicated by shock,<br>haemorrhage (acute circulatory<br>failure) |
| G10. Proctitis | Perianal pruritus, haemorrhoids<br>(new onset), transient, or<br>intermittent, relieved by OTC<br>meds | Tenesmus or ulcerations, anal fissure, responsive to treatment, minimal interference with function | Unresponsive to treatment, marked interference with function | Mucosal necrosis with haemorrhage, infection, surgery required. |
| H. Musculoskeletal | | | | |
| H1. Avascular necrosis | Asymptomatic MRI changes, non-progressive | MRI changes and symptoms responsive to rest and analgesia | MRI changes, symptoms requiring surgical intervention | Wheelchair bound; surgical repair not possible |
| H2. Arthralgia | Intermittent transient symptoms, no meds or relieved by OTC meds | Persistent or recurrent symptoms, resolve with meds, little effect on function | Severe symptoms despite meds impairs function | Debilitating, hospitalisation required for treatment |
| H3. Leg cramps | Transient, intermittent, does not interfere with function | Recurrent symptoms, minimally interferes with function or sleep, responds to meds | Persistent, prolonged interference<br>with function or sleep, partial or no<br>response to meds | NA |
| H4. Myalgia | Occasional; does not interfere with function | Frequent, requires meds<br>(non-narcotic); minor effects on<br>function | Major change in function/lifestyle, narcotic pain meds | Debilitating, profound weakness, requires wheelchair, unresponsive to meds |



| I1. Anxiety or | Symptomatic, does not interfere | Frequent symptoms, responds to | Persistent, prolonged symptoms, | Suicidal ideation or danger to self |
|---|---|---|---|---|
| Depression (mood alteration) | with function; no meds | meds; interferes with ADL at times | partial or no response to meds,<br>limits daily function | Sulcidar ideation of danger to sen |
| I2. Cerebrovascular ischaemia | NA | Single transient ischaemic event, responsive to treatment | Recurrent transient ischaemic events | Cerebrovascular vascular accident with permanent disability |
| I3. Cognitive disturbance | Subjective symptoms, transient, intermittent, not interfering with function | Objective symptoms, persisting, interferes with daily function occasionally | Persistent, or worsening objective symptoms; interferes with routine daily routine | Debilitating/disabling and permanent; toxic psychosis |
| I4. Depressed consciousness (somnolence) | Observed, transient, intermittent, not interfering with function | Somnolence or sedation, interfering with function | Persistent, progressive, obundation, stupor | Coma |
| I5. Inability to concentrate | Subjective symptoms, does not interfere with function | Objective findings, interferes with function | Persistent, prolonged objective findings or organic cause | NA |
| I6. Insomnia (in absence of pain) | Occasional difficulty sleeping,<br>transient intermittent, not<br>interfering with function | Recurrent difficulty sleeping;<br>requires meds for relief; occasional<br>interference with function | Persistent or worsening difficulty sleeping; severely interferes with routine daily function | NA |
| I7. Libido decreased | Decrease in interest | Loss of interest; influences relationship | Persistent, prolonged interfering with relationship | NA |
| I8. Peripheral motor neuropathy | Subjective or transient loss of deep tendon reflexes; function maintained | Objective weakness, persistent, no significant impairment of daily function | Objective weakness with substantial impairment of function | Paralysis |
| I9. Peripheral sensory neuropathy (sensory disturbance) | Subjective symptoms without objective findings, transient, not interfering with function | Objective sensory loss, persistent, not interfering with function | Prolonged sensory loss or paraethesias interfering with function | NA |
| I10. Seizure | NA | Recurrence of old seizures,<br>controlled with adjustment of<br>medication | Recurrence/exacerbation with partial response to medication | Recurrence not controlled, requiring hospitalization; new seizures |



| I. Neuropsychiatric | (continued) | | | |
|---|---|---|---|---|
| II1. Vertigo (dizziness) | Subjective symptoms, transient, intermittent, no treatment | Objective findings, recurrent, meds relieve, occasionally interfering with function | Persistent, prolonged, interfering with daily function; partial response to medication | Debilitating without response to medication, hospitalization |
| J. Pulmonary | | | | |
| J1. Asthma | Occasional wheeze, no interference with activities | Wheezing, requires oral meds, occasional interference with function | Debilitating, requires nasal O <sub>2</sub> | Requires ventilator assistance |
| J2. Cough | Transient, intermittent, occasional OTC meds relieve | Persistent, requires narcotic or other prescription meds for relief | Recurrent, persistent coughing spasms without consistent relief by meds, interferes with function | Interferes with oxygenation; debilitating |
| J3. Dyspnea | Subjective, transient, no interference with function | Symptomatic, intermittent or recurring, interferes with exertional activities | Symptomatic during daily routine activities, interferes with function, treatment with intermittent nasal O <sub>2</sub> relieves | Symptomatic at rest, debilitating, requires constant nasal O <sub>2</sub> |
| J4. Pleuritic pain (pleurisy) | Transient, intermittent symptoms, no treatment or OTC meds relieve | Persistent symptoms, requires prescription meds for relief | Prolonged symptoms, interferes with function, requires frequent narcotic pain relief | Debilitation, requiring hospitalisation |
| J5. Pneumonitis<br>(pulmonary<br>infiltrates) | Asymptomatic radiographic changes, transient, no treatment required | Symptomatic, persistent, requiring corticosteroids | Symptomatic, requiring treatment including O <sub>2</sub> | Debilitating, not reversible; or requiring assisted ventilation |
| J6. Pulmonary<br>function decreased<br>(FVC or carbon<br>monoxide diffusion<br>capacity – DLCO) | 76% – 90% of pre-treatment value | 51% – 75% of pre-treatment value | 26% – 50% of pre-treatment value | ≤ 25% of pre-treatment value |



| Laboratory Data | | | | |
|---|---|---|---|---|
| K. Haematology | | | | |
| K1. Hgb (g/dl)<br>decrease from<br>pre-treatment | 1.0 – 1.4 | 1.5 – 2.0 | 2.1 - 2.9, or Hgb $< 8.0$ , $> 7.0$ | ≥ 3.0; or Hgb < 7.0 |
| K2. Leukopenia<br>(total WBC) × 1000 | 3.0 – 3.9 | 2.0 – 2.9 | 1.0 – 1.9 | <1.0 |
| K3. Neutropenia (× 1000) | 1.5 – 1.9 | 1.0 – 1.4 | 0.5 – 0.9 | < 0.5 |
| K4. Lymphopenia (× 1000) | 1.5 – 1.9 | 1.0 – 1.4 | 0.5 – 0.9 | < 0.5 |
| K5. Platelets (× 1000) | 75 – LLN | 50 – 74.9 | 20 – 49.9; platelet transfusion required | < 20; recurrent platelet transfusions |
| L. Chemistry | • | | | |
| L1. Hypercalcaemia (mg/dl) | 1.1 × ULN – 11.5 | 11.6 – 12.5 | 12.6 – 13.5; or symptoms present | > 13.5; or associated coma |
| L2. Hyperglycemia (mg/dl) Fasting | 140 – 160 | 161 – 250 | 251 – 500 | > 500, or associated with ketoacidosis |
| L3. Hyperkalaemia (mg/dl) | 5.5 – 5.9 | 6.0 – 6.4 | 6.5 – 7.0 or any ECG change | > 7.0 or any arrhythmia |
| L5. Hypocalcaemia (mg/dl) | 0.9 × LLN – 7.8 | 7.7 – 7.0 | 6.9 – 6.5; or associated with symptoms | < 6.5 or occurrence of tetany |
| L6. Hypoglycemia (mg/dl) | 55 – 64 (no symptoms) | 40 – 54 (or symptoms present) | 30 – 39 (symptoms impair function) | < 30 or coma |
| L7. Hyponatraemia (mg/dl) | | 125 – 129 | 120 – 124 | < 120 |
| L8. Hypokalaemia (mg/dl) | | 3.0 – 3.4 | 2.5 – 2.9 | < 2.5 |



| L. Chemistry (contin | ued) | | | |
|---|---|---|---|---|
| L9. CPK (also if polymyositis-disease* | 1.2 – 1.9 × ULN | 2.0 – 4.0 × ULN | 4.0 × ULN with weakness but<br>without life-threatening signs or<br>symptoms | > 4.0 × ULN with signs or<br>symptoms of rhabdomyolysis or<br>life-threatening |
| L10. Serum uric acid | $1.2 - 1.6 \times ULN$ | $1.7 - 2.9 \times ULN$ | $3.0 - 5.0 \times ULN$ or gout | NA |
| L11. Creatinine (mg/dL)* | 1.1 – 1.3 × ULN | 1.3 – 1.8 × ULN | 1.9 – 3.0 × ULN | > 3.0 × ULN |
| L12. SGOT (AST) | $1.2 - 1.5 \times ULN$ | $1.6 - 3.0 \times ULN$ | $3.1 - 8.0 \times ULN$ | > 8.0 × ULN |
| L13. SGPT (ALT) | $1.2 - 1.5 \times ULN$ | $1.6 - 3.0 \times ULN$ | $3.0 - 8.0 \times ULN$ | > 8.0 × ULN |
| L14. Alkaline phosphatase | $1.1 - 2.0 \times ULN$ | $1.6-3.0 \times ULN$ | $3.0-5.0 \times ULN$ | > 5.0 × ULN |
| L15. T. bilirubin | 1.1 – 1.4 × ULN | 1.5 – 1.9 × ULN | $2.0 - 3.0 \times ULN$ | > 3.0 × ULN |
| L16. LDH | $1.3 - 2.4 \times ULN$ | $2.5 - 5.0 \times ULN$ | 5.1 – 10 × ULN | > 10 × ULN |
| M. Urinalysis | | · | • | |
| M1. Haematuria | Micro only | Gross, no clots | Clots, transfusion < 2 units | Transfusion required |
| M2. Proteinuria (per 24 h) | 300 – 500 mg (tr/1+) | 501 – 1999 mg (2+) | 2 – 5.0 g (3+) nephrotic syndrome | 5.0 g (4+) anasarca |
| M3. WBC in urine | NA | NA | Indicating acute interstitial nephritis | Associated with acute renal failure |
| M4. Uric acid crystals | Present without symptoms | NA | With stones or symptoms of stones (e.g., renal colic) | Causing renal outflow obstruction and hospitalization |

OTC = over-the-counter medication; ADL = activities of daily living; IV = intravenous; ECG = electrocardiogram; CHF = congestive heart failure; MRI = magnetic resonance imaging; Hb = haemglobin; LLN = lower limit of normal; ULN = upper limit of normal; WBC = white blood cells; SLE = systemic lupus erythematosus; ANA = antinuclear antibodies; H-2 blockers = histamine-2 blockers; FVC = forced vital capacity

<sup>\*</sup> For CPK and Creatinine NCI CTC grading will be used. For CPK the following gradings apply: Grade 1: > ULN - 2.5 × ULN; Grade 2: > 2.5 - 5.0 × ULN; Grade 3: > 5.0 - 10.0 × ULN; Grade 4: > 10.0 × ULN; For Creatinine the following gradings apply: Grade 1: > 1 - 1.5 × Baseline; > ULN - 1.5 × ULN; Grade 2: > 1.5 - 3.0 × Baseline; > 1.5 - 3.0 × ULN; Grade 3: > 3.0 baseline; > 3.0 - 6.0 × ULN; Grade 4: > 6.0 × ULN.